Protocol: 331-10-238

- **Protocol number:** 331-10-238.
- **Document title:** A Long-term, Phase 3, Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Oral OPC-34712 as Adjunctive Therapy in Adults with Major Depressive Disorder, the Orion Trial.
- Version number: Amendment 4.
- **Date of the document:** 13 Jun 2014.
- **NCT number:** NCT01360866.

# Otsuka Pharmaceutical Development & Commercialization, Inc.

## Investigational Medicinal Product

Brexpiprazole (OPC-34712)

#### REVISED CLINICAL PROTOCOL

A Long-term, Phase 3, Multicenter, **O**pen-label T**r**ial to Evaluate the Safety and Tolerab**i**lity of **O**ral OPC-34712 as Adju**n**ctive Therapy in Adults with Major Depressive Disorder, the Orion Trial

Protocol No. 331-10-238 IND No. 103,958 EudraCT No. 2011-001351-37

#### CONFIDENTIAL - PROPRIETARY INFORMATION

| Drug Development Phase: | 3 |
|---|---|
| Sponsor: | Otsuka Pharmaceutical Development & Commercialization, Inc. 2440 Research Boulevard Rockville, Maryland 20850, United States |
| Sponsor Representatives: | Phone Fax E-mail |
| | Phone Fax E-mail |
| | Phone Fax E-mail |
| Immediately Reportable Event | INC Research (see Appendix 2) |
| Issue Date: Date of Amendment 1: Date of Amendment 2: Date of Amendment 3: | 11 May 2011<br>23 Nov 2011<br>16 Nov 2012<br>11 Apr 2014 |
| Date of Amendment 4: | 13 Jun 2014 |

## **Protocol Synopsis**

| Name of Company: O Development & Comm Name of Product: Bre Protocol Title: | | |
|---|---|---|
| Clinical Phase: | 3 | |
| Treatment Indication: | Major Depressive Disorder (MD | D) |
| Objective(s): | OPC-34712 (hereafter referred to | Primary: To assess the long-term safety and tolerability of oral OPC-34712 (hereafter referred to by the generic name "brexpiprazole") as adjunctive therapy in the treatment of adults with MDD. |
| | • | Secondary: To assess the long-term efficacy of oral brexpiprazole as adjunctive therapy in the treatment of adults with MDD. |
| Trial Design: | This is a multicenter, 26-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive brexpiprazole in depressed adults on concurrent antidepressant therapy (ADT). The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed the last scheduled visit of a double-blind, phase 3 brexpiprazole MDD trial and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral brexpiprazole for MDD. The original 52 week open-label trial design has been modifie in this Amendment 3 to shorten the duration of the trial to 26 weeks; ongoing subjects who have not reached their Week 26 visit will be re-consented and will follow Amendment 3 schedule of assessments. Ongoing subjects who have already completed their Week 26 visit at the time of Amendment 3 will follow Amendment 3 week 26/ET schedule of assessments at their next scheduled visit. | |
| | The trial will be organized as fol | lows: |
| | Screening/Baseline: Subjects will be screened for eligibility at the last scheduled visit of the prior double-blind phase 3 trial. Subjects will sign a separate informed consent form for participation in Trial 331-10-238 before any procedures | |

specific to the open-label trial are performed. The assessments from the last scheduled visit of the prior double-blind phase 3 trial will serve as the baseline measures for Trial 331-10-238 for any assessment that is not unique to the open-label trial. Medical history will be updated, if necessary.

Treatment Phase: Eligible subjects will receive daily treatment with open-label brexpiprazole and ADT as described in the Investigational Medicinal Product, Dose, Formulation, Mode of Administration section. Visits will occur at the end of Weeks 1, 2, 4, 8, 14, 20, and 26. All subjects will receive up to 26 weeks of open-label treatment in Trial 331-10-238.

Follow-up: Subjects will be followed for safety via telephone contact or clinic visit 30 (+ 2) days after the last dose of openlabel medication.

#### **Subject Population:**

The subject population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with brexpiprazole for MDD according to the following criteria:

- Subjects who participated in Trial 331-10-227, Trial 331-10-228 or 331-13-214 will be eligible for the 331-10-238 trial if they meet one of the following conditions:
- Subjects who completed participation in the double-blind randomization phase (ie, Week 14 visit of Phase B) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214 or
- Subjects who continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214, BUT DID NOT meet criteria for remission (defined as a Montgomery Asberg Depression Rating Scale Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214.
- Subjects who participated in another double-blind phase 3 brexpiprazole MDD trial will be eligible for 331-10-238 Trial if they have completed the last scheduled visit of the prior double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last scheduled visit of the prior double-blind phase 3 trial and

must be able to continue therapy without interruption between the double-blind and open label trials. Based on the projected enrollment estimates for the prior double-blind phase 3 brexpiprazole MDD trials, up to approximately 3,000 subjects may enroll into Trial 331-10-238.

Investigational Medicinal Product, Dose, Formulation, Mode of Administration: Trial medication (ie, investigational medicinal product [IMP]) will be provided to the investigator(s) by the sponsor (or designated agent) and will consist of open-label brexpiprazole and open-label ADTs.

Brexpiprazole: Open-label brexpiprazole will be supplied as 0.5, 1, 2, and 3-mg tablets packaged in weekly blister cards, each containing sufficient tablets for 7 (+ 2 days). Blister cards will be dispensed at each scheduled visit and at unscheduled visits if the dose of brexpiprazole is changed. All doses of brexpiprazole should be taken orally once daily and can be administered without regard to meals. For convenience, brexpiprazole may be taken with the first daily dose of ADT.

All subjects will be dosed as follows:

- The first dose of open-label brexpiprazole will be taken one day after the last dose is taken for the prior double-blind, phase 3 brexpiprazole MDD trial so that adjunctive treatment will continue without interruption. It is anticipated that the last dose of the double-blind, phase 3 brexpiprazole MDD trial will be taken the day of the last scheduled visit, ie, the day of the Screening/Baseline visit for the open-label trial. Subjects will initiate open-label dosing with brexpiprazole 0.5 mg/day for 1 week. Subjects unable to tolerate brexpiprazole 0.5 mg/day must be withdrawn from the trial.
- The dose of brexpiprazole will be increased to 1 mg/day at the Week 1 visit. Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit.
- Investigators may further increase the dose to brexpiprazole 2 mg/day and then to brexpiprazole 3 mg/day, with an interval of at least 5 days between dose increases. An interval of at least 5 days between dose adjustments is recommended for dose decreases; however, the dose of brexpiprazole can be decreased at the investigator's discretion in a step-wise manner at any time after the

- Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response.
- Subjects who tolerate a reduced dose of brexpiprazole 0.5 mg/day should be rechallenged with brexpiprazole 1 mg/day at least once during the trial. In addition, the dose of brexpiprazole can be re-escalated as necessary following any dose decrease if, in the investigator's judgment, rechallenge with a higher dose is warranted in order to identify an optimum dose for the subject. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

ADT: During the Treatment Phase of Trial 331-10-238, subjects will remain on the same assigned open-label ADT from the prior double-blind, phase 3 brexpiprazole MDD trial. The initial dose of ADT will be the same as the ADT dose taken on the last scheduled visit of the prior double-blind phase 3 trial. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). After the Week 4 visit, the dose of ADT can be modified if necessary to achieve optimum efficacy and tolerability for the treatment regimen using the following rules: 1) at least 5 days must elapse between dose increases (either brexpiprazole or ADT), 2) an interval of at least 5 days between dose adjustments (either brexpiprazole or ADT) is recommended for dose decreases; however, the ADT dose can be decreased at the investigator's discretion at any time as needed for tolerability, and 3) subjects must return to the clinic for unscheduled visits if changes to the ADT dose are required between scheduled visits.

ADTs for open-label treatment will be provided in commercial packaging (eg, bottles), with additional labeling for use in this trial, as necessary to fulfill regulatory requirements. Numbered ADT bottles to be dispensed to the subject will be assigned by the IVRS or IWRS. The ADTs to be used in this trial, including allowable doses within the therapeutic range, are as follows:

Selective Serotonin Reuptake Inhibitors:

Escitalopram (Lexapro<sup>®</sup>) tablets, 10 and 20 mg/day Fluoxetine (Prozac<sup>®</sup>) capsules, 20 and 40 mg/day Paroxetine CR (Paxil CR<sup>®</sup>) controlled-release (CR) tablets,

Paroxetine CR (Paxil CR<sup>®</sup>) controlled-release (CR) tablets 37.5 and 50 mg/day

Sertraline (Zoloft®) tablets, 100, 150, and 200 mg/day

Serotonin-norepinephrine Reuptake Inhibitors:

Duloxetine (Cymbalta<sup>®</sup>) delayed-release capsules, 40 and 60 mg/day

Venlafaxine XR (Effexor XR®) extended-release (XR) capsules, 75, 150, and 225 mg/day

All doses of ADT will be administered orally once daily except for duloxetine 40 mg/day that can be administered once daily or as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily. All ADTs can be given without regard to meals, except for venlafaxine XR which should be taken with food. Subjects should be instructed to take the ADT at approximately the same time each day, if possible.

# Criteria for Evaluation:

Primary Outcome Variable:

The primary outcome variable is the safety and tolerability of brexpiprazole which will be assessed by examining the frequency and severity of adverse events (AEs).

Secondary Outcome Variables:

Efficacy: Efficacy variables will be as follows:

- Change from baseline in Clinical Global Impression -Severity of Illness scale score;
- Mean Clinical Global Impression Improvement scale score;
- Change from baseline in Sheehan Disability Scale score.
- Change from baseline in the Inventory of Depressive Symptomatology (Self-Report) Total Score

<u>Safety:</u> In addition to AEs, safety variables to be examined in this trial will include physical examinations, vital signs, body weight, waist circumference, clinical laboratory tests (hematology, serum chemistry, urinalysis, and pregnancy tests), and electrocardiograms (ECGs). In general, descriptive

statistics of changes from baseline will be provided for safety variables based on all available data. Prospectively defined criteria will be used to identify potentially clinically relevant abnormal values for clinical laboratory tests, vital signs, ECGs, and body weight. Change from baseline in body mass index (derived programmatically from body weight and height measurements) will be summarized. In addition to the analysis of standard safety variables, other safety variables including the Simpson Angus Scale, the Abnormal Involuntary Movement Scale, the Barnes Akathisia Rating Scale, the Columbia-Suicide Severity Rating Scale, and the Massachusetts General Hospital Sexual Functioning Questionnaire will also be evaluated.

Other Outcomes: Responses to the Resource Utilization Form (RUF) will be summarized appropriately to explore the impact of treatment on health care resources.

#### Trial Duration:

The duration of this trial from first subject enrolled to last subject completed is estimated to be approximately 57 months, of which approximately 51 months are allotted for rollover of subjects from the prior double-blind phase 3 brexpiprazole MDD trials. Individual participation for subjects who complete the trial without early withdrawal will be approximately 30 weeks (26 weeks of treatment and 30-day follow-up).

## **Table of Contents**

| Protoc | col Synopsis | 2 |
|--------------|------------------------------------------|----|
| <b>Table</b> | of Contents | 8 |
| List of | f In-text Tables | 13 |
| List of | f In-text Figures | 14 |
| | f Appendices | |
| | f Abbreviations and Definitions of Terms | |
| | Introduction | |
| 1.1 | Nonclinical Studies. | |
| 1.1.1 | Efficacy Pharmacology | |
| 1.1.2 | Safety Pharmacology | |
| 1.2 | Clinical Studies | |
| 1.2.1 | Pharmacokinetics/Pharmacodynamics | |
| 1.2.2 | Major Depressive Disorder | 23 |
| 1.2.3 | Schizophrenia | |
| 1.2.4 | Other Indications | 24 |
| 1.3 | Known and Potential Risks and Benefits | 24 |
| 2 7 | Frial Rationale and Objectives | 25 |
| 2.1 | Trial Rationale | 25 |
| 2.2 | Dosing Rationale | 26 |
| 2.3 | Trial Objectives | 26 |
| 3 7 | Frial Design | 27 |
| 3.1 | Type/Design of Trial | 27 |
| 3.2 | Trial Treatments | 29 |
| 3.2.1 | Treatment Administration | 29 |
| 3.2.1.1 | Brexpiprazole | 29 |
| 3.2.1.2 | ADT | 30 |
| 3.2.2 | Dose Adjustments | 31 |
| 3.2.2.1 | Brexpiprazole | 31 |

| 3.2.2.2 | ADT | 32 |
|-----------|-------------------------------------------------|----|
| 3.3 | Trial Population | 33 |
| 3.4 | Eligibility Criteria | 33 |
| 3.4.1 | Informed Consent | 33 |
| 3.4.2 | Inclusion Criteria | 34 |
| 3.4.3 | Exclusion Criteria | 35 |
| 3.5 | Primary and Secondary Outcome Variables | 38 |
| 3.5.1 | Primary Outcome Variable | 38 |
| 3.5.2 | Secondary Outcome Variables | 38 |
| 3.5.2.1 | Efficacy Variables | 38 |
| 3.5.2.2 | Safety Variables | 39 |
| 3.5.2.3 | Other Outcome Variables | 39 |
| 3.6 | Trial Procedures | 39 |
| 3.6.1 | Schedule of Assessments | 43 |
| 3.6.1.1 | Screening/Baseline | 43 |
| 3.6.1.2 | Week 1 | 44 |
| 3.6.1.3 | Week 2 | 44 |
| 3.6.1.4 | Week 4 | 45 |
| 3.6.1.5 | Week 8 | 46 |
| 3.6.1.6 | Week 14 | 47 |
| 3.6.1.7 | Week 20 | 48 |
| 3.6.1.8 | End of Treatment (Week 26/ET) | 48 |
| 3.6.1.9 | Follow-up | 49 |
| 3.6.2 | Safety Assessments | 49 |
| 3.6.2.1 | Clinical Laboratory Tests | 49 |
| 3.6.2.2 | Physical Examination and Vital Sign Assessments | 52 |
| 3.6.2.2.1 | Physical Examination | 52 |
| 3.6.2.2.2 | Vital Signs | 53 |
| 3.6.2.3 | ECG Assessments | 54 |
| 3.6.2.4 | Other Safety Assessments | 52 |
| 3.6.2.4.1 | Simpson Angus Scale (SAS) | 55 |
| 3.6.2.4.2 | Abnormal Involuntary Movement Scale (AIMS) | 55 |

| 3.6.2.4.3 | Barnes Akathisia Rating Scale (BARS) | 55 |
|---|---|---|
| 3.6.2.4.4 | Suicidality | 56 |
| 3.6.2.4.5 | Sexual Function | 56 |
| 3.6.3 | Efficacy Assessments | 56 |
| 3.6.3.1 | Clinical Global Impression - Severity of Illness Scale (CGI-S) | 57 |
| 3.6.3.2 | Clinical Global Impression - Improvement Scale (CGI-I) | 57 |
| 3.6.3.3 | Subject Assessment Recording | 57 |
| 3.6.3.3.1 | Sheehan Disability Scale (SDS) | 57 |
| 3.6.3.3.2 | Inventory of Depressive Symptomatology (Self-Report) | 57 |
| 3.6.3.3.3 | Resource Utilization Form (RUF) | 58 |
| 3.6.4 | End of Trial | 58 |
| 3.7 | Stopping Rules, Withdrawal Criteria and Procedures | 58 |
| 3.7.1 | Entire Trial or Treatment Arm(s) | 58 |
| 3.7.2 | Individual Center | 58 |
| 3.7.3 | Individual Subject | 58 |
| 3.8 | Screen Failures | 59 |
| 3.9 | Definition of Completed Subjects | 59 |
| 3.10 | Definition of Lost to Follow-up | 60 |
| 3.11 | Subject Compliance | 60 |
| 3.12 | Protocol Deviations | 60 |
| 4 R | estrictions | 61 |
| 4.1 | Prohibited Medications | 61 |
| 4.2 | Other Restrictions | 62 |
| 4.2.1 | Restricted Therapies and Precautions | 62 |
| 4.2.2 | Non-therapy Precautions and Restrictions | 64 |
| 4.2.2.1 | Precautions | 64 |
| 4.2.2.2 | Restrictions | 64 |
| 5 R | eporting of Adverse Events | 65 |
| 5.1 | Definitions | |
| 5.2 | Eliciting and Reporting Adverse Events | |
| 5.3 | Immediately Reportable Events (IRE) | 67 |

### Protocol 331-10-238

| 5.4 | Potential Hy's Law Cases | 68 |
|---|---|---|
| 5.5 | Pregnancy | 68 |
| 5.6 | Follow-up of Adverse Events | 69 |
| 5.6.1 | Follow-up of Non-serious Adverse Events | 69 |
| 5.6.2 | Follow-up of Post Trial Serious Adverse Events | 70 |
| 5.6.3 | Follow-up and Reporting of Serious Adverse Events Occurring after Last Scheduled Contact | 70 |
| 6 | Pharmacokinetic Analysis | 70 |
| 7 | Statistical Analysis | 70 |
| 7.1 | Primary and Secondary Outcome Variable Analysis | |
| 7.1.1 | Data Sets for Analysis | 70 |
| 7.1.2 | Handling of Missing Data | 71 |
| 7.1.3 | Primary Outcome Analysis | 71 |
| 7.1.4 | Secondary Outcome Analysis | 71 |
| 7.2 | Sample Size | 71 |
| 7.3 | Analysis of Demographic and Baseline Characteristics | 72 |
| 7.4 | Safety Analyses | 72 |
| 7.4.1 | Adverse Events | 72 |
| 7.4.2 | Clinical Laboratory Data | 72 |
| 7.4.3 | Physical Examination and Vital Signs Data | 73 |
| 7.4.4 | ECG Data | 73 |
| 7.4.5 | Other Safety Data | 73 |
| 7.5 | Other Outcomes | 73 |
| 8 | Trial Drug Management | 74 |
| 8.1 | Packaging and Labeling | 74 |
| 8.2 | Storage | 75 |
| 8.3 | Accountability | 75 |
| 8.4 | Returns and Destruction | 75 |
| 8.5 | Reporting of Product Quality Complaints | 75 |
| 8.5.1 | Eliciting and Reporting Product Quality Complaints | 76 |
| 8.5.2 | Information Required for Reporting Purposes | 76 |

### Protocol 331-10-238

| 8.5.3 | Return Process | 77 |
|-----------|----------------------------------------------|----|
| 8.5.4 | Assessment/Evaluation | 77 |
| 9 | Records Management | 77 |
| 9.1 | Source Documents | 77 |
| 9.2 | Data Collection | 77 |
| 9.3 | File Management at the Trial Site | 78 |
| 9.4 | Records Retention at the Trial Site | 78 |
| 10 | <b>Quality Control and Quality Assurance</b> | 79 |
| 10.1 | Monitoring | 79 |
| 10.2 | Auditing | 79 |
| 11 | Ethics and Responsibility | 79 |
| <b>12</b> | Confidentiality | 80 |
| 13 | Amendment Policy | 80 |
| 14 | References | |

## **List of In-text Tables**

| Table 3.2.1.1-1 | Dosing Schedule for Brexpiprazole | 30 |
|---|---|---|
| Table 3.2.1.2-1 | Open-label Antidepressant Therapy (ADT) Allowable Doses Within Therapeutic Dose Ranges for MDD | 31 |
| Table 3.2.2.1-1 | Dose Modifications for Brexpiprazole | 32 |
| Table 3.4.2-1 | Inclusion Criteria | 34 |
| Table 3.4.3-1 | Exclusion Criteria | 35 |
| Table 3.6-1 | Schedule of Assessments | 40 |
| Table 3.6.2.1-1 | Safety Clinical Laboratory Tests | 51 |
| Table 4.1-1 | List of Medications Prohibited During the Trial | 61 |

## **List of In-text Figures**

| Figure 3.1-1 | Trial Design Scl | hematic 28 |
|--------------|--------------------|------------|
| | 11101 2 001811 001 | |

## **List of Appendices**

| Appendix 1 | Names of Sponsor Personnel | 84 |
|---|---|---|
| Appendix 2 | Institutions Concerned With the Trial | 86 |
| Appendix 3 | Criteria for Identifying Vital Signs of Potential Clinical Relevance 89 | |
| Appendix 4 | Criteria for Identifying Laboratory Values of Potential Clinical Relevance | 90 |
| Appendix 5 | Criteria for Identifying ECG Measurements of Potential Clinical Relevance | 91 |
| Appendix 6 | Clinical Global Impression - Severity of Illness Scale (CGI-S) 92 | |
| Appendix 7 | Clinical Global Impression - Improvement Scale (CGI-I) | 93 |
| Appendix 8 | Sheehan Disability Scale (SDS) | 94 |
| Appendix 9 | Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) 96 | |
| Appendix 10 | Simpson Angus Scale (SAS) | 99 |
| Appendix 11 | Abnormal Involuntary Movement Scale (AIMS) | 102 |
| Appendix 12 | Barnes Akathisia Rating Scale (BARS) | 103 |
| Appendix 13 | Columbia-Suicide Severity Rating Scale (C-SSRS) | 105 |
| Appendix 14 | Massachusetts General Hospital Sexual Functioning Questionnaire (MSFQ) | 110 |
| Appendix 15 | Resource Utilization Form (RUF) | 111 |
| Appendix 16 | Protocol Amendment(s)/Administrative Change(s) | 113 |

**BARS** 

#### List of Abbreviations and Definitions of Terms

**Abbreviation Definition** 

ADHD Attention-deficit/hyperactivity disorder

ADT Antidepressant therapy

AE Adverse event

AIMS Abnormal Involuntary Movement Scale

ALP Alkaline phosphatase ALT (SGPT) Alanine transaminase

APO Apomorphine

aPTT Activated partial thromboplastin time

AST (SGOT) Aspartate transaminase

AUC<sub>t</sub> Area under the concentration-time curve calculated to the last

observable concentration at time t Barnes Akathisia Rating Scale

BMI Body mass index
BUN Blood urea nitrogen

CFR Code of Federal Regulations

CGI-I Clinical Global Impression - Improvement scale
CGI-S Clinical Global Impression - Severity of Illness scale
C<sub>max</sub> Maximum (peak) plasma concentration of the drug

CNS Central nervous system
CPK Creatine phosphokinase
CR Controlled-release

C-SSRS Columbia-Suicide Severity Rating Scale

CYP Cytochrome P450

D2 Dopamine type 2 receptor
D3 Dopamine type 3 receptor
DBP Diastolic blood pressure

DSM-IV-TR Diagnostic and Statistical Manual of Mental Disorders, Fourth

Edition, Text Revision

ECG Electrocardiogram

eCRF Electronic case report form ECT Electroconvulsive therapy EPS Extrapyramidal symptoms

ET Early termination

EudraCT European Clinical Trial Data Base FDA Food and Drug Administration

5-HT Serotonin

5-HT1A Serotonin type 1A receptor 5-HT2A Serotonin type 2A receptor GABA Gamma-aminobutyric acid GCP Good Clinical Practice GGT Gamma glutamyl transferase

HAM-D17 17-item Hamilton Depression Rating Scale

HbA1c Glycosylated hemoglobin HDL High density lipoprotein

HEENT Head, eyes, ears, nose, and throat

hERG Human ether-a-go-go

HIV Human immunodeficiency virus

ICF Informed consent form

ICH International Conference on Harmonization

ID Identification

IDDM Insulin-dependent diabetes mellitus

IDS-SR Inventory of Depressive Symptomatology (Self-Report)

IEC Independent ethics committee
IMP Investigational medicinal product
INR International Normalized Ratio
IRB Institutional review board
IRE Immediately reportable event

IUD Intrauterine device

IVRS Interactive voice response system IWRS Interactive web response system

LDH Lactate dehydrogenase LDL Low density lipoprotein

LOCF Last-observation-carried-forward

MADRS Montgomery Asberg Depression Rating Scale

MDD Major depressive disorder

MedDRA Medical Dictionary for Regulatory Activities

MSFQ Massachusetts General Hospital Sexual Functioning

Questionnaire

NMS Neuroleptic malignant syndrome

OC Observed cases

OPC Otsuka Pharmaceutical Co.

OPDC Otsuka Pharmaceutical Development & Commercialization,

Inc.

OTC Over-the-counter

PET Positron emission tomography

PK Pharmacokinetic
PT Prothrombin time
OTc Corrected OT interval

QTcB QT interval as corrected by Bazett's formula QTcF QT interval as corrected by Fridericia's formula

QTcN QT interval as corrected by the FDA Neuropharm Division

formula

RBC Red blood cell

RUF Resource Utilization Form
SAE Serious adverse event
SAS Simpson Angus Scale
SBP Systolic blood pressure

#### Protocol 331-10-238

SDS Sheehan Disability Scale

**SNRI** Serotonin-norepinephrine reuptake inhibitor **SSRI** Selective serotonin reuptake inhibitor

Sequenced Treatment Alternatives to Relieve Depression STAR\*D

Thyroxine  $T_4$ 

**TEAE** Treatment-emergent adverse event

Time to maximum (peak) plasma concentration  $t_{max}$ 

Thyroid-stimulating hormone **TSH** 

Upper limit of normal **ULN** 

**United States** US **WBC** White blood cell

Women of childbearing potential **WOCBP** 

Extended-release XR

#### **Definition** Term

Investigational For the purposes of this protocol, IMP refers to all trial medicinal product medication supplied to the sites by the sponsor (or designated (IMP)

agent) and includes bottles of protocol-specified ADTs and blister

cards containing brexpiprazole.

Remission Montgomery Asberg Depression Rating Scale Total Score  $\leq 10$ .

#### 1 Introduction

Major depressive disorder (MDD) is a debilitating and chronic illness characterized by a broad spectrum of emotional and physical symptoms. Despite the availability of numerous treatments (eg, pharmacotherapy, cognitive behavioral psychotherapy, electroconvulsive therapy [ECT], etc.), achievement of consistent and favorable long-term outcomes still represents an unmet medical need. For patients who experience an initial major depressive episode, the probability of experiencing another episode at some point in the future can be as high as 85%. In addition, 15% of patients may endure chronic symptoms after the first episode, while 35% may experience recurrent episodes.<sup>2</sup> Remission rates are low for initial antidepressant monotherapy treatment (less than 30%) and partial response is common.3 Incomplete response to treatment for MDD is associated with an increased risk of relapse, 4,5 impaired social and occupational functioning, 6 and consequently, an increased economic burden. <sup>7,8</sup> Practice guidelines emphasize the importance of adequate treatment for MDD, including continuation of pharmacotherapy after an initial response is achieved to prevent relapse and maintenance treatment in individuals at risk of recurrence. Augmentation of ADT with agents such as lithium, thyroid hormone, anticonvulsants, or psychostimulants has also been explored as a possible means of achieving a more robust response to treatment.

Antipsychotics have been used in combination with antidepressants for treatment of psychotic or delusional forms of depression. However, the use of antipsychotics as adjunctive therapy for non-psychotic depression has been limited due to safety concerns, specifically, the potential for extrapyramidal symptoms (EPS), hyperprolactinemia, weight gain, and excessive sedation. The introduction of atypical antipsychotics has created a renewed interest in adjunctive therapy for MDD, particularly for treatment-resistant MDD. Although initial studies produced mixed results, several atypical antipsychotics have been shown to enhance the response to ADT. 10,11,12,13,14



schizophrenia and bipolar mania. Hence, brexpiprazole is expected to be a promising antipsychotic agent. As the relative activity at these and other receptors appears to be related to the side effect profiles of antipsychotic drugs, <sup>15,16,17,18</sup> brexpiprazole may have the potential to exhibit improved safety compared to other agents. The more potent antagonism at 5-HT2A receptors for brexpiprazole relative to aripiprazole may afford a more favorable profile with respect to sleep quality; whereas, the low binding affinities for histamine and muscarinic receptors suggest that brexpiprazole may have less potential to cause H1-receptor-related weight gain than olanzapine. Preclinical data also suggest that brexpiprazole will have lower potential for hyperprolactinemia than risperidone. Results from initial phase 2 trials showed brexpiprazole to be well tolerated by subjects with MDD and schizophrenia (see Section 1.3).

#### 1.1 Nonclinical Studies

Efficacy and safety pharmacology are summarized in Section 1.1.1 and Section 1.1.2. A complete description of the available data from nonclinical studies, including pharmacokinetic and toxicology studies in different animal species can be found in the Investigator Brochure.<sup>19</sup>

## 1.1.1 Efficacy Pharmacology

Brexpiprazole functions as a partial agonist at the D2 receptor. In in vitro assay systems based on forskolin-induced cyclic AMP accumulation and calcium (Ca<sup>2+</sup>) mobilization in human dopamine D2L receptor-expressing cells, its intrinsic activity at the D2 receptor was slightly lower than that of aripiprazole, another D2 receptor partial agonist. Brexpiprazole inhibited apomorphine (APO)-induced hyperlocomotion, APO-induced stereotyped behavior, and conditioned avoidance response in rats, which are predictive animal models for antipsychotic-like efficacy. The inhibitory effects of brexpiprazole were more potent than those of aripiprazole. Moreover, in contrast to the D2 receptor antagonist risperidone, brexpiprazole did not increase plasma prolactin levels in reserpine-treated rats, thus demonstrating a D2 receptor partial agonistic profile in vivo. Despite its lower intrinsic activity at the D2 receptor, the in vivo catalepsy liability of brexpiprazole, an index of EPS, was similar to that of aripiprazole, but still lower than that of the typical antipsychotic haloperidol. Furthermore, brexpiprazole showed high binding affinity for the 5-HT2A receptor and dose-dependently inhibited  $(\pm)$ -2,5-dimethoxy-4-iodoamphetamine-induced head twitch response in rats, indicating that the compound has 5-HT2A receptor antagonistic activity; the effect of brexpiprazole was more potent than that of aripiprazole. In addition, brexpiprazole exhibited high

binding affinities for the D3 and 5-HT1A receptors, acting as a partial agonist at these receptors.

#### 1.1.2 Safety Pharmacology

In safety pharmacology studies in rats at an oral dose of 30 mg/kg or higher, brexpiprazole induced pharmacologically mediated clinical signs considered to be due to depression of the central nervous system (CNS) and dose-dependent decreases in body temperature. When orally administered at up to 30 mg/kg in conscious male beagle dogs, brexpiprazole showed no effect on respiratory parameters or heart rate at any dose tested. Brexpiprazole decreased blood pressure at doses of 3 mg/kg or higher and prolonged both QT interval and corrected QT interval (QTc, by Van de Water's formula) at 30 mg/kg. Brexpiprazole inhibited human ether-a-go-go related gene (hERG) current in Chinese hamster ovary cells (CHO-K1) at concentrations of 10<sup>-8</sup> mol/L or higher, with a 50% inhibitory concentration of  $1.17 \times 10^{-7}$  mol/L. The mechanism for the blood pressure decreasing effect of brexpiprazole was suggested to result from a blockade of the  $\alpha_1$ -adrenoceptor in peripheral blood vessels, which is a part of the compound's pharmacological profile. Proarrhythmic risk was also evaluated by examining the effects of brexpiprazole on monophasic action potential parameters in halothane-anesthetized dogs. Brexpiprazole did not affect the terminal repolarization period even at an intravenous dose of 3 mg/kg, suggesting a low potential for proarrhythmic effects. In general, the changes in the CNS, respiratory, and cardiovascular systems observed with brexpiprazole occurred at doses or exposure levels higher than those at which efficacy was confirmed in rats (3 mg/kg), and similar changes were shown to occur after administration of risperidone at similar or lower doses.

#### 1.2 Clinical Studies

#### 1.2.1 Pharmacokinetics/Pharmacodynamics

The pharmacokinetics of single and multiple doses of brexpiprazole was studied in healthy subjects and in subjects with MDD, attention-deficit/hyperactivity disorder (ADHD), and schizophrenia or schizoaffective disorder. Based on preclinical data and human clinical trials, brexpiprazole (OPC-34712) and one metabolite, DM-3411, were identified as the major analytes that are present in human plasma. In vitro, the activity of DM-3411 is 17 times lower than that of brexpiprazole and thus is considered as an inactive metabolite. Both brexpiprazole and DM-3411 pharmacokinetics were linear following single oral doses of brexpiprazole 0.2 to 8 mg to healthy subjects. The

terminal phase elimination half-life of brexpiprazole and DM-3411 was 48.3 to 80.8 hours and 48.6 to 77.5 hours, respectively. The median time to maximum (peak) plasma concentration (t<sub>max</sub>) occurred at approximately 2 to 6 hours postdose for brexpiprazole and at approximately 10 to 24 hours postdose for DM-3411. In healthy subjects, administration of single-dose brexpiprazole with a high-fat meal did not affect its rate and extent of absorption.

Steady state pharmacokinetics also appeared to be linear following multiple daily doses of brexpiprazole in the range of 0.5 to 2 mg to healthy subjects. The accumulation factor based on maximum (peak) plasma concentration ( $C_{max}$ ) and area under the concentration-time curve calculated to the last observable concentration at time t ( $AUC_t$ ) was approximately 4 times. After multiple dose administration of brexpiprazole (1 to 12 mg/day) to subjects with schizophrenia or schizoaffective disorder, brexpiprazole and DM-3411 mean terminal elimination half-life at steady state was 95.4 and 89.3 hours, respectively; median  $t_{max}$  was 3.0 and 8.0 hours, respectively.

In drug interaction trials in healthy subjects, brexpiprazole was shown to be metabolized by CYP3A4 and CYP2D6 isozymes and was not an inhibitor of CYP3A4, CYP2B6, CYP2D6, or P-glycoprotein. Coadministration of potent CYP3A4 or CYP2D6 inhibitors with brexpiprazole resulted in about a 2-fold higher exposure and about a 1.5-fold increase in the terminal elimination half life of brexpiprazole. Of note, administration of brexpiprazole with fluoxetine, paroxetine, or duloxetine (MDD medications coadministered in this trial) may potentially increase brexpiprazole plasma concentrations by up to 2-fold.

In a single-dose trial in healthy subjects, approximately 46.0% and 24.6% of administered radioactivity following an oral dose of  $^{14}$ C-brexpiprazole was excreted in feces and urine, respectively. In this same trial, brexpiprazole did not preferentially bind to red blood cells. Brexpiprazole showed high protein binding in human serum ( $\geq 99.8\%$ ) in vitro.

The binding of brexpiprazole to dopamine receptors was assessed using positron emission tomography (PET). The mean D2/D3 receptor occupancies at 4 and 24 hours postdose after 0.25, 0.5, 1, 2, 4, 5, and 6 mg single dose administration of brexpiprazole to healthy subjects were 11.4% to 17.4%, 36.5% to 46.3%, 45.6% to 60.2%, 52.7% to 68.6%, 67.9% to 79.5%, 71.9% to 88.2%, and 69.5% to 92.6%, respectively (Trial 331-07-202). Based on the single-dose D2/D3 receptor occupancy data and steady-state pharmacokinetic/pharmacodynamic modeling, it was predicted that the

D2/D3 receptor occupancy after multiple daily dose administration of 1 to 2 mg and higher doses of brexpiprazole will result in at least 80% to 90% D2/D3 receptor occupancy.

Additional information on the pharmacokinetics/pharmacodynamics of brexpiprazole and its metabolites in humans can be found in the Investigator Brochure.<sup>19</sup>

#### 1.2.2 Major Depressive Disorder

The efficacy of brexpiprazole as adjunctive therapy for the treatment of MDD has been studied in one completed placebo-controlled trial (Trial 331-08-211). An additional placebo-controlled efficacy trial (Trial 331-09-222) and one long-term open-label safety trial (Trial 331-08-212) are ongoing. Trial 331-08-211 was a multicenter, randomized, double-blind, placebo-controlled trial designed to assess the safety and efficacy of brexpiprazole (0.15 to 2 mg daily) as adjunctive treatment to an assigned open-label ADT in subjects with MDD who have demonstrated an incomplete response to prospective treatment with the same ADT. Subjects with an incomplete response after 8 weeks of treatment with single-blind placebo plus open-label ADT were randomized to 6 weeks of double-blind treatment with either brexpiprazole-plus-ADT or placebo-plus-ADT. Responders continued to receive placebo-plus-ADT for an additional 6 weeks. Randomized subjects received brexpiprazole 0.15 mg/day,  $0.50 \pm 0.25$  mg/day,  $1.5 \pm 0.50$  mg/day, or matching placebo. Subjects randomized to the brexpiprazole  $0.50 \pm 0.25$  mg/day and brexpiprazole  $1.5 \pm 0.50$  mg/day arms were titrated to the target doses (0.50 and 1.5 mg, respectively) over a 2-week period. Dose adjustments were permitted after the subjects received 1 week of treatment at the target dose. Subjects who could not tolerate the lowest dose (brexpiprazole 0.15, 0.25, or 1.0 mg/day or matching placebo, respectively) were to be discontinued from the trial. In this trial, adjunctive brexpiprazole dosed at  $1.5 \pm 0.50$  mg/day was superior to adjunctive placebo with respect to the primary endpoint (change from Week 8 to Week 14 in Montgomery Asberg Depression Rating Scale [MADRS] Total Score) and several secondary efficacy endpoints. Ongoing Trial 331-09-222 is of similar design to Trial 331-08-211, but is exploring an expanded dose range (brexpiprazole 1 to 3 mg/day).

#### 1.2.3 Schizophrenia

A dose-ranging, placebo-controlled trial for the monotherapy treatment of adults with schizophrenia has been performed in subjects experiencing an acute exacerbation of schizophrenia (Trial 331-07-203). The outcome of this trial suggests an active dose range

of brexpiprazole 1 to 6 mg/day for the treatment of schizophrenia.<sup>21</sup> In addition to the double-blind, placebo-controlled trial, a long-term open-label safety trial (Trial 331-08-210) is ongoing.

#### 1.2.4 Other Indications

Brexpiprazole is being investigated in a proof-of-concept trial in adult ADHD (Trial 331-08-213). This is a multicenter, randomized, double-blind, placebo-controlled, flexible-dose trial in which adults with ADHD who have an incomplete/partial response to stimulant therapy in a prospective treatment phase are randomized to double-blind treatment with either brexpiprazole-plus-stimulant or placebo-plus-stimulant. This trial is ongoing; therefore, results are not available.

#### 1.3 Known and Potential Risks and Benefits

As of 31 Dec 2010, 14 clinical trials involving brexpiprazole have been completed worldwide, including 10 in the United States (US), 1 in multiple countries (including the US), 2 in Japan, and 1 in Korea. An additional 4 trials are currently ongoing (3 in the US and 1 in multiple countries [including the US]). The collective trials can be classified as follows: four phase 1 pharmacokinetic (PK) trials in healthy subjects, 2 drug interaction trials in healthy subjects, one phase 1 PET trial in healthy subjects, one phase 1b polysomnography trial in subjects with schizophrenia, five phase 1 PK trials in specific patient populations, and six phase 2 efficacy and/or safety trials. Brexpiprazole has been well tolerated by healthy volunteers at single doses up to 6 mg and at multiple doses up to 2 mg/day. In patient trials, brexpiprazole has been well tolerated at multiple doses up to 12 mg/day in subjects with schizophrenia or schizoaffective disorder, up to 4 mg/day in subjects with MDD who received concomitant ADT, and up to 4 mg/day in adults with ADHD who received concomitant stimulant therapy.

In the 11 completed phase 1 and 2 clinical trials performed under the US IND (two phase 2 trials, one phase 1b trial, and eight phase 1 trials), 673/973 (69.2%) subjects who received brexpiprazole either alone or coadministered with another marketed medication reported at least one treatment-emergent adverse event (TEAE) compared to 158/253 (62.5%) subjects who received placebo either alone or coadministered with another marketed medication. The most common TEAEs reported for brexpiprazole in the completed trials ( $\geq 5\%$  in the total brexpiprazole group and more than the total placebo group) were headache (10.6%), dizziness (8.0%), anxiety (7.1%), akathisia (7.0%), and nausea (5.5%). In the total placebo group, TEAEs that occurred in  $\geq 5\%$  of subjects were headache (9.9%), insomnia (9.1%), and constipation (5.5%).

One death was reported in the completed phase 2 trial in adults with acute schizophrenia (Trial 331-07-203). The subject was not on any investigational medicinal product (IMP) at the time of death, and the death was not considered by the investigator to be related to IMP. The incidence of serious TEAEs (fatal and non-fatal) that were reported during treatment with brexpiprazole administered either alone or coadministered with another medication (19/973 subjects, 2.0%) was comparable to placebo administered either alone or coadministered with another medication (4/253 subjects, 1.6%). Furthermore, treatment with brexpiprazole does not appear to promote suicidal behavior in subjects with MDD or schizophrenia.

Brexpiprazole did not result in any consistent, clinically relevant changes in laboratory values, vital signs (blood pressure or heart rate), or electrocardiogram (ECG) parameters in the completed phase 1 and 2 clinical trials in subjects with MDD or schizophrenia. Statistically significant increases in weight were observed with brexpiprazole relative to placebo in both sample populations. Brexpiprazole exhibited a favorable profile with respect to movement disorders in subjects with MDD at doses up to 3 mg/day (Trial 331-09-221) and in subjects with schizophrenia at doses up to 12 mg/day (Trial 331-08-205). In the dose-ranging trial that enrolled subjects who were experiencing an acute exacerbation of schizophrenia (Trial 331-07-203), an increase in the incidence of EPS was observed at the highest dose (ie, brexpiprazole  $5.0 \pm 1.0$  mg/day).

Please refer to the current Investigator Brochure for a summary of available nonclinical and clinical safety data. <sup>19</sup>

Risks associated with use of the selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs) used in Trial 331-10-238 can be found in the prescribing information for the open-label ADTs.

## 2 Trial Rationale and Objectives

#### 2.1 Trial Rationale

Investigations of the interactions between serotonin and norepinephrine following sustained treatment with SSRIs provide a pharmacological basis for use of atypical antipsychotics as an augmentation strategy in treatment-resistant MDD. At the cellular level, increased serotonergic activity from prolonged reuptake inhibition appears to attenuate the firing of noradrenergic neurons indirectly through increased activation of

5-HT2A receptors.<sup>22</sup> The resulting decrease in noradrenergic tone may contribute to the suboptimal therapeutic response observed clinically with long-term administration of SSRIs.<sup>23</sup> As brexpiprazole demonstrated antagonism at 5-HT2A receptors, the attenuated response to SSRIs may be reversed with coadministration of brexpiprazole and SSRIs, thus enhancing clinical outcomes.

Because the management of MDD may require prolonged administration of ADT(s) with or without an augmenting agent, safety monitoring for longer than the period required to achieve initial response is warranted. In the brexpiprazole clinical development program for MDD, phase 2 and phase 3 trials examined the 6-week safety and efficacy of brexpiprazole augmentation of ADTs. For phase 2, subjects who completed either of the trials had the option to enroll into an open-label rollover trial in which they received brexpiprazole for up to 52 weeks (Trial 331-08-212). The current trial (Trial 331-10-238) provides an open-label rollover option for double-blind phase 3 brexpiprazole MDD trials and will expand on the knowledge gained in these trials by assessing the long-term safety, tolerability, and efficacy of brexpiprazole when administered concomitantly with antidepressant medications.

### 2.2 Dosing Rationale

A dose range of brexpiprazole 0.5 to 3 mg/day was selected for the current open-label trial to encompass the dose range of the double-blind efficacy trials (ie, brexpiprazole 1 to 3 mg/day) and to include an option for a reduced dose for tolerability (ie, 0.5 mg/day) in order to maximize subject retention in the long-term trial. Therapeutic dose ranges of ADT are based on product labels and clinical practice. Data from phase 1 drug interaction trials (Trial 331-08-207 and Trial 331-08-208) indicated that coadministration of CYP2D6 inhibitors (eg, paroxetine, fluoxetine, and duloxetine) with brexpiprazole could cause potentially higher plasma concentrations of brexpiprazole (up to 2-fold). In order to limit the potential higher exposure of brexpiprazole when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine in the current trial.

#### 2.3 Trial Objectives

Primary: To assess the long-term safety and tolerability of oral brexpiprazole as adjunctive therapy in the treatment of adults with MDD.

Secondary: To assess the long-term efficacy of oral brexpiprazole as adjunctive

therapy in the treatment of adults with MDD.

## 3 Trial Design

#### 3.1 Type/Design of Trial

This is a multicenter, 26-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive brexpiprazole in depressed adults on concurrent ADT. The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed the last scheduled visit of a double-blind phase 3 brexpiprazole MDD trial and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral brexpiprazole for MDD. A schematic of the trial design is presented in Figure 3.1-1.

The trial will be organized as follows:

Screening/Baseline: Subjects will be screened for eligibility at the last scheduled visit of the prior double-blind phase 3 trial. Subjects will sign a separate informed consent form (ICF) for participation in Trial 331-10-238 before any procedures specific to the open-label trial are performed. The assessments from the last scheduled visit of the prior double-blind phase 3 trial will serve as the baseline measures for Trial 331-10-238 for any assessment that is not unique to the open-label trial. Medical history will be updated, if necessary.

*Treatment Phase:* Eligible subjects will receive daily treatment with open-label brexpiprazole and ADT as described in Section 3.2. Visits will occur at the end of Weeks 1, 2, 4, 8, 14, 20, and 26. All subjects will receive up to 26 weeks of open-label treatment in Trial 331-10-238 and follow the schedule of assessments described in Table 3.6-1.

*Follow-up:* Subjects will be followed for safety via telephone contact or clinic visit 30 (+ 2) days after the last dose of open-label medication.



Figure 3.1-1 Trial Design Schematic

#### 3.2 Trial Treatments

#### 3.2.1 Treatment Administration

#### 3.2.1.1 Brexpiprazole

The first dose of open-label brexpiprazole will be taken one day after the last dose is taken for the prior double-blind, phase 3 efficacy trial so that adjunctive treatment will continue without interruption. It is anticipated that the last dose of the double-blind, phase 3 efficacy trial will be taken the day of the last scheduled visit ie, the day of the Screening/Baseline visit for the open-label trial. Subjects will initiate open-label dosing with brexpiprazole 0.5 mg/day for 1 week. Subjects unable to tolerate brexpiprazole 0.5 mg/day must be withdrawn from the trial. The dose of brexpiprazole will be increased to 1 mg/day at the Week 1 visit. Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit.

Investigators may further increase the dose to brexpiprazole 2 mg/day and then to brexpiprazole 3 mg/day, with an interval of at least 5 days between dose increases. An interval of at least 5 days between dose adjustments is recommended for dose decreases; however, the dose of brexpiprazole can be decreased at the investigator's discretion in a step-wise manner at any time after the Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits. The dosing schedule is summarized in Table 3.2.1.1-1. Additional information on dose adjustments is provided in Section 3.2.2.1.

All doses of brexpiprazole should be taken orally once daily and can be administered without regard to meals. For convenience, brexpiprazole may be taken with the first daily dose of ADT.

| Table 3.2.1.1-1 Dosing Schedule for Brexpiprazole | | | | | |
|---|---|---|---|---|---|
| | Trial Visit | | | | |
| IMP | Screening/<br>Baseline | Week 1 <sup>a</sup> | Week 2 <sup>b</sup> | Week 4 <sup>b</sup> | Visits at Weeks 8, 14, and 20 b |
| Brexpiprazole (mg/day) <sup>c</sup> | 0.5 | 1 | 0.5, 1 or 2 | 0.5, 1, 2 or 3 | 0.5, 1, 2, or 3 |
| ADT <sup>d</sup> | Final dose<br>from double-<br>blind trial | No change | No change | No change | Change to ADT dose is permitted as described in Section 3.2.2.2. |

<sup>&</sup>lt;sup>a</sup>Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit.

#### 3.2.1.2 ADT

During the Treatment Phase of Trial 331-10-238, subjects will remain on the same assigned open-label ADT from the prior double-blind, phase 3 efficacy trial. Numbered ADT bottles to be dispensed to the subject will be assigned by the IVRS or IWRS. The initial dose of ADT for the open-label trial will be the same as the ADT dose taken on the last scheduled visit of the prior double-blind phase 3 trial. The ADTs to be used in Trial 331-10-238, including allowable doses within the therapeutic range, are listed in Table 3.2.1.2-1. Adjustments to the ADT dose are permitted as described in Section 3.2.2.2. If in the clinical judgment of the investigator a subject should permanently discontinue their assigned ADT or change to a different ADT, the subject must be withdrawn from the trial. All doses of ADT will be administered orally once daily except for duloxetine 40 mg/day that can be administered once daily or as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily. All ADTs can be given without regard to meals, except for venlafaxine XR, which should be taken with food. Subjects should be instructed to take the ADT at approximately the same time each day, if possible.

bStep-wise increases in the dose of brexpiprazole must be separated by at least 5 days. Although step-wise decreases in the brexpiprazole dose are permitted at any time after the Week 1 visit to a minimum of 0.5 mg/day, an interval of at least 5 days between dose adjustments is recommended. See Section 3.2.2.1 for additional information on dose adjustments. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

<sup>&</sup>lt;sup>c</sup>Subjects unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial.

<sup>&</sup>lt;sup>d</sup>Throughout Trial 331-10-238, the subject must remain on the same ADT that was assigned in the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>e</sup>It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized.

| Table 3.2.1.2-1 | Open-label Antidepressant Therapy (ADT) Allowable Doses<br>Within Therapeutic Dose Ranges for MDD | | |
|---|---|---|---|
| Generic Name Brand Nam | | Dosage Form | Allowable Doses<br>Within Therapeutic<br>Dose Range (mg/day) <sup>a</sup> |
| SSRIs | | <u>.</u> | |
| Escitalopram Lexapro® | | Tablet | 10 and 20 |
| Fluoxetine | Prozac® | Capsule | 20 and 40 |
| Paroxetine CR Paxil CR ® | | Controlled-release<br>Tablet | 37.5 and 50 |
| Sertraline | ertraline Zoloft <sup>®</sup> | | 100, 150, and 200 |
| SNRIs | | | |
| Duloxetine | Cymbalta® | Delayed-release capsule | 40 and 60 |
| Venlafaxine XR | Effexor XR Extended-release capsule | | 75, 150, and 225 |

CR = controlled release; XR = extended release.

### 3.2.2 Dose Adjustments

Dose modifications to both brexpiprazole and ADT will be permitted to optimize therapeutic benefit according to the rules described below for each treatment. However, the dose of brexpiprazole and the dose of ADT should not both be changed at the same visit.

#### 3.2.2.1 Brexpiprazole

Allowable dose modifications to the daily dose of brexpiprazole are summarized in Table 3.2.2.1-1. At least 5 days must elapse between dose increases for brexpiprazole. An interval of at least 5 days between dose adjustments is recommended for dose decreases; however, the dose of brexpiprazole can be decreased at the investigator's discretion in a step-wise manner at any time after the Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

Subjects who are unable to tolerate the 0.5 mg/day dose of brexpiprazole must be withdrawn from the trial. However, subjects whose brexpiprazole dose is decreased to

<sup>&</sup>lt;sup>a</sup>All doses are to be administered orally once daily except for duloxetine 40 mg/day that can be administered once daily or as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily. All doses should be taken at approximately the same time each day, if possible.

0.5 mg/day and who demonstrate adequate tolerability at this dose should be rechallenged with a 1 mg/day dose within approximately 6 to 8 weeks after the dose is decreased to 0.5 mg/day. If tolerability issues arise following the rechallenge, the dose may be decreased again to 0.5 mg/day. Further rechallenge at 1 mg/day may be performed at the investigator's discretion. The dose of brexpiprazole can be increased as necessary following a dose decrease at any other dose if, in the investigator's judgment, rechallenge with a higher dose is warranted in order to identify an optimum dose for the subject. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response.

| <b>Table 3.2.2.1-1 Dose M</b> | Iodifications for Brexpipraz | zole |
|---|---|---|
| Dose Increases a,b | | |
| Current Dose of Brexpiprazole | Incremental Increase | Adjusted Brexpiprazole dose |
| 0.5 mg | 0.5 mg | 1 mg |
| 1 mg | 1 mg | 2 mg |
| 2 mg | 1 mg | 3 mg |
| Dose Decreases b,c | | |
| Current Dose of Brexpiprazole | Incremental Decrease | Adjusted Brexpiprazole dose |
| 0.5 mg | Not permitted <sup>d</sup> | 0.5 mg <sup>d</sup> |
| 1 mg | 0.5 mg | 0.5 mg |
| 2 mg | 1 mg | 1 mg |
| 3 mg | 1 mg | 2 mg |

<sup>&</sup>lt;sup>a</sup>At least 5 days must elapse between dose increases.

#### 3.2.2.2 ADT

It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). *After the Week 4 visit*, the dose of ADT can be modified if necessary to achieve optimum efficacy and tolerability for the treatment regimen using the following rules: 1) at least 5 days must elapse between dose increases (either brexpiprazole or ADT), 2) an interval of at least 5 days between dose adjustments (either brexpiprazole or ADT) is recommended for dose decreases; however, the ADT dose can be decreased at the investigator's discretion at any time as needed for tolerability, and 3) subjects must return to the clinic for unscheduled visits if changes to the ADT dose are required between scheduled visits.

<sup>&</sup>lt;sup>b</sup>Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

An interval of at least 5 days between dose adjustments is recommended for dose decreases; however, the investigator may decrease the dose of brexpiprazole at any time after the Week 1 visit for tolerability.

<sup>&</sup>lt;sup>d</sup>Subjects unable to tolerate 0.5 mg/day of brexpiprazole must be withdrawn from the trial.

The Sponsor reserves the right to use a generic equivalent should any marketed antidepressant become unavailable during the course of the trial.

#### 3.3 Trial Population

The trial population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with brexpiprazole for MDD according to the following criteria:

- Subjects who participated in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214 will be eligible for Trial 331-10-238 if they meet one of the following conditions:
- Subjects who completed participation in the double-blind randomization phase (ie, Week 14 visit of phase B) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214 or
- Subjects who continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214, BUT DID NOT meet criteria for remission (defined as a MADRS Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214.
- Subjects who participated in a double-blind phase 3 brexpiprazole MDD trial will be eligible for the 331-10-238 trial if they have completed the last scheduled visit of the double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last scheduled visit of the prior double-blind phase 3 trial and must be able to continue therapy without interruption between the double-blind and open-label trials. Based on the projected enrollment estimates for the prior double-blind phase 3 brexpiprazole MDD trials, up to approximately 3,000 subjects may enroll into Trial 331-10-238.

### 3.4 Eligibility Criteria

#### 3.4.1 Informed Consent

Written informed consent will be obtained from all subjects (or their guardian or legal representative, as applicable for local laws). Consent will be documented on a written ICF. The ICF will be approved by the same Institutional Review Board/Independent Ethics Committee (IRB/IEC) that approves this protocol. Each ICF will comply with the FDA regulations in 21 Code of Federal Regulations (CFR) Part 50, International Conference on Harmonization Good Clinical Practice (ICH GCP), and local regulatory requirements. The investigator agrees to obtain approval from the sponsor of any written ICF used in the trial, prior to submission to the IRB/IEC.

Investigators may discuss trial availability and the possibility for entry with a potential subject without first obtaining consent. However, informed consent must be obtained and documented prior to initiation of any procedures that are performed solely for the purpose of determining eligibility for this trial, including withdrawal from current medication(s). The ICF for the open-label trial may be provided to potential candidates for review and discussion toward completion of the prior double-blind phase 3 trial, but the form must not be signed until the day of the Screening/Baseline visit for Trial 331-10-238 (ie, the last scheduled visit of the prior double-blind phase 3 trial).

Once appropriate essential information has been provided and fully explained in layman's language to the subject by the investigator (or a qualified designee), the IRB/IEC-approved written ICF will be signed and dated by both the subject and the person obtaining consent (investigator or designee), as well as by any other parties required by the IRB/IEC. The subject will receive a copy of the signed ICF; the original shall be kept on file by the investigator.

In addition to the English version of the ICF, the document may also be translated by the central translation vendor into local languages for use in this trial. Translation with backtranslation for confirmation will be utilized to ensure accuracy.

#### 3.4.2 Inclusion Criteria

Subjects are required to meet the following inclusion criteria:

| Tabl | Table 3.4.2-1 Inclusion Criteria |
|---|---|
| | All Subjects |
| 1. | Subjects who are able to provide written informed consent and/or consent obtained from a legally acceptable representative (as required by IRB/IEC) prior to the initiation of any protocol-required procedures. |
| 2. | Ability, in the opinion of the principal investigator, to understand the nature of the trial and follow protocol requirements, including the prescribed dosage regimens, tablet/capsule ingestion, and discontinuation of prohibited concomitant medication; to read and understand the written word in order to complete subject-reported outcomes measures; and to be reliably rated on assessment scales. |
| 3 | Male and female outpatients 18 to 65 years of age, inclusive, at the time of informed consent for Trial 331-10-238. |
| 4 | Subjects willing to discontinue all prohibited psychotropic medications starting from the time of signing the ICF and during the trial period (refer to Section 4). |

| Tab | le 3.4.2-1 Inclusion Criteria |
|---|---|
| | 331-10-227, 331-10-228 and 331-13-214 Subjects Only |
| 5. | <ul> <li>Subjects who, in the opinion of the investigator, could potentially benefit from administration of brexpiprazole as adjunctive therapy to their antidepressant therapy and who meet one of the following criteria:</li> <li>a) Subjects who completed participation in the double-blind randomization phase (ie, Week 14 visit of Phase B) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214 or</li> <li>b) Subjects who continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214, BUT DID NOT meet criteria for remission (defined as a MADRS Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227, Trial 331-10-228 or Trial 331-10-227, Trial 331-10-228 or Trial 331-10-227, Trial 331-10-228 or Trial 331-10-227, Trial 331-10-228 or Trial 331-10-227, Trial 331-10-228 or Trial 331-10-228 or Trial 331-10-227, Trial 331-10-228 or Trial 331-10-228 or Trial 331-10-229.</li> </ul> |
| | Eligible Subjects From Other Double-Blind Phase 3 Brexipiprazole MDD Trials |
| 6. | Subjects who completed the last scheduled visit of the prior double-blind phase 3 trial, and who in the opinion of the investigator, could potentially benefit from administration of brexpiprazole as adjunctive therapy to their antidepressant therapy. |

#### 3.4.3 Exclusion Criteria

Subjects entering the open-label trial at the last scheduled visit of the prior double-blind phase 3 trial will be excluded from Trial 331-10-238 if they meet any of the following exclusion criteria.

| Tabl | e 3.4.3-1 Exclusion Criteria | | |
|---|---|--|--|
| Sex a | nd Reproductive Status | | |
| 1. | Sexually active females of childbearing potential (see Section 5.5) and male subjects who are not practicing two different methods of birth control with their partner during the trial and for 30 days after the last dose of trial medication or who will not remain abstinent during the trial and for 30 days after the last dose. If employing birth control, each couple must use two of the following precautions: vasectomy, tubal ligation (subject or partner), vaginal diaphragm, IUD, birth control pill, birth control implant, birth control depot injections, condom, or sponge with spermicide. | | |
| 2. | Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving open-label brexpiprazole in Trial 331-10-238. | | |
| Admi | Administrative | | |
| 3. | Subjects with a major protocol violation during the course of their participation in the prior double-blind phase 3 trial. Minor violations such as occasional visits outside of the acceptable window or a missing blood draw will not exclude a subject from participation in Trial 331-10-238; however, continual lack of compliance with the visit schedule, trial assessments, or treatment regimen in the prior double-blind phase 3 trial would be considered a major violation that would result in exclusion from Trial 331-10-238. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility. | | |
| Targe | et Disease | | |
| 4. | Subjects who have received ECT for the current depressive episode. | | |
| 5. | Subjects who have had an inadequate response to ECT at any time in the past or who have had a vagus nerve stimulation or deep brain stimulation device implanted at any time for management of treatment-resistant depression. Subjects who have had Transcranial Magnetic Stimulation during the current major depressive episode. | | |
| 6. | Subjects with a current need for involuntary commitment or who have been hospitalized during the prior double-blind phase 3 trial for the current major depressive episode. | | |
| Tabl | e 3.4.3-1 Exclusion Criteria |
|---|---|
| 7. | Subjects with a current Axis I (DSM-IV-TR) diagnosis of: |
| | Delirium, dementia, amnestic or other cognitive disorder |
| | Schizophrenia, schizoaffective disorder, or other psychotic disorder |
| | Bipolar I or II disorder |
| | Eating disorder (including anorexia nervosa or bulimia) |
| | Obsessive compulsive disorder |
| | Panic disorder |
| | Post-traumatic stress disorder |
| 8. | Subjects with a current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, |
| 0 | schizoid, schizotypal or histrionic personality disorder. |
| 9. | Subjects experiencing hallucinations, delusions or any psychotic symptomatology in the current |
| 10 | depressive episode. |
| 10. | Subjects receiving new onset psychotherapy (individual, group, marriage, or family therapy) during the prior double-blind phase 3 trial. |
| Modi | cal History and Concurrent Diseases |
| 11. | Subjects with a response of "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal |
| 11. | Ideation with Some Intent to Act, Without Specific Plan) at entry, <b>OR</b> |
| | Subjects with a response of "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal |
| | Ideation with Specific Plan and Intent) at entry, <b>OR</b> |
| | Subjects with a response of "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual |
| | attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) at entry, <b>OR</b> |
| | Subjects who, in the opinion of the investigator (including consideration of responses on the |
| | C-SSRS throughout the prior double-blind phase 3 trial), present a serious risk of suicide. |
| | Note: "Entry" is defined as the last scheduled visit of the prior double-blind phase 3 trial. |
| 12. | Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 |
| | days; including alcohol and benzodiazepines, but excluding caffeine and nicotine. |
| 13. | Subjects with hypothyroidism or hyperthyroidism (unless condition has been stabilized with |
| | medications for at least the past 90 days) and/or an abnormal result for free T4 at |
| | screening/baseline. Eligibility of subjects excluded based on an abnormal free T4 result can be discussed with the medical monitor if, in the investigator's judgment, the subject is a suitable |
| | candidate for the trial. |
| 14. | Subjects who currently have clinically significant neurological, hepatic, renal, metabolic, |
| 1 | hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any |
| | history of myocardial infarction, congestive heart failure, HIV seropositive status/acquired |
| | immunodeficiency syndrome, chronic hepatitis B or C. Medical conditions that are minor or well- |
| | controlled may be considered acceptable if the condition does not expose the subject to an undue |
| | risk of a significant adverse event or interfere with assessments of safety or efficacy during the |
| | course of the trial. The medical monitor should be contacted in any instance where the investigator |
| | is uncertain regarding the stability of a subject's medical condition(s) and the potential impact of |
| 1.5 | the condition(s) on trial participation. |
| 15. | Subjects with IDDM (ie, any subjects using insulin) are excluded. Subjects with non-IDDM may |
| | be eligible for the trial if their condition is stable as determined by satisfying <b>ALL</b> of the following |
| | criteria: • Screening/baseline HbA1c < 7.0%, AND |
| | <ul> <li>Screening/baseline HbA1c &lt; 7.0%, AND</li> <li>Screening/baseline fasting glucose must be ≤ 125 mg/dL, AND</li> </ul> |
| | <ul> <li>Streening/baseline rasting glucose must be ≤ 123 ing/dL, AND</li> <li>Subject has been maintained on a stable regimen of oral anti-diabetic medication(s) or diabetes</li> </ul> |
| | has been well-controlled by diet during the prior double-blind phase 3 trial, <b>AND</b> |
| | Subject has not had any hospitalizations due to diabetes or complications related to diabetes |
| | during the prior double-blind phase 3 trial, AND |
| | <ul> <li>Subject's diabetes is not newly diagnosed during screening/baseline for Trial 331-10-238.</li> </ul> |
| | Continuation of subjects excluded based on abnormal laboratory test results from the |
| | J |

| Tabl | e 3.4.3-1 Exclusion Criteria |
|---|---|
| | screening/baseline visit should be discussed with the medical monitor, if in the investigator's judgement the subject is a suitable candidate for the trial. |
| 16. | Subjects with uncontrolled hypertension (DBP > 95 mmHg) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in SBP and/or a decrease of ≥ 20 mmHg in DBP after at least 3 minutes standing compared to the previous supine blood pressure, <b>OR</b> development of symptoms. |
| 17. | Subjects with known ischemic heart disease or history of myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery. |
| 18. | Subjects with epilepsy or a history of seizures, except for a single seizure episode, for instance childhood febrile seizure, post traumatic, or alcohol withdrawal. |
| Physic | eal and Laboratory Results |
| 19. | Subjects with a positive drug screen for cocaine, marijuana, or other illicit drugs are excluded and may not be retested or rescreened. Subjects with a positive urine drug screen resulting from use of prescription or OTC medications or products that in the investigator's documented opinion do not signal a clinical condition that would impact the safety of the subject or interpretation of the trial results may continue evaluation for the trial following consultation and approval by the medical monitor. |
| 20. | The following Screening/baseline laboratory test and ECG results are exclusionary: |
| | 1) Platelets $\leq 75,000/\text{mm}$ |
| | 2) Hemoglobin ≤ 9 g/dL |
| | 3) Neutrophils, absolute ≤ 1000/mm <sup>3</sup> 4) AST > 2 × ULN 5) ALT > 2 × ULN |
| | <ul> <li>6) CPK &gt; 3 × ULN, unless discussed with and approved by the medical monitor</li> <li>7) Creatinine ≥ 2 mg/dL</li> <li>8) HbA1c ≥ 7.0%</li> </ul> |
| | <ul> <li>9) Abnormal free T<sub>4</sub>, unless discussed with and approved by the medical monitor. (Note: Free T<sub>4</sub> is measured only if result for TSH is abnormal.)</li> <li>10) QTcF ≥ 450 msec</li> </ul> |
| | NOTE: In addition, subjects should be excluded if they have any other abnormal laboratory tests, vital sign results, or ECG findings which in the investigator's judgment are medically significant and that would impact the safety of the subject or the interpretation of the trial results. Criteria are provided in Appendix 3, Appendix 4, and Appendix 5 to assist investigators in their assessments of results that may be potentially medically significant, depending on the subject's medical history and clinical presentation. Eligibility should be based on the Screening/baseline laboratory test and ECG results. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility. Continuation of subjects excluded based on abnormal laboratory test and ECG results should be discussed with the medical monitor, if in the investigator's judgement, the subject is a suitable candidate for the trial. |
| Prohi | bited Therapies or Medications |
| 21. | Subjects who would be likely to require prohibited concomitant therapy during the trial (see Table 4.1-1) <sup>a</sup> . |
| Allero | ies and Adverse Drug Reactions |
| 22. | Subjects with a history of neuroleptic malignant syndrome or serotonin syndrome. |
| 23. | Subjects with a history of true allergic response (ie, not intolerance) to more than one class of medications. |

| Table | e 3.4.3-1 Exclusion Criteria |
|---|---|
| Other | |
| 24. | Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of |
| | either a psychiatric or physical (eg, infectious disease) illness must not be enrolled into this trial. |
| 25. | Any subject who, in the opinion of the investigator, should not participate in the trial. |

ALT = alanine transaminase; AST = aspartate transaminase; CPK = creatine phosphokinase; C-SSRS = Columbia-Suicide Severity Rating Scale; DBP = diastolic blood pressure; DSM-IV-TR = Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision; HbA1c = glycosylated hemoglobin; HIV = human immunodeficiency virus; IDDM = insulin-dependent diabetes mellitus; IUD = intrauterine device; NMS = neuroleptic malignant syndrome; OTC = over-the-counter; QTcF = QT interval as corrected for heart rate by Fridericia's formula; SBP = systolic blood pressure; T<sub>4</sub> = thyroxine; TSH = thyroid-stimulating hormone; ULN = upper limit of normal.

Subjects who do not qualify for the open-label trial at the Screening/Baseline visit may not be rescreened at a later date. If results of clinical laboratory tests from the last scheduled visit of the prior double-blind phase 3 trial are not available to assess eligibility, the assessment for the affected criteria should be based on the last available measurement during the respective double-blind trial. Results from the last visit of the double-blind trial should be reviewed when they become available and action should be taken as described in Section 3.6.2.1 if there are any clinically significant and/or exclusionary values.

## 3.5 Primary and Secondary Outcome Variables

#### 3.5.1 Primary Outcome Variable

The primary outcome variable is the safety and tolerability of brexpiprazole, which will be assessed by examining the frequency and severity of adverse events (AEs).

## 3.5.2 Secondary Outcome Variables

## 3.5.2.1 Efficacy Variables

Efficacy variables will be as follows:

- Change from baseline in Clinical Global Impression Severity of Illness scale (CGI-S) score;
- Mean Clinical Global Impression Improvement scale (CGI-I) score;
- Change from baseline in Sheehan Disability Scale (SDS) score.

Use of CYP2D6 inhibitors or CYP3A4 inhibitors and inducers is prohibited during the trial. Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs that are also CYP2D6 inhibitors. In order to limit the potential higher exposure of brexpiprazole when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine.

 Change from baseline in the Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) Total Score

## 3.5.2.2 Safety Variables

In addition to AEs, safety variables to be examined in this trial will include physical examinations, vital signs, body weight, waist circumference, clinical laboratory tests (hematology, serum chemistry, urinalysis, and pregnancy tests), ECGs, the Simpson Angus Scale (SAS), the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), the Columbia-Suicide Severity Rating Scale (C-SSRS), and the Massachusetts General Hospital Sexual Functioning Questionnaire (MSFQ).

Mean change from baseline and the incidence of potentially clinically relevant abnormal values will be calculated for vital signs, body weight, routine laboratory tests (including prolactin), and ECG parameters. Mean change from baseline will be calculated for coagulation parameters (prothrombin time [PT], activated partial thromboplastin time [aPTT], and International Normalized Ratio [INR]), glycosylated hemoglobin (HbA1c), thyroid-stimulating hormone (TSH), waist circumference, and body mass index (BMI; derived programmatically from body weight and height measurements). A central ECG service will be utilized to review all ECGs in order to standardize interpretations for the safety analysis. EPS will be evaluated by calculating mean change from baseline on the SAS, AIMS, and BARS. Sexual dysfunction will be evaluated as change from baseline in MSFQ score. The C-SSRS will be used to assess and classify reported suicidal behavior. By-patient listings of physical examination findings will be reviewed as a further assessment of safety.

#### 3.5.2.3 Other Outcome Variables

Responses to the Resource Utilization Form (RUF) will be summarized appropriately to explore the impact of treatment on health care resources.

#### 3.6 Trial Procedures

The duration of this trial from first subject enrolled to last subject completed is estimated to be approximately 57 months, of which approximately 51 months are allotted for rollover of subjects from prior double-blind phase 3 brexpiprazole MDD trials. Individual participation for subjects who complete the trial without early withdrawal will be approximately 30 weeks (26 weeks of treatment and 30-day follow-up). Trial assessment time points are summarized in Table 3.6-1.

| Table 3.6-1 Schedule of Assessments | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screening/<br>Baseline | O | Follow-up <sup>c</sup> | | | | | | |
| | Baseline | 1 | 2 | 4 | 8 | 14 | 20 | 26/ET <sup>b</sup> | 30 (+2) days |
| ENTRANCE CRITERIA | | | l . | I. | ı | ı | I | | |
| Informed consent d | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | |
| Medical history | X <sup>e</sup> | | | | | | | | |
| EFFICACY | | 1 | | | | | | 1 | |
| CGI-S | X | X | X | X | X | X | X | X | |
| CGI-I <sup>f</sup> | X | | | | | X | | X | |
| SDS | X | | | | | X | | X | |
| IDS-SR | X | | | | | X | | X | |
| SAFETY | <u>.</u> | • | • | • | | | • | | |
| Physical examination | X | | | | | | | X | |
| Waist circumference | X | | | | | X | | X | |
| Vital signs <sup>g</sup> | X | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>h</sup> | X | | | | | X | | X | |
| Clinical laboratory tests <sup>i</sup> | X <sup>j</sup> | | | | | $X^k$ | | $X^k$ | |
| HbA1c | x <sup>j</sup> | | | | | $X^k$ | | $X^k$ | |
| Drug screen/blood alcohol | X | X | | X | X | X | | X | |
| Urine pregnancy test | X | X | X | X | X | X | X | X | |
| (WOCBP only) <sup>m</sup> | | | | | | | | | |
| SAS | X | X | X | X | X | X | X | X | |
| AIMS | X | | | | | X | | X | |
| BARS | X | X | X | X | X | X | X | X | |
| C-SSRS <sup>n</sup> | X | X | X | X | X | X | X | X | |
| MSFQ | X | | | | | | | X | |
| Adverse events | X <sup>o</sup> | X | X | X | X | X | X | X | X |

| Table 3.6-1 Schedule of Assessments | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screening/<br>Baseline | 0 | Follow-up <sup>c</sup><br>30 (+2) days | | | | | | |
| | Dasenne | 1 | 2 | 4 | 8 | 14 | 20 | <b>26/ET</b> <sup>b</sup> | 50 (+2) days |
| Concomitant medications <sup>p</sup> | X | X | X | X | X | X | X | X | X |
| OTHER | | | | | | | | | |
| Dose adjustments q | | X | X | X | X | X | X | | |
| RUF <sup>r</sup> | X | | | | | | | X | |
| Register visit in IVRS/IWRS <sup>8</sup> | X | X | X | X | X | X | X | X | |
| IMP dispensing | X | X | X | X | X | X | X | | |
| IMP accountability | | X | X | X | X | X | X | X | |

IVRS = interactive voice response system; IWRS = interactive web response system; WOCBP = women of childbearing potential.

<sup>&</sup>lt;sup>a</sup>Screening for Trial 331-10-238 occurs simultaneously with Baseline at the last scheduled visit of the prior double-blind phase 3 trial. All assessments listed under screening need to be performed at Screening/Baseline of Trial 331-10-238; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.

<sup>&</sup>lt;sup>b</sup>If a subject discontinues prematurely before Week 26, procedures noted for Week 26 must be completed at the early termination (ET) visit. Subjects who have completed 26 weeks or more, will have the Week 26/ET procedures at their next scheduled visit.

<sup>&</sup>lt;sup>c</sup>Consists of telephone contact or clinic visit (investigator's discretion) for evaluation of safety and applies to all subjects (completers and early withdrawals).

d Informed consent for Trial 331-10-238 will occur at Screening/Baseline and must be obtained before any trial-related procedures specific to the open-label trial are performed.

<sup>&</sup>lt;sup>e</sup>Update, if necessary.

Improvement should be based on the subject's status at the last scheduled visit of the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>g</sup>Vital signs include body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Blood pressure and heart rate will be measured in the following order: supine, sitting, and standing after the subject has been in each position for at least 3 minutes. Vital signs scheduled for the same visit as blood samples are to be completed before blood is drawn.

h Standard 12-lead ECGs will be performed after the subject has been supine and at rest for ≥ 5 minutes prior to the ECG. A central ECG service will be utilized to review all ECGs in order to standardize interpretations for the safety analysis. In addition, ECG results will be evaluated at the investigational site to monitor safety during the trial. Subjects will be enrolled in Trial 331-10-238 based on the screening/baseline ECG results from the trial site. If the screening/baseline ECG results from the central reader (ie, the last scheduled visit of the prior double-blind phase 3 trial), when available, indicate a QTcF

- $\geq$  450 msec at screening/baseline, the investigator must contact the medical monitor to discuss the subject's continued participation in the trial. ECGs scheduled for the same visit as blood samples are to be completed before blood is drawn.
- <sup>1</sup>Includes hematology (including PT, aPTT, and INR), serum chemistry (including prolactin and TSH, with reflex to free thyroxine [T<sub>4</sub>] if the result for TSH is abnormal), and urinalysis.
- <sup>j</sup>Subjects must be fasting for a minimum of 8 hours prior to blood draws for screening/baseline laboratory assessments (ie, the last scheduled visit of the prior double-blind phase 3 trial).
- <sup>k</sup>Clinical laboratory tests should be drawn fasting, if possible, but must be drawn after a minimum 8-hour fast at Week 26/ET. Vital sign and ECG assessments should be completed before any blood samples are collected.
- A urine drug screen and a blood alcohol test are required at the designated times, but either or both can be conducted at any time during the trial at the discretion of the investigator.
- <sup>m</sup>All positive urine pregnancy test results must be confirmed by a serum test. Subjects with a positive serum pregnancy test result at Screening/Baseline must not be enrolled in Trial 331-10-238 and subjects with a positive serum pregnancy test result during the trial must discontinue treatment and be withdrawn from the trial. Pregnancy tests can be performed at any point during the trial if pregnancy is suspected.
- <sup>n</sup> "Since Last Visit" C-SSRS form.
- <sup>o</sup>AE recording will begin with the signing of the ICF for Trial 331-10-238.
- <sup>p</sup>All prescription and non-prescription medications taken during the trial will be recorded as concomitant medications. Details of prohibited and restricted medications are provided in Section 4.
- <sup>q</sup>Adjustments to the dose of brexpiprazole or ADT are permitted to optimize efficacy and tolerability as described in Section 3.2. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). At least 5 days must elapse between dose increases for brexpiprazole and ADT. An interval of at least 5 days between dose adjustments is also recommended for dose decreases; however, the investigator may decrease the dose of brexpiprazole or ADT as needed for tolerability according to the rules described in Section 3.2.2. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole or ADT (increases or decreases) are required between scheduled visits. All eligible subjects entering from prior double-blind phase 3 brexpiprazole MDD trials must be able to continue therapy without interruption between the double-blind and open label trials.
- <sup>r</sup>Baseline RUF is completed at Screening/Baseline for all subjects. The Follow-up RUF (as well as hospitalization questions) is completed at Week 26/ET visit.
- <sup>s</sup>The IVRS/IWRS will be accessed at unscheduled visits if new blister cards are dispensed for dose adjustment of brexpiprazole.

#### 3.6.1 Schedule of Assessments

# 3.6.1.1 Screening/Baseline

Subjects entering Trial 331-10-238 must sign the ICF for the open-label trial before any procedures specific to Trial 331-10-238 can be performed. Subjects will retain the same subject identification (Subject ID) number assigned in the prior double-blind phase 3 trial. The following procedures need to be performed at Screening/Baseline of Trial 331-10-238; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.

- Inclusion/exclusion criteria for Trial 331-10-238 will be reviewed to assure the subject's eligibility.
- Medical history will be updated, if necessary, using information from the prior double-blind phase 3 trial.
- Subjects will submit to a physical examination and assessments of waist circumference, vital signs, and ECG.
- The investigator (or qualified designee) will administer the CGI-S and CGI-I.
- Subjects will complete any Baseline instrument (ie, SDS, IDS-SR, and MSFQ).
- An adequately trained and experienced clinician will administer any EPS scale (ie, SAS, AIMS, and BARS).
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Concomitant medications will be reviewed to assure that the subject is not receiving any prohibited medications.
- Subjects will complete the Baseline RUF.
- For subjects entering Trial 331-10-238 after completing the last scheduled visit of the prior double-blind phase 3 trial, a fasting blood sample will be drawn for analysis of any clinical laboratory parameter (ie, the clinical laboratory parameters specified in Table 3.6.2.1-1) that was not drawn at the last scheduled visit of the prior double-blind phase 3 trial.
- AE recording will begin with the signing of the ICF for Trial 331-10-238.
- Trial personnel will call the interactive voice response system (IVRS) or access the interactive web response system (IWRS) to register the visit and to obtain blister card and ADT bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed. Treatment will begin with brexpiprazole 0.5 mg/day for 1 week. The ADT will be the same as the one taken during the prior double-blind phase 3 trial. The dose of ADT should not be changed at this time.

#### 3.6.1.2 Week 1

All subjects will attend a visit at Week 1 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S.
- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urine screen(s) for drugs of abuse.
- Women of childbearing potential (WOCBP) will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The dose of brexpiprazole will be increased to 1 mg/day. Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

#### 3.6.1.3 Week 2

All subjects will attend a visit at Week 2 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S.
- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.

- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized. Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

#### 3.6.1.4 Week 4

All subjects will attend a visit at Week 4 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S.
- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. If necessary, the dose of

ADT can be changed after the Week 4 visit, but not at the same visit as a change to the dose of brexpiprazole (see Section 3.2.2.2). Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.

• AEs and concomitant medications will be recorded.

#### 3.6.1.5 Week 8

All subjects will attend a visit at Week 8 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S.
- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

#### 3.6.1.6 Week 14

All subjects will attend a visit at Week 14 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S and CGI-I.
- Waist circumference will be measured.
- An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS.
- The subject will complete the IDS-SR and SDS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, and TSH, with reflex to free T4 if the result for TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing. Additional blood alcohol testing may be performed at any other time at the discretion of the investigator.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse. Additional urine drug screens may be performed at any other time at the discretion of the investigator.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

#### 3.6.1.7 Week 20

All subjects will attend a visit at Week 20 ( $\pm$  2 days) where the following evaluations will be performed:

- The investigator (or qualified designee) will administer the CGI-S.
- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

## 3.6.1.8 End of Treatment (Week 26/ET)

The Week 26 visit signifies the end of treatment. Therefore, all subjects will undergo a complete evaluation at Week 26 (± 2 days). In addition, Week 26 evaluations are to be completed, if possible, for any subject withdrawn from the trial prematurely. Since the original 52 week open-label trial design has been modified as a part of Amendment 3 to shorten the duration of the trial to 26 weeks, ongoing subjects who have not reached their Week 26 visit will be re-consented and will follow Amendment 3 schedule of assessments. Ongoing subjects who have already completed their Week 26 visit at the time Amendment 3 is approved will follow Amendment 3 week 26/ET schedule of assessments at their next scheduled visit. The following activities and assessments will occur at Week 26 (or at the ET visit, if applicable):

• The investigator (or qualified designee) will administer the CGI-S and CGI-I.

- An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- The subject will complete the MSFQ, SDS, IDS-SR, and the Follow-up RUF.
- A complete physical examination (including waist circumference) will be performed.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, and TSH, with reflex to free T<sub>4</sub> if TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test.
- Final drug accountability will be performed.
- Trial personnel will call the IVRS or access the IWRS to register completion or discontinuation from the trial.
- AEs and concomitant medications will be recorded.

#### 3.6.1.9 Follow-up

Follow-up safety information (AEs and concomitant medications) will be collected 30 (+ 2) days after the last dose of open-label medication for all subjects (completers and early withdrawals). Follow-up information can be obtained via telephone contact or clinic visit at the investigator's discretion.

# 3.6.2 Safety Assessments

#### 3.6.2.1 Clinical Laboratory Tests

As it is unlikely that the final laboratory test results from the last scheduled visit of the prior double-blind phase 3 trial will be available at the time of enrollment in Trial 331-10-238, the investigator is to review the subject's most recent laboratory test results from the prior double-blind phase 3 trial for compliance with the exclusion criteria

and the presence of abnormal laboratory test results that, in the investigator's judgment, are medically significant and would impact the safety of the subject or the interpretation of the trial results. Subjects meeting any of these criteria will be excluded from Trial 331-10-238. Appendix 4 is included to assist investigators in their assessments of results that may be potentially medically significant, depending on the subject's medical history and clinical presentation. If one or more results from the screening/baseline sample are clinically significant and/or exclusionary when the results from the last scheduled visit of the prior double-blind phase 3 trial become available, the test(s) should be repeated. The subject may continue to receive trial medication pending results of the repeat laboratory tests at the investigator's discretion. If the abnormality remains upon retest, the medical monitor should be contacted to discuss the subject's eligibility for continued participation in Trial 331-10-238.

A central laboratory designated by the sponsor will be used for all laboratory testing required during the trial. The central laboratory should be used for all laboratory testing whenever possible (including unscheduled and follow-up labs, if needed). In cases where an immediate result is required for a particular laboratory test, the sample should be divided and sent to both a local laboratory and the designated central laboratory. Urine will be collected and blood will be drawn from subjects at the scheduled visits designated in Table 3.6-1. Additional urine and blood samples may be collected for further evaluation of safety as warranted by the investigator's judgment. Screening/baseline laboratory assessments will be performed after a minimum 8-hour fast per the protocol instructions for the double-blind phase 3 trials. All subjects must be fasting for a minimum of 8 hours prior to the blood draw at Week 26/ET and should be fasting for a minimum of 8 hours prior to all other blood draws during the Treatment Phase, if possible. If a subject is not fasting at a visit other than Week 26/ET, the blood draw should still be performed and the status documented as nonfasting on the laboratory requisition sheet. The Week 26/ET blood draw must be rescheduled to accommodate the fasting requirement. Reports from the central laboratory should be filed with the source documents for each subject. The central laboratory will provide laboratory results to the sponsor electronically.

| Table 3.6.2.1-1 Safety Clinical Laboratory Tests | |
|---|---|
| Hematology: | Serum Chemistry: |
| WBC count with differential | ALP |
| RBC count | ALT or SGPT |
| Hematocrit | AST or SGOT |
| Hemoglobin | BUN |
| Platelet count | CPK |
| | Creatinine |
| <u>Urinalysis:</u> | LDH |
| pH | Total bilirubin |
| Specific gravity | Triglycerides |
| Protein | Cholesterol (total, LDL, and HDL) |
| Ketones | Calcium |
| Glucose | Chloride |
| Blood | Glucose |
| Microscopic exam (performed only if any part of | Insulin |
| the urinalysis is not negative) | Magnesium |
| | Bicarbonate |
| <u>Urine Drug Screens:</u> | Inorganic phosphorous |
| Amphetamines | Sodium |
| Barbiturates | Potassium |
| Benzodiazepines | Total protein |
| Cannabinoids | Uric acid |
| Cocaine | GGT |
| Marijuana | Prolactin |
| Methadone | Albumin |
| Opiates | |
| Phencyclidine | Additional Tests: |
| Propoxyphene | Urine pregnancy (WOCBP) <sup>a</sup> |
| Other: | TSH, with reflex to free T <sub>4</sub> if TSH is abnormal |
| Blood alcohol | PT, aPTT, and INR |
| Dioda diconor | HbA1c |
| A I D = -111:1 A I T CCDT = -1: | 4 |

ALP = alkaline phosphatase; ALT or SGPT = alanine transaminase; AST or SGOT = aspartate transaminase; BUN = blood urea nitrogen; CPK = creatine phosphokinase; GGT = gamma glutamyl transferase; HbA1c = glycosylated hemglobin; HDL = high density lipoprotein; LDH = lactic dehydrogenase; LDL = low density lipoprotein; RBC = red blood cell.

Any value outside the normal range will be flagged for the attention of the investigator who must indicate whether or not a flagged value is of clinical significance. If one or more values are questionable, the test(s) may be repeated. Follow-up unscheduled labs should be performed on clinically significant abnormalities. Unscheduled laboratory tests may be repeated at any time at the discretion of the investigator for appropriate medical care.

<sup>&</sup>lt;sup>a</sup> All positive urine pregnancy test results must be confirmed by a serum test. Subjects with a positive serum pregnancy test result at Screening/Baseline must not be enrolled and subjects with a positive serum pregnancy test result during the trial must discontinue treatment and be withdrawn from the trial.

To be eligible for Trial 331-10-238, subjects are not permitted to have laboratory values within the following exclusionary ranges:

- 1) Platelets  $\leq 75,000/\text{mm}^3$
- 2) Hemoglobin  $\leq 9 \text{ g/dL}$
- 3) Neutrophils, absolute  $\leq 1000/\text{mm}^3$
- 4) Aspartate transaminase (AST)  $\geq 2 \times$  upper limit of normal (ULN)
- 5) Alanine transaminase (ALT)  $\geq$  2 × ULN
- 6) Creatine phosphokinase (CPK)  $> 3 \times$  ULN, unless discussed with and approved by the medical monitor
- 7) Creatinine  $\geq 2 \text{ mg/dL}$
- 8) HbA1c  $\geq 7.0\%$
- 9) Abnormal free T<sub>4</sub>, unless discussed with and approved by the medical monitor. (Note: Free T<sub>4</sub> is measured only if result for TSH is abnormal.)

#### 3.6.2.2 Physical Examination and Vital Sign Assessments

## 3.6.2.2.1 Physical Examination

The complete physical examination at the last scheduled visit of the prior double-blind phase 3 trial will serve as the screening/baseline physical examination for the current protocol. A complete physical examination will consist of a review of the following body systems: HEENT, thorax, abdomen, urogenital, extremities, neurological, and skin and mucosae. Repeat measurement of height is not required during Trial 331-10-238 if a Screening/Baseline value is available from the prior double-blind phase 3 trial. Waist circumference will be measured at Screening/Baseline, Week 14, and Week 26/ET. The following procedures will aid in the standardization of these measurements:

- The subject should be minimally clothed (ie, lightweight clothing; no heavy overgarments).
- Waist circumference should be recorded before a subject's meal and at approximately the same time at each visit.
- Measurement will be accomplished by locating the upper hip bone and the top of the right iliac crest and placing a weighted measuring tape in a horizontal plane around the abdomen at the level of the crest. Before reading the tape measure, the assessor should assure that the tape is snug, but does not compress the skin, and is parallel to the floor. The measurement is to be made at the end of a normal exhalation.<sup>24</sup>

The principal investigator or his/her appointed designee is primarily responsible to perform the physical examination. If the appointed designee is to perform the physical examination, he/she must be permitted by local regulations and his/her name must be included on the FDA Form 1572. Whenever possible, the same individual should perform all physical examinations. Any condition present at the post-treatment physical examination that was not present at the screening/baseline examination should be documented as an AE and followed to a satisfactory conclusion.

# 3.6.2.2.2 Vital Signs

Vital sign measurements will include body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. The following guidelines will aid in the standardization of body weight measurements:

- The same scale should be used to weigh a given subject each time, if possible.
- Scales should be calibrated and reliable; scales should be at zero just prior to each subject's weigh-in session.
- A subject should void prior to being weighed and be minimally clothed (ie, no shoes or heavy overgarments).
- Weight should be recorded before a subject's meal and at approximately the same time at each visit.

Blood pressure and heart rate measurements will be made in the supine, sitting, and standing positions after the subject has been in each position for at least 3 minutes. The supine measurements will be performed first, followed by sitting, and finally standing. Vital signs scheduled at the same visit as blood samples are to be completed before blood is drawn.

Subjects with uncontrolled hypertension (Screening/Baseline DBP > 95 mmHg) or symptomatic hypotension are excluded from the trial as are subjects with orthostatic hypotension defined as a decrease of  $\geq$  30 mmHg in SBP and/or a decrease of  $\geq$  20 mmHg in DBP after at least 3 minutes standing compared to the previous supine blood pressure **OR** development of symptoms (see Table 3.4.3-1). In addition, subjects should be excluded if they have any other vital sign measurement at Screening/Baseline that, in the investigator's judgment, is medically significant in that it would impact the safety of the subject or the interpretation of the trial results. However, any abnormal screening/baseline vital sign result(s) considered to be clinically significant should be repeated to confirm the finding(s) before excluding the subject from the trial. Appendix 3 is included to assist investigators in their assessments of results that may be potentially

medically significant, depending on the subject's medical history and clinical presentation.

#### 3.6.2.3 ECG Assessments

Twelve-lead ECGs will be recorded at the visits specified in Table 3.6-1. ECG recordings will be obtained after the subject has been supine and at rest for at least 5 minutes. Additional 12-lead ECGs may be obtained at the investigator's discretion and should always be obtained in the event of an early termination. A central ECG service will be utilized for reading all ECGs in order to standardize interpretations for the safety analysis. In addition, ECG results will be evaluated at the investigational site to monitor safety during the trial. The principal investigator or qualified designee will review, sign, and date each ECG reading, noting whether or not any abnormal results are of clinical significance. The ECG will be repeated if any results are considered to be clinically significant.

As the results from the central reader will not be available at the Screening/Baseline visit, the subject will be enrolled into Trial 331-10-238 based on the local ECG results. A screening/baseline ECG finding of QTc corrected for heart rate by Fridericia's formula  $(QTcF) \ge 450$  msec is exclusionary (see Table 3.4.3-1). In addition, subjects should be excluded if they have any other abnormal ECG finding at Screening/Baseline that, in the investigator's judgment, is medically significant in that it would impact the safety of the subject or the interpretation of the trial results. However, any screening/baseline ECG with abnormal result(s) considered to be clinically significant should be repeated to confirm the finding(s) before excluding the subject from the trial. Appendix 5 is provided as a guide for determining potentially clinically relevant ECG abnormalities. If the results from the central reader, when available, indicate a screening/baseline  $QTcF \ge 450$  msec, the investigator must contact the medical monitor to discuss the subject's continued participation in the trial.

# 3.6.2.4 Other Safety Assessments

It is required that a trained and experienced clinician administer the safety assessments, including the EPS scales (SAS, AIMS, and BARS) and C-SSRS. The number of raters within each trial center should be kept to a minimum. All efforts will be made to ensure that the same clinician administers the scales for a given subject. Notations in the subject's trial records should substantiate the ratings. Training and materials for rating will be provided by Bracket.

# 3.6.2.4.1 Simpson Angus Scale (SAS)

The SAS<sup>25</sup> (Appendix 10) consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item will be rated on a 5-point scale, with a score of zero representing absence of symptoms, and a score of 4 representing a severe condition. The SAS Total Score is the sum of the scores for all 10 items.

Anticholinergics, propranolol, benzodiazepines, and non-benzodiazepine sleep aids are not permitted within 12 hours of scale administration (see Section 4). Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of the scale is not feasible, the SAS should still be administered and the use of the medication documented, including a notation of the drug name, dose, and time of administration on the electronic case report form (eCRF).

# 3.6.2.4.2 Abnormal Involuntary Movement Scale (AIMS)

The AIMS<sup>26</sup> assessment (Appendix 11) consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) will be observed unobtrusively while the subject is at rest (eg, in the waiting room), and the investigator will also make global judgments on the subject's dyskinesias (items 8 through 10). Each item will be rated on a 5-point scale, with a score of zero representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness, severe distress). For this scale, the subject is to be sitting on a hard, firm chair. In addition, the AIMS includes two yes/no questions that address the subject's dental status. Anticholinergics, propranolol, benzodiazepines, and non-benzodiazepine sleep aids are not permitted within 12 hours of scale administration (see Section 4). Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of the scale is not feasible, the AIMS should still be administered and the use of the medication documented, including a notation of the drug name, dose, and time of administration on the eCRF.

The AIMS Movement Rating Score is defined as the sum of items 1 through 7 (ie, items 1 through 4, facial and oral movements; items 5 and 6, extremity movements; and item 7, trunk movements).

# 3.6.2.4.3 Barnes Akathisia Rating Scale (BARS)

The BARS<sup>27</sup> (Appendix 12) consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the

subject, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items will be rated on a 4-point scale, with a score of zero representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation will be made on a 6-point scale, with zero representing absence of symptoms and a score of 5 representing severe akathisia. To complete this scale, subjects will be observed while they are seated and then standing for a minimum of 2 minutes in each position. Symptoms observed in other situations (eg, while engaged in neutral conversation or engaged in other activity) may also be rated. Subjective phenomena are to be elicited by direct questioning. Anticholinergics, propranolol, benzodiazepines, and non-benzodiazepine sleep aids are not permitted within 12 hours of scale administration (see Section 4). Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of the scale is not feasible, the BARS should still be administered and the use of the medication documented, including a notation of the drug name, dose, and time of administration on the eCRF.

The BARS Global Score is defined as the global clinical assessment of akathisia.

# 3.6.2.4.4 Suicidality

Suicidality will be monitored during the trial using the C-SSRS. Subjects completed the "Baseline/Screening" C-SSRS form at the beginning of the prior double-blind phase 3 trial; therefore, only the "Since Last Visit" C-SSRS form will be used in Trial 331-10-238. A copy of the "Since Last Visit" C-SSRS form is provided in Appendix 13.

#### 3.6.2.4.5 Sexual Function

The MSFQ<sup>28</sup> is a measure of a subject's self-reported sexual functioning. It consists of 5 items that are each rated as one of six defined grades of functioning (Appendix 14). The investigator or designated trial personnel should ensure that a subject completes this instrument completely and legibly.

# 3.6.3 Efficacy Assessments

It is required that appropriately trained and qualified individuals administer the CGI-S and CGI-I. The number of raters within each trial center should be kept to a minimum. All efforts will be made to ensure that the same clinician administers the scales for a given subject. Notations in the subject's trial records should substantiate the ratings. Training and materials for rating will be provided by Bracket.

# 3.6.3.1 Clinical Global Impression - Severity of Illness Scale (CGI-S)

The severity of illness for each subject will be rated using the CGI-S. To perform this assessment, the rater or investigator will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices include: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. A sample of the CGI-S is provided in Appendix 6.

# 3.6.3.2 Clinical Global Impression - Improvement Scale (CGI-I)

The efficacy of trial treatment will be rated for each subject using the CGI-I.<sup>26</sup> The rater or investigator will rate the subject's total improvement whether or not it is due entirely to drug treatment. All responses will be compared to the subject's condition at Screening/Baseline (ie, last scheduled visit of the prior double-blind phase 3 trial). Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. A sample of the CGI-I is provided in Appendix 7.

# 3.6.3.3 Subject Assessment Recording

# 3.6.3.3.1 Sheehan Disability Scale (SDS)

The SDS  $^{29,30}$  is a self-rated instrument used to measure the effect of the subject's symptoms on work/school, social life, and family/home responsibilities (Appendix 8). The SDS is a visual analogue scale that uses spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the three domains. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0 = not at all, to 10 = extremely. Scores of 5 and above are associated with significant functional impairment. In addition to the visual scale, the SDS includes two questions related to productivity losses due to the psychiatric symptoms and impairment.

# 3.6.3.3.2 Inventory of Depressive Symptomatology (Self-Report)

The IDS-SR<sup>31</sup> is a 30-item self-report measure used to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of MDD (Appendix 9). The investigator or designated trial personnel should ensure that a subject completes this instrument completely and legibly.

# 3.6.3.3.3 Resource Utilization Form (RUF)

The RUF is a self-report tool designed to collect information regarding the extent of medical care sought by subjects while participating in the trial (Appendix 15). The number of hospitalizations and days of hospitalization within the past 12 months will be collected on the Baseline Form at Screening/Baseline, including any hospitalizations that may have occurred during the subject's participation in the prior double-blind phase 3 trial. The number of visits to various practitioners for mental health and other reasons within the 3 months prior to Screening/Baseline (excluding any visits from the prior double-blind phase 3 trial) will be collected on the Baseline Form and the number of such visits occurring during the trial (excluding visits related to the trial) will be collected on the Follow-up Form at Week 26/ET.

#### 3.6.4 End of Trial

The End of Trial Date is defined as the last Date of Contact or the Date of Final Contact Attempt from the Post-treatment Follow-up eCRF page for the last subject completing or withdrawing from the trial.

## 3.7 Stopping Rules, Withdrawal Criteria and Procedures

# 3.7.1 Entire Trial or Treatment Arm(s)

If the sponsor terminates or suspends the trial for safety or unanticipated other reasons, prompt notification will be given to investigators, IRBs/IECs, and regulatory authorities in accordance with regulatory requirements.

#### 3.7.2 Individual Center

A particular center may be terminated from the trial at the discretion of the investigator, sponsor, or IRB, eg, for non-enrollment of subjects or noncompliance with the protocol. The investigator will notify the sponsor promptly if the trial is terminated by the investigator or the IRB/EC at the site.

#### 3.7.3 Individual Subject

If a subject discontinues from the trial prematurely, the reason must be fully evaluated and recorded appropriately in source documents and the eCRF. If the subject is being withdrawn because of an AE, that AE should be indicated as the reason for withdrawal. All subjects have the right to withdraw at any point during treatment without prejudice. The investigator can discontinue a subject's participation in the trial at any time if

medically necessary. In addition, subjects meeting the following criteria must be withdrawn from the trial:

- a) occurrence of any AE, intercurrent illness or abnormality in a laboratory assessment which, in the opinion of the investigator, warrants the subject's permanent withdrawal from the trial;
- b) treatment with a prohibited concomitant medication other than the use of appropriate medications for the treatment of AEs under direction of the investigator;
- c) subject noncompliance, defined as refusal or inability to adhere to the trial schedule or procedures (see Section 3.11, Subject Compliance);
- d) at the request of the subject, investigator, sponsor or designee, or regulatory authority;
- e) subject becomes pregnant;
- f) subject cannot tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day), the minimum protocol-defined therapeutic dose of ADT (see Table 3.2.1.2-1), or requires a different ADT; or
- g) subject is lost to follow-up.

The investigator will notify the sponsor promptly when a subject is withdrawn. Subjects withdrawn prior to Week 26 must complete the Week 26/ET evaluations at the time of withdrawal. In addition, all subjects who withdraw prematurely from the trial will be assessed 30 (+ 2) days after the last dose of IMP for evaluation of safety. This assessment can be accomplished via telephone contact or clinic visit at the investigator's discretion. Withdrawn subjects will not be replaced.

#### 3.8 Screen Failures

A screen failure subject is one from whom informed consent is obtained and is documented in writing (ie, subject signs an ICF), but who is not started on treatment, whether through randomization or open assignment. For the purposes of Trial 331-10-238, treatment begins with the first dose of open-label brexpiprazole in the Treatment Phase. Subjects who do not qualify for Trial 331-10-238 at the last scheduled visit of the prior double-blind phase 3 trial may not be rescreened.

#### 3.9 Definition of Completed Subjects

The treatment period is defined as the time period during which subjects are evaluated for primary and/or secondary objectives of the trial irrespective of whether or not the subject actually consumed all doses of IMP. Subjects who are evaluated at the last scheduled

visit during the treatment period will be defined as trial completers. For purposes of this trial, subjects who complete the Week 26 visit will be defined as completers. Protocol-specified post-treatment follow-up contacts will not qualify as the "last scheduled visit." Subjects who are not completers are defined as those who "discontinued the trial."

## 3.10 Definition of Lost to Follow-up

Subjects who cannot be contacted on or before the Week 26 visit during the treatment period and who do not have a known reason for discontinuation (eg, withdrew consent or AE) will be classified as "lost to follow-up" as the reason for discontinuation. The site will make three attempts to contact the subject by telephone and in the event the site is unable to reach the subject by telephone, the site will attempt to contact the subject via certified mail or an alternative similar method where appropriate.

## 3.11 Subject Compliance

Responsible trial personnel will dispense the IMP (ie, brexpiprazole and ADTs). Accountability and compliance verification should be documented in the subject's trial records. Subjects must be counseled on the importance of taking the IMP as directed at all trial visits. If poor compliance continues (eg, multiple missed doses resulting in less than 80% overall compliance at any point in the trial), discontinuation of the subject from the trial should be considered. Subjects who habitually miss visits or habitually attend visits outside of the protocol-defined visit window are also noncompliant and should be considered for discontinuation. The medical monitor should be contacted if the investigator is uncertain whether a subject's lack of compliance merits discontinuation from the trial.

#### 3.12 Protocol Deviations

This trial is intended to be conducted as described in this protocol. In the event of a significant deviation from the protocol due to an emergency, accident, or mistake (eg, violation of informed consent process, IMP dispensing or subject dosing error, subject enrolled in violation of eligibility criteria or concomitant medication criteria), the investigator or designee will contact the sponsor's designee (medical monitor) at the earliest possible time by telephone. Investigator and sponsor (or sponsor's designee) will come as quickly as possible to a joint decision regarding the subject's continuation in the trial. This decision will be documented by the investigator and the designated medical monitor, and reviewed by the site monitor.

#### 4 Restrictions

#### 4.1 Prohibited Medications

Concomitant medications taken by subjects who are rolling over into Trial 331-10-238 from a prior double-blind phase 3 trials should be reviewed for the prohibited medications listed in Table 4.1-1. Any subject taking a prohibited concomitant medication should not be enrolled in Trial 331-10-238.

## **Table 4.1-1 List of Medications Prohibited During the Trial** 1. All psychotropic agents including, but not limited to, the following: a) Antipsychotics, including depot or long-acting injectable formulations b) Anticonvulsants c) Antidepressants other than the ADTs listed in Table 3.2.1.2-1 d) Mood stabilizers (ie, lithium) e) Benzodiazepines, except when used to manage treatment emergent AEs such as agitation and anxietva f) Hypnotics, including ramelteon and other non-benzodiazepine sleep aids, except for specific medications when used to manage treatment-emergent AEs related to insomnia g) Stimulants h) Opioid analgesics, unless permission is obtained from the medical monitor. Permission for opioid use may be considered for a documented and clinically appropriate indication (eg, episodic pain condition, tooth extraction) if prescribed at a medically appropriate dose and frequency. Nutritional supplements and non-prescription herbal preparations with CNS effects (eg, St. John's Wort, omega-3 fatty acids, kava extracts, GABA supplements, etc) Investigational agents CYP2D6 inhibitors or CYP3A4 inhibitors and inducers. Selected CYP2D6 inhibitors <sup>c</sup> are: celecoxib, hydroxyzine, chloroquine, methadone, chloroheniramine, moclobemide, clemastine, clomipramine, pyrilamine, diphenhydramine, quinidine, terbinafine, halofantrine, tripelennamine. Selected CYP3A4 inhibitors are: amiodarone, fluvoxamine, amprenavir, indinavir, aprepitant, itraconazole, chloramphenicol, ketoconazole, cimetidine, nefazodone, clarithromycin, nelfinavir, clotrimazole (if used orally), quinupristin/dalfopristin, delavirdine, ritonavir, diltiazem, saquinavir, erythromycin, troleandomycin, fluconazole, verapamil. Selected CYP3A4 inducers are: carbamazepine, oxcarbazepine, phenytoin, dexamethasone, primidone, efavirenz, rifampin, nevirapine, St. John's Wort, phenobarbitol, troglitazone. The medical monitor should be consulted for any questions regarding the potential for pharmacokinetic interactions with concomitant medications used by subjects during the trial. Barbiturates, except for the treatment of migraine headaches, provided that in the opinion of the

GABA = gamma-aminobutyric acid.

investigator the dosing is medically appropriate.

Administration of specific oral benzodiazepines is permitted for the short-term management of treatment emergent AEs such as anxiety and agitation up to a maximum of 6 mg/day lorazepam (or equivalent) in divided doses. Short-acting benzodiazepines are to be used whenever possible. In countries where no short-acting benzodiazepines are commercially available, use of oral diazepam or clonazepam may be acceptable if prior authorization is obtained from the medical monitor. The following guide should be used to determine approximate lorazepam equivalents: 1 mg lorazepam = 15 mg oxazepam = 0.5 mg alprazolam = 5 mg diazepam = 0.5 mg clonazepam. The prescribed benzodiazepine should be discontinued as soon as the AE for which it was initiated subsides, as per

the investigator's discretion to avoid any withdrawal effects. Benzodiazepines must not be administered within 12 hours prior to scheduled efficacy and safety assessments, including EPS scales. Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of efficacy and safety scales is not feasible, the scales should still be administered and the use of benzodiazepine documented, including a notation of the drug name, dose, and time of administration on the eCRF.

Non-benzodiazepine sleep aids (ie, zolpidem, zaleplon, zopiclone, and eszopiclone only) are permitted for the treatment of insomnia, but not on the same day as administration of a benzodiazepine, regardless of indication. For the non-benzodiazepine sleep aids, sites should only utilize one of the listed medications that are approved for this indication in their respective countries and the country-specific prescribing information is to be used to determine the maximum allowable daily dose for the treatment of insomnia. Non-benzodiazepine sleep aids must not be administered within 12 hours prior to scheduled efficacy and safety assessments, including EPS scales. Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of efficacy and safety scales is not feasible, the scales should still be administered and the use of the sleep aid documented, including a notation of the drug name, dose, and time of administration on the eCRF.

Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs that are also CYP2D6 inhibitors. In order to limit the potential higher exposure of brexpiprazole when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine (see Section 4.2.1).

#### 4.2 Other Restrictions

# 4.2.1 Restricted Therapies and Precautions

The subject's best medical interests should guide the investigator in the management of conditions that are pre-existing or that develop during the trial (intercurrent illness or AEs). The investigator should examine the acceptability of all concomitant medications not explicitly prohibited. In order to ensure that appropriate concomitant therapy is administered, it is essential that subjects be instructed not to take any medications (either self-administered non-prescription drugs or prescription therapy prescribed by another physician) without prior consultation with the investigator. In particular, the investigator should caution the subject about concomitant use of the following during the trial:

- Non-steroidal anti-inflammatory drugs, aspirin, or other drugs that interfere with coagulation since the combined use of psychotropic drugs that interfere with serotonin reuptake and these agents has been associated with an increased risk of upper gastrointestinal bleeding.<sup>32</sup>
- Triptans (eg, sumatriptan, naratriptan, almotriptan, frovatriptan, rizatriptan, eletriptan, and zolmitriptan), linezolid, and methylene blue since there have been rare post-marketing reports of serotonin syndrome or serotonin syndrome-like reactions (eg, mental status changes, hyperreflexia, autonomic effects, lack of coordination, and diarrhea) following the concomitant use of SSRIs or SNRIs and these drugs. 33,34,35

Electroconvulsive therapy was prohibited during the prior double-blind phase 3 trials and is also prohibited for the duration of Trial 331-10-238. Transcranial magnetic stimulation is also prohibited. In addition, subjects may not undergo implantation of a device for vagus nerve stimulation or deep brain stimulation during the trial.

Use of intramuscular benzodiazepines and continual use of oral benzodiazepines are prohibited throughout the trial. However, administration of specific oral benzodiazepines is permitted for the short-term management of treatment emergent AEs such as anxiety and agitation up to a maximum of 6 mg/day lorazepam (or equivalent) in divided doses. Short-acting benzodiazepines are to be used whenever possible. In countries where no short-acting benzodiazepines are commercially available, use of oral diazepam or clonazepam may be acceptable if prior authorization is obtained from the medical monitor. The following guide should be used to determine approximate lorazepam equivalents: 1 mg lorazepam = 15 mg oxazepam = 0.5 mg alprazolam = 5 mg diazepam = 0.5 mg clonazepam. The prescribed benzodiazepine should be discontinued as soon as the AE for which it was initiated subsides, as per the investigator's discretion to avoid any withdrawal effects.

Non-benzodiazepine sleep aids (ie, zolpidem, zaleplon, zopiclone, and eszopiclone only) are permitted for the treatment of insomnia, but not on the same day as administration of a benzodiazepine, regardless of indication. For the non-benzodiazepine sleep aids, sites should only utilize one of the listed medications that are approved for this indication in their respective countries and the country-specific prescribing information is to be used to determine the maximum allowable daily dose for the treatment of insomnia.

Anticholinergics are permitted for the treatment of EPS up to a maximum of 4 mg/day benztropine or its equivalent and propranolol is permitted for akathisia or tremor up to a maximum of 20 mg three times daily (total of 60 mg/day). Sites should only utilize medications that are approved for these indications in their respective countries.

Benzodiazepines, non-benzodiazepine sleep aids, anticholinergics, and propranolol must not be administered within 12 hours prior to scheduled efficacy and safety assessments, including EPS scales. Investigators are encouraged to delay scale administration until 12 hours have elapsed, if at all possible. However, if delaying administration of efficacy and safety scales is not feasible, the scales should still be administered and the use of the medication documented, including a notation of the drug name, dose, and time of administration on the eCRF.

Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs in this trial; however, they are also CYP2D6 inhibitors. Data from Trial 331-08-207 and Trial 331-08-208 indicate that coadministration of CYP2D6 inhibitors with brexpiprazole can cause potentially higher plasma concentrations of brexpiprazole (up to 2-fold). In order to limit the potential higher exposure of brexpiprazole when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine. The investigator should consider the potential for higher brexpiprazole plasma concentrations when adjusting the dose of brexpiprazole for subjects who are receiving fluoxetine, paroxetine CR, or duloxetine as the assigned ADT.

All trial personnel should be familiar with the content of the Investigator Brochure for brexpiprazole in order to manage the subject's condition adequately and select appropriate concomitant medications, if needed.

# 4.2.2 Non-therapy Precautions and Restrictions

#### 4.2.2.1 Precautions

Subjects should not undergo any elective medical procedure without prior consultation with the investigator. An elective procedure (minor surgery, dental surgery, orthopedic surgery, etc) that might require hospitalization or general anesthesia should be deferred until after the trial whenever clinically appropriate.

## 4.2.2.2 Restrictions

Subjects may only receive psychotherapy (eg, individual, group, marriage, or family therapy) if they initiated the therapy at least 42 days before enrollment in the prior double-blind phase 3 trial, participated in the therapy regularly during the prior double-blind phase 3 trial, and commit to maintain their participation during the course of Trial 331-10-238, or unless permission is obtained from the medical monitor.

Consumption of grapefruit, grapefruit products, Seville oranges, or Seville orange products within 72 hours prior to dosing and during the trial is prohibited. Subjects will be instructed to refrain from drinking alcoholic beverages or using illicit drugs during participation in the trial. The investigator may request a blood or urine drug screen at any time during the trial if there is a suspicion of illicit drug use.

# 5 Reporting of Adverse Events

#### 5.1 Definitions

An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

A suspected adverse reaction means any AE for which there is a reasonable possibility that the drug caused the AE. For the purpose of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the AE. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any AE caused by a drug.

A serious adverse event (SAE) includes any event that results in any of the following outcomes:

- death
- life-threatening, ie, the subject was, in the opinion of the investigator or the sponsor, at <u>immediate</u> risk of death from the event as it occurred. It does not include an event that, had it occurred in a more severe form, might have caused death.
- persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- requires in-patient hospitalization or prolongs an existing hospitalization NOTE: A pre-scheduled hospitalization is not considered an SAE; however, SAE forms must be completed for all other hospitalizations, including hospitalization for psychiatric reasons. Psychosocial hospitalizations (eg, homelessness or need for shelter that is unrelated to the subject's underlying psychiatric condition) should not be reported as SAEs.
- congenital anomaly/birth defect
- other medically significant events that, based upon appropriate medical
  judgment, may jeopardize the subject and may require medical or surgical
  intervention to prevent one of the outcomes listed above, eg, allergic
  bronchospasm requiring intensive treatment in an emergency room or home,
  blood dyscrasias or convulsions that do not result in hospitalization, or the
  development of drug dependency or drug abuse.

Non-serious adverse events are all AEs that do not meet the criteria for a "serious" AE.

If a subject is experiencing an extrapyramidal symptom, the specific extrapyramidal symptom must be indicated on the AE page of the eCRF. Examples of AEs that are considered extrapyramidal symptoms include, but are not limited to: generalized rigidity,

hyperkinesia, dyskinesia, bradykinesia, akinesia, dystonia, hypertonia, akathisia, tremor, flexed posture, involuntary muscle contractions, athetosis, and chorea. If a subject is experiencing two or more of these symptoms, whether or not treatment with an anticholinergic is required, this is considered as extrapyramidal syndrome and must be entered as "extrapyramidal syndrome" on the AE page of the eCRF instead of the individual symptoms. Permitted treatments for EPS are described in Section 4.2.1.

## <u>Immediately Reportable Event (IRE):</u>

- Any SAE
- Any AE that necessitates discontinuation of IMP.
- Potential Hy's Law cases (any increase of AST or ALT  $\geq 3$  times the upper normal limit with an increase in total bilirubin  $\geq 2$  times the upper normal limit).
- Pregnancies are also defined as IREs. Although normal pregnancy is not an AE, it will mandate IMP discontinuation and must be reported on an IRE form to INC Research. Pregnancy will only be documented on the AE eCRF if there is an abnormality or complication.

Clinical Laboratory Changes: It is the investigator's responsibility to review the results of all laboratory tests as they become available. This review will be documented by the investigator's dated signature on the laboratory report. For each abnormal laboratory test result, the investigator needs to ascertain if this is an abnormal (ie, clinically significant) change from baseline for that individual subject. (This determination, however, does not necessarily need to be made the first time an abnormal value is observed. The investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory tests). If this laboratory value is determined by the investigator to be an abnormal change from baseline for that subject, this is considered an AE.

<u>Severity</u>: Adverse events will be graded on a 3-point scale and reported as indicated on the eCRF. The intensity of an adverse experience is defined as follows:

**1 = Mild:** Discomfort noticed, but no disruption to daily activity.

**2 = Moderate:** Discomfort sufficient to reduce or affect normal daily activity.

**3 = Severe:** Inability to work or perform normal daily activity.

<u>IMP Causality:</u> Assessment of causal relationship of an AE to the use of the IMP is defined as follows:

**Related**: There is a reasonable possibility of a causal relationship.

Possibly related: There is a reasonable causal relationship between the IMP and the

AE. Dechallenge is lacking or unclear.

Unlikely related: There is a temporal relationship to IMP administration, but there is

not a reasonable causal relationship between the IMP and the AE.

**Not Related**: There is no temporal or reasonable relationship to the IMP

administration.

Investigators will assess IMP causality based on brexpiprazole.

# 5.2 Eliciting and Reporting Adverse Events

The investigator will periodically assess subjects for the occurrence of AEs. In order to avoid bias in eliciting AEs, subjects should be asked the following non-leading question: "How have you felt since your last visit?" All AEs (serious and non-serious) reported by the subject must be recorded on the source documents and on the eCRFs provided by the sponsor or designee.

Note: Normal pregnancy is not an AE and should not be recorded on the eCRFs; guidelines outlined in Section 5.5 should be followed for pregnancy reporting.

In addition, INC Research (Appendix 2) must be notified immediately by telephone or fax of any <u>immediately reportable events</u> according to the procedure outlined below in Section 5.3. Special attention should be paid to recording hospitalization and concomitant medications.

# 5.3 Immediately Reportable Events (IRE)

The investigator must immediately (ie, within 24 hours) report any <u>serious adverse event</u>, <u>potential Hy's law cases</u>, <u>or confirmed pregnancy</u> by telephone or by fax to INC Research as outlined in <u>Appendix 2</u> after either the investigator or site personnel become aware of the event. An Immediately Reportable Event (IRE) form must be completed and transmitted per the instructions in the Operations Manual. (Please note that the IRE form is NOT the AE eCRF.)

<u>Non-serious events</u> that require <u>discontinuation</u> of IMP (including laboratory abnormalities) should be reported to INC Research within 3 working days. The IRE form must be completed and sent by fax or overnight courier to INC Research.

Subjects experiencing SAEs should be followed clinically until their health has returned to baseline status or until all parameters have returned to normal, or have otherwise been explained. It is expected that the investigator will provide or arrange appropriate supportive care for the subject.

# 5.4 Potential Hy's Law Cases

For a subject that experiences an elevation in AST or ALT that is  $\geq 3$  times the upper normal limit, a total bilirubin level should also be evaluated. If the total bilirubin is  $\geq 2$  times the upper normal limit, confirmatory repeat laboratory samples should be drawn within 48 to 72 hours of the initial draw. If these values are confirmed, trial personnel will complete an IRE form with all values listed and also report the event as an AE on the eCRFs. Please note: If the subject was enrolled into the trial with non-exclusionary elevated transaminase levels at baseline, please discuss any potential druginduced liver injury events with the Medical Monitor.

# 5.5 Pregnancy

WOCBP and men who are sexually active must use an effective method of birth control during the course of the trial and for at least 30 days after the last dose in a manner such that risk of failure is minimized. Unless the subject is sterile (ie, women who have had an oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months; or men who have had orchidectomy) or remains abstinent, two of the following precautions must be used: vasectomy or tubal ligation (subject and partner), vaginal diaphragm, intrauterine device, birth control pills, birth control depot injection, birth control implant, condom or sponge with spermicide. Any single method of birth control, including vasectomy and tubal ligation, may fail, leading to pregnancy.

Before enrolling WOCBP in this clinical trial, investigators must review guidelines about trial participation for WOCBP. The topics should generally include:

- General information
- Informed consent form
- Pregnancy prevention information
- Drug interactions with hormonal contraceptives
- Contraceptives in current use
- Guidelines for the follow-up of a reported pregnancy

Prior to trial enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. The subject must sign an ICF stating that the above-mentioned risk factors and the consequences were discussed with her.

During the trial, all WOCBP should be instructed to contact the investigator immediately if they suspect they might be pregnant (eg, missed or late menstrual cycle).

If a subject or investigator suspects that the subject may be pregnant prior to IMP administration, the IMP administration must be withheld until the results of serum pregnancy tests are available. If the pregnancy is confirmed, the subject must not receive the IMP and must not be enrolled in the trial. If pregnancy is suspected while the subject is taking IMP, the IMP must be withheld immediately (if reasonable, taking into consideration any potential withdrawal risks) until the result of the pregnancy is known. If pregnancy is confirmed, the IMP will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for subject safety) and the subject withdrawn from the trial. Exceptions to trial discontinuation may be considered for life-threatening conditions only after consultations with the Drug Safety and Pharmacovigilance Department of INC Research (see Appendix 2 for contact information).

The investigator must immediately notify INC Research of any pregnancy associated with IMP exposure, including at least 30 days after the last dose for female subjects and the female partner(s) of a male subject and record the event on the IRE form and forward it to INC Research. INC Research will forward Pregnancy Surveillance Form(s) for monitoring the outcome of the pregnancy.

Protocol required procedures for trial discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (eg, x-ray studies). Other appropriate pregnancy follow-up procedures should be considered if indicated. In addition, the investigator must report to INC Research, on appropriate Pregnancy Surveillance form(s), follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants will be followed for a minimum of six months.

# 5.6 Follow-up of Adverse Events

For this trial, information on AEs will be followed for up to 30 (+2) days after the last dose of IMP has been administered.

#### 5.6.1 Follow-up of Non-serious Adverse Events

Non-serious AEs that are identified on the last scheduled contact must be recorded on the AE eCRF with the current status noted. All non-serious events that are ongoing at this time will be recorded as ongoing on the eCRF.

# 5.6.2 Follow-up of Post Trial Serious Adverse Events

Serious adverse events that are **identified on the last scheduled contact** must be recorded on the AE eCRF page and reported to INC Research according to the reporting procedures outlined in Section 5.3. This may include **unresolved previously reported** SAEs, or **new SAEs.** The investigator will follow SAEs until the events are resolved, or the subject is lost to follow-up. Resolution means the subject has returned to the baseline state of health, or the investigator does not expect any further improvement or worsening of the subject's condition. The investigator will continue to report any significant follow-up information to INC Research up to the point the event has been resolved.

This trial requires that subjects be actively monitored for SAEs up to 30 (+ 2) days after discharge from the trial.

# 5.6.3 Follow-up and Reporting of Serious Adverse Events Occurring after Last Scheduled Contact

Any new SAEs reported by the subject to the investigator that occur **after the last scheduled contact**, and are determined by the investigator to be reasonably associated with the use of the IMP, should be reported to INC Research. This may include SAEs that are captured on follow-up visit or telephone contact or at any other time point after the defined trial period (ie, up to last scheduled contact). The investigator should follow related SAEs identified after the last scheduled contact until the events are resolved, or the subject is lost to follow-up. The investigator should continue to report any significant follow-up information to INC Research up to the point the event has been resolved.

# 6 Pharmacokinetic Analysis

Not Applicable

# 7 Statistical Analysis

# 7.1 Primary and Secondary Outcome Variable Analysis

# 7.1.1 Data Sets for Analysis

The following analysis samples are defined for this trial:

Enrolled Sample: comprises all subjects who sign an ICF for the trial.

Safety Sample: comprises those subjects who receive at least one dose of open-label brexpiprazole as adjunctive therapy to one of the allowed ADTs.

Efficacy Sample: comprises those subjects in the Safety Sample who have at least one postbaseline efficacy evaluation of CGI-S.

The Safety Sample will be used for all baseline and safety summaries.

The Efficacy Sample will be used for the CGI-S summaries.

The observed cases (OC) dataset will consist of the actual observations recorded at each visit and will be used to present summaries per trial week.

The last-observation-carried-forward (LOCF) data set will include data recorded at a given visit in the Treatment Phase or, if no observation is recorded at that visit, data carried forward from the previous visit in the Treatment Phase. Data collected prior to or on the first day of Treatment Phase dosing will not be carried forward or averaged with Treatment Phase data to impute missing values for the LOCF data set.

# 7.1.2 Handling of Missing Data

In order to assess sensitivity of results due to missing data, two types of analyses will be performed for analyses by visit: LOCF and OC. The LOCF and OC data sets are defined in Section 7.1.1. The OC data set will be used for analyses at each visit and the LOCF data set will be used for the last visit analyses.

# 7.1.3 Primary Outcome Analysis

The primary safety analysis is the frequency and severity of AEs (see Section 7.4.1).

#### 7.1.4 Secondary Outcome Analysis

Secondary efficacy endpoints are as follows:

- 1) Change from baseline in CGI-S score, by trial week and at the last visit;
- 2) Mean CGI-I score, by trial week and at the last visit;
- 3) Change from baseline in SDS score, by trial week and at the last visit;
- 4) Change from baseline in IDS-SR Total Score, by trial week and at the last visit.

Descriptive statistics will be provided for each endpoint. The analysis will be carried out on the Efficacy Sample. Descriptive statistics will be summarized at each trial visit using the OC data set and at the last visit using the LOCF data set.

#### 7.2 Sample Size

The sample size is not based on statistical power considerations. The trial population will be derived from eligible subjects from the prior double-blind phase 3 brexpiprazole MDD
trials. Therefore, the number of eligible subjects will be limited by the number of subjects enrolled into these protocols. Based on the projected enrollment estimates for the prior double-blind phase 3 trials, up to approximately 3,000 subjects may enroll into Trial 331-10-238.

### 7.3 Analysis of Demographic and Baseline Characteristics

Baseline demographic characteristics including age, race, ethnicity, gender, weight, height, and BMI will be summarized by descriptive statistics (frequency, mean, median, standard deviation, maximum, minimum, and percentage when applicable).

### 7.4 Safety Analyses

Standard safety variables to be analyzed include AEs, clinical laboratory tests, vital signs, ECGs, body weight, waist circumference, and BMI. In addition, data from the following safety scales will be evaluated: SAS, AIMS, BARS, C-SSRS, and MSFQ. Analyses regarding safety and tolerability will be conducted based on the Safety Sample, which is defined in Section 7.1.1. In general, baseline measurements of safety variables are defined as their last measurements prior to the first dose of open-label brexpiprazole.

### 7.4.1 Adverse Events

All AEs will be coded by system organ class and Medical Dictionary for Regulatory Activities (MedDRA) preferred term. The incidence of the following events will be summarized:

- a) TEAEs by severity
- b) Potentially drug-related TEAEs
- c) TEAEs with an outcome of death
- d) Serious TEAEs
- e) Discontinuations due to TEAEs

### 7.4.2 Clinical Laboratory Data

Summary statistics for changes from baseline in the routine clinical laboratory measurements, prolactin concentrations, coagulation parameters (PT, aPTT, and INR), HbA1c, and TSH will be provided. In addition, potentially clinically significant results in laboratory tests identified using prospectively defined criteria will be summarized.

### 7.4.3 Physical Examination and Vital Signs Data

By-patient listings will be provided for physical examination. Summary statistics for changes from baseline in vital signs will be provided. Potentially clinically significant results in vital signs will also be summarized.

### 7.4.4 ECG Data

Mean change from baseline and incidence of clinically significant changes will be calculated for ECG parameters.

For the analysis of QT and QTc, data from three consecutive complexes (representing three consecutive heart beats) will be measured to determine average values. The following QT corrections will be used for reporting purposes in the clinical study report:

- 1) QTcB is the length of the QT interval corrected for heart rate by the Bazett formula: QTcB=QT/(RR)<sup>0.5</sup>
- 2) QTcF is the length of the QT interval corrected for heart rate by the Fridericia formula: QTcF=QT/(RR)<sup>0.33</sup>
- 3) QTcN is the length of the QT interval corrected for heart rate by the FDA Neuropharm Division formula: QTcN=QT/(RR)<sup>0.37</sup>

### 7.4.5 Other Safety Data

Descriptive statistics will be provided for the SAS, AIMS, BARS, and MSFQ scales. Change from baseline in body weight will be summarized by descriptive statistics, as well as incidence of clinically significant changes in body weight. Descriptive statistics will also be provided for change from baseline in waist circumference and BMI. Descriptive statistics will be summarized at each visit using the OC data set and at the last visit using the LOCF data set.

Suicidality monitored during the trial using the C-SSRS will be summarized as number and percentage of subjects reporting any suicidal behavior, ideation, behavior by type (4 types), ideation by type (5 types), and treatment-emergent suicidal behavior and ideation.

### 7.5 Other Outcomes

The percentage of subjects hospitalized for exacerbation of symptoms (including emergency department visits) will be tabulated as a measure of healthcare resource

utilization. The frequency of outpatient visits to various healthcare providers (eg, primary care physician, psychiatrists, other mental health practitioners, etc.) not required per the protocol will also be examined.

### 8 Trial Drug Management

### 8.1 Packaging and Labeling

Trial drugs will be provided to the investigator(s) by the sponsor (or designated agent). The IMP will consist of open-label brexpiprazole and open-label ADTs. Open-label brexpiprazole will be supplied as 0.5, 1, 2, and 3-mg tablets packaged in weekly blister cards, each containing sufficient tablets for 7 (+ 2 days). Blister cards will contain single tablet strengths (ie, brexpiprazole 0.5, 1, 2, or 3 mg/day) and subjects will take 1 tablet daily. When accessed by the site, the IVRS or IWRS will assign a specific blister card number to be dispensed to a subject. New weekly blister cards will be dispensed at each scheduled visit and at unscheduled visits if the dose of brexpiprazole is changed.

Each blister card used in the trial will be given an identifying number and will be labeled to clearly disclose the blister card number, Subject ID (to be filled in by the site staff/investigator), subject's initials or other unique identifier, name of the investigator (to be filled in by the site staff/investigator), site number (to be filled in by the site staff/investigator), subject's initials (to be filled in by the site staff/investigator), date dispensed (to be filled in by the site staff/investigator), compound ID, protocol number, the sponsor's name and address, instructions for use, route of administration, and appropriate precautionary statements. Once a blister card has been assigned to a subject via the IVRS or IWRS, it cannot be dispensed to another subject.

ADTs will be supplied as bulk drug in commercial packaging (eg, bottles) with an ancillary trial-specific label that will be positioned such that it will not obscure the original commercial label. The sponsor reserves the right to use a generic equivalent, should any marketed antidepressant become unavailable during the course of the trial. Each ADT bottle used in the trial will be labeled to clearly disclose the bottle number, Subject ID, subject's initials, protocol number, ADT drug name, the sponsor's name and address, instructions for use, route of administration, and appropriate precautionary statements. Once an ADT bottle has been assigned to a subject via the IVRS or IWRS, it cannot be dispensed to another subject. The amount of open-label ADT dispensed to a subject at each visit will be contingent upon the prescribed daily dose of ADT as well as the duration between trial visits. Subjects must remain on the same ADT for the duration

of the trial (ie, Screening/Baseline through Week 26/ET). Any subject who cannot tolerate the minimum protocol-defined therapeutic dose of ADT (see Table 3.2.1.2-1) or who is required to change from one ADT to another must be withdrawn from the trial.

### 8.2 Storage

Trial drugs will be stored in a securely locked cabinet or enclosure. Access will be limited to the investigators and their designees. Neither investigators nor any designees may provide trial drugs to any subject not participating in this protocol.

Brexpiprazole should be stored according to the storage conditions indicated on the clinical label. The open-label ADTs should be stored as per the individual manufacturers' label recommendations on the package insert or the ADT clinical label. The clinical site staff will maintain a temperature log in the drug storage area recording the temperature at least once each working day.

### 8.3 Accountability

The investigator, or designee, must maintain an inventory record of trial drugs (including brexpiprazole and ADTs) received, dispensed, administered, and returned.

### 8.4 Returns and Destruction

Upon completion or termination of the trial, all unused and/or partially used IMP (including brexpiprazole and ADTs) must be returned to Otsuka Pharmaceutical Development & Commercialization, Inc. (OPDC) (or a designated contractor).

All IMP returned to OPDC (or the designated contractor) must be accompanied by the appropriate documentation and be clearly identified by protocol number and trial site number. Returned supplies should be in the original containers (eg, blister cards and ADT commercial packaging). The assigned trial monitor will facilitate the return of unused and/or partially used IMP.

### 8.5 Reporting of Product Quality Complaints

A Product Quality Complaint (PQC) is any written, electronic, or verbal communication by a healthcare professional, consumer, subject, medical representative, Competent Authority, regulatory agency, partner, affiliate or other third party that alleges deficiencies or dissatisfaction related to identity, quality, labeling, packaging, reliability, safety, durability, tampering, counterfeiting, theft, effectiveness or performance of a drug product or medical device after it is released for distribution. Examples include, but are not limited to, communications involving:

- Failure/malfunction of a product to meet any of its specifications
- Incorrect or missing labeling
- Packaging issues (eg, damaged, dirty, crushed, missing product)
- Blister defects (eg, missing, empty blisters)
- Bottle defects (eg, under/over-fill, no safety seal)
- Vial defects
- Product defect (eg, odor, chipped, broken, embossing illegible)
- Loss or theft of product

### 8.5.1 Eliciting and Reporting Product Quality Complaints

The investigator or designee must record all PQCs identified through any means from the receipt of the IMP from sponsor through and including reconciliation and up to destruction, including subject dosing. The investigator or designee must notify the sponsor (or sponsor's designee) within 24 hours of becoming aware of the PQC by e-mail or telephone and according to the procedure outlined below:

- Online Send information required for reporting purposes (listed below) to
- Phone Call Center at

Identification of a PQC by the subject should be reported to the site investigator, who should then follow one of the reporting mechanisms above.

### 8.5.2 Information Required for Reporting Purposes

- Description of compliant
- Reporter identification (eg, subject, investigator, site, etc)
- Reporter contact information (eg, address, phone number, e-mail address.)
- ID of material (product/compound name, coding)
- Clinical protocol reference (number and/or trial name)
- Dosage form/strength (if known)
- Pictures (if available)
- Availability for return

### 8.5.3 Return Process

Indicate during the report of the PQC if the complaint sample is available for return. If complaint sample is available for return, return it in the product retrieval package, which will be provided by OAPI-EQC.

It should be documented in the site accountability record that a complaint sample for a dispensed kit has been forwarded to OAPI-EQC for complaint investigation.

### 8.5.4 Assessment/Evaluation

Assessment and evaluation of Product Quality complaints will be handled by OAPI EQC-QM group.

### 9 Records Management

### 9.1 Source Documents

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include but are not limited to progress notes, electronic data, screening logs, and recorded data from automated instruments. All source documents pertaining to this trial will be maintained by the investigators and made available for direct inspection by authorized persons. Investigator(s)/institution(s) will permit trial-related monitoring, audits, IRB/IEC review, and regulatory inspection(s) by providing direct access to source data/documents by authorized persons as defined in the ICF.

### 9.2 Data Collection

During each subject's visit to the clinic, a clinician participating in the trial will record progress notes to document all significant observations. At a minimum, these notes will contain:

- Documentation of the informed consent process, including any revised consents;
- The date of the visit and the corresponding Visit in the trial schedule;
- General subject status remarks, including any *significant* medical findings. The severity, frequency, and duration of any AEs and the investigator's assessment of relationship to the IMP must also be recorded;
- Any changes in concomitant medications or dosages;
- A general reference to the procedures completed;
- The signature (or initials) and date of all clinicians who made an entry in the progress notes.

In addition, any contact with the subject via telephone or other means that provides significant clinical information will also be documented in the progress notes as described above. Any changes to information in the trial progress notes or other source documents will be <u>initialed and dated on the day the change is made</u> by a site trial staff member authorized to make the change. Changes will be made by striking a single line through erroneous data, and clearly entering the correct data (eg, wrong data right data). If the reason for the change is not apparent, a brief explanation for the change will be written in the source documentation by the clinician.

Information from the trial progress notes and other source documents will be data entered by investigative site personnel directly onto eCRFs in the sponsor's electronic data capture system.

### 9.3 File Management at the Trial Site

The investigator will ensure that the trial center file is maintained in accordance with Section 8 of the ICH GCP and as required by applicable local regulations. The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

### 9.4 Records Retention at the Trial Site

Regulatory requirements for the archival of records for this trial necessitate that participating investigators maintain detailed clinical data for the longest of the following three periods:

- A period of at least 2 years following the date on which approval to market the drug is obtained (or if IMP development is discontinued, the date regulatory authorities were notified of discontinuation); OR
- A period of at least 3 years after the sponsor notifies the investigator that the final report has been filed with regulatory authorities.
- Longer, region-specific storage requirements, if applicable.

The investigator must not dispose of any records relevant to this trial without either (1) written permission from the sponsor or (2) provision of an opportunity for the sponsor or designated agent to collect such records. The investigator will be responsible to maintain adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial, including the eCRF data on the CD-ROM and any data clarification forms received from the sponsor (or sponsor's

designee). Such documentation is subject to inspection by the sponsor, sponsor's designee, and relevant regulatory agencies. If the investigator withdraws from the trial (eg, due to relocation or retirement), all trial related records should be transferred to a mutually agreed upon designee within a sponsor-specified timeframe. Notice of such transfer will be given to the sponsor (or designee) in writing.

### 10 Quality Control and Quality Assurance

### 10.1 Monitoring

The sponsor has ethical, legal, and scientific obligations to follow this trial in a detailed and orderly manner in accordance with established research principles, the ICH GCP Guideline, FDA regulations and applicable regulatory requirements and local laws. As part of a concerted effort to fulfill these obligations (maintain current personal knowledge of the progress of the trial), the sponsor's monitors or designee will visit the site during the trial, as well as communicate frequently via telephone and written communications.

### 10.2 Auditing

The sponsor's Quality Management Unit (or representative) may conduct trial site audits. Audits will include, but are not be limited to, drug supply, presence of required documents, the informed consent process, and comparison of eCRFs with source documents. The investigator agrees to participate with audits.

Regulatory authorities may inspect the investigator during or after the trial. The investigator will cooperate with such inspections and will contact the sponsor immediately if such an inspection occurs.

## 11 Ethics and Responsibility

This trial must be conducted in compliance with the protocol, FDA regulations, the ICH GCP Guideline, and all other applicable local laws and regulatory requirements. Each trial site will seek approval by an IRB or EC according to regional requirements. The IRB/IEC will evaluate the ethical, scientific and medical appropriateness of the trial. Further, in preparing and handling eCRFs, the investigator, subinvestigator, and their staff will take measures to ensure adequate care in protecting subject privacy. To this end, a subject number and subject identification code will be used to identify each subject.

### 12 Confidentiality

All information generated in this trial will be considered highly confidential and will not be disclosed to anyone not directly concerned with the trial without the sponsor's prior written permission. However, authorized regulatory officials and sponsor personnel (or their representatives) will be allowed full access to inspect and copy the records. All IMPs, subject bodily fluids, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the sponsor.

Subjects will be identified only by initials and unique subject numbers in eCRFs. Per country regulations, if subject initials cannot be collected, another unique identifier will be used. Their full names may, however, be made known to a regulatory agency or other authorized officials if necessary.

### 13 Amendment Policy

The investigator will not make any changes to this protocol without prior written consent from the sponsor (or sponsor's designee) and subsequent approval by the IRB/IEC. Any permanent change to the protocol, whether it be an overall change or a change for specific trial site(s), must be handled as a protocol amendment. Any amendment will be written by the sponsor. Each amendment will be submitted to the IRB/IEC. Except for non-substantial (ie, administrative) amendments, investigators will wait for IRB/IEC approval of the amended protocol before implementing the change(s). Administrative amendments are defined as having no effect on the safety or physical or mental integrity of subjects, the conduct or management of the trial, the scientific value of the trial or the quality or safety of IMP(s) used in the trial. However, a protocol change intended to eliminate an apparent immediate hazard to subjects should be implemented immediately, followed by IRB/IEC notification within 5 working days. The sponsor (or sponsor's designee) will submit protocol amendments to the FDA or other regulatory agencies.

When the IRB/IEC, investigators, and/or the sponsor conclude that the protocol amendment substantially alters the trial design and/or increases the potential risk to the subject, the currently approved written ICF will require similar modification. In such cases, after approval of the new ICF by the IRB/IEC, repeat informed consent will be obtained from subjects in a timely manner before expecting continued participation in the trial.

### 14 References

- 1 Mueller TI, Leon AC, Keller MB, Solomon DA, Endicott J, et al. Recurrence after recovery from Major Depressive Disorder during 15 years of observational follow-up. Am J Psychiatry. 1999;156:1000-6.
- 2 Eaton WW, Shao H, Nestadt G, Lee BH, Bienvenu OJ, Zandi P. Population-based study of first onset and chronicity in Major Depressive Disorder. Arch Gen Psychiatry. 2008;65:513-20.
- 3 Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, et al. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR\*D: Implications for clinical practice. Am J Psychiatry. 2006;163:28-40.
- 4 Moller HJ. Outcomes in major depressive disorder: the evolving concept of remission and its implications for treatment. World J Biol Psychiatry. 2008;9:102-14.
- 5 Mulder RT, Frampton CM, Luty SE, Joyce PR. Eighteen months of drug treatment for depression: Predicting relapse and recovery. J Affect Disord. 2009;114:263-70.
- 6 Judd LL, Schettler PJ, Akiskal HS. The prevalence, clinical relevance, and public health significance of subthreshold depressions. Psychiatr Clin North Am. 2002;25:685-98.
- 7 McIntyre RS, O'Donovan C. The human cost of not achieving full remission in depression. Can J Psychiatry. 2004;49(Suppl 1):10S-16S.
- 8 Sobocki P, Jonsson B, Angst J, Rehnberg C. Cost of depression in Europe. J Ment Health Policy Econ. 2006;9:87-98.
- 9 American Psychiatric Association. Practice Guideline for the Treatment of Patients with Major Depressive Disorder, Second Edition. Arlington, VA: American Psychiatric Association; 2000.
- 10 Trivedi MH, Thase ME, Osuntokun O, Henley DB, Case M, Watson SB, et al. An integrated analysis of olanzapine/fluoxetine combination in clinical trials of treatment-resistant depression. J Clin Psychiatry. 2009;70:387-96.
- 11 Bauer M, El-Khalili N, Dato C, Szamosi J, Eriksson H. A pooled analysis of two randomised, placebo-controlled studies of extended release quetiapine fumarate adjunctive to antidepressant therapy in patients with major depressive disorder. J Affect Disord. 2010;127:19-30.
- 12 Marcus RN, McQuade RD, Carson WH, Hennicken D, Fava M, Simon J, et al. The efficacy and safety of aripiprazole as adjunctive therapy in major depressive disorder. A second multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychopharmacol. 2008;28:156-65.
- 13 Berman RM, Marcus RN, Swanink R, McQuade RD, Carson WH, Corey-Lisle PK, et al. The efficacy and safety of aripiprazole as adjunctive therapy in major depressive disorder: A multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2007;68:843-853.

- 14 Mahmoud RA, Pandina GJ, Turkoz I, Kosik-Gonzalez C, Canuso CM, Kujawa MJ, et al. Risperidone for treatment-refractory major depressive disorder: a randomized trial. Ann Intern Med. 2007;147:593-602.
- 15 Reynolds GP, Kirk SL. Metabolic side effects of antipsychotic drug treatment pharmacological mechanisms. Pharmacol Ther. 2010;125:169-79.
- 16 Sharpley AL, Attenburrow ME, Hafizi S, Cowen PJ. Olanzapine increases slow wave sleep and sleep continuity in SSRI-resistant depressed patients. J Clin Psychiatry. 2005;66(4):450-4.
- 17 Miller DD. Atypical antipsychotics: Sleep, sedation, and efficacy. Prim Care Companion J Clin Psychiatry. 2004;6(Suppl 2):3-7.
- 18 Ohno Y. New insight into the therapeutic role of 5-HT1A receptors in central nervous system disorders. Cent Nerv Syst Agents Med Chem. 2010;10:148-57.
- 19 OPC-34712 Investigator's Brochure, Otsuka Pharmaceutical Development & Commercialization, Inc. Version No. 6, 03 Mar 2011.
- 20 A phase 2, multicenter, randomized, double-blind, placebo-controlled study of the safety and efficacy of OPC-34712 as adjunctive therapy in the treatment of patients with major depressive disorder. Otsuka Clinical Study Report for Protocol 331-08-211, issued 23 Mar 2011.
- 21 A phase 2, 6-week, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of oral OPC-34712 once daily and aripiprazole once daily for treatment of hospitalized adult patients with acute schizophrenia. Otsuka Clinical Study Report for Protocol 331-07-203, issued 09 Mar 2011.
- 22 Blier P and Szabo SR. Potential mechanisms of action of atypical antipsychotic medications in treatment-resistant depression and anxiety. J Clin Psychiatry. 2005;66(Suppl 8):30-40.
- 23 Trivedi MH, Hollander E, Nutt D, Blier P. Clinical evidence and potential neurobiological underpinnings of unresolved symptoms of depression. J Clin Psychiatry. 2008;69:246-58.
- 24 The Practical Guide: Identification, evaluation, and treatment of overweight and obesity in adults. Developed by National Institutes of Health National Heart, Lung and Blood Institute. North American Association for the Study of Obesity. NIH Publication Number 00-4084, October 2000.
- 25 Simpson GN, Angus JWS. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand. 1970;212(Suppl 44):S11-S19.
- 26 Guy W. ECDEU Assessment Manual for Psychopharmacology. US Department of Health, Education, and Welfare publication (ADM) 76-338. Rockville, MD: National Institute of Mental Health; 1976.
- 27 Barnes TR. A rating scale for drug-induced akathisia. Br J Psychiatry. 1989;154:672 6.

- 28 Labbate LA, Lare SB. Sexual dysfunction in male psychiatric outpatients: validity of the Massachusetts General Hospital Sexual Functioning Questionnaire. Psychother Psychosom. 2001;70:221-5.
- 29 Sheehan DV. The Anxiety Disease. New York: Charles Scribner & Sons; 1983.
- 30 Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996;11(Suppl 3):89-95.
- 31 Rush AJ, Gullion CM, Basco MR, Jarrett RB, Trivedi MH. The Inventory of Depressive Symptomatology (IDS): Psychometric properties. Psychol Med. 1996;26:477-86.
- 32 Loke YK, Trivedi AN, Singh S. Meta-analysis: gastrointestinal bleeding due to interaction between selective serotonin uptake inhibitors and non-steroidal anti-inflammatory drugs. Aliment Pharmacol Ther. 2008;27:31-40.
- 33 US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Public Health Advisory 2006 19 Jul [cited 24 Oct 2011]. Available at www.fda.gov/DrugS/DrugSafety/PostmarketDrugSafetyInformationforPatientsandPro viders/DrugSafetyInformationforHeathcareProfessionals/PublicHealthAdvisories/ucm 124349.htm
- 34 US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Drug Safety Communication 2011 26 Jul [updated 2011 21 Oct; cited 24 Oct 2011]. Available at www.fda.gov/Safety/MedWatch/SafetyInformation/SafetyAlertsforHumanMedicalPr oducts/ucm265479.htm
- 35 US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Drug Safety Communication 2011 26 Jul [updated 2011 21 Oct; cited 24 Oct 2011]. Available at www.fda.gov/Safety/MedWatch/SafetyInformation/SafetyAlertsforHumanMedicalPr oducts/ucm265476.htm

### Appendix 1 Names of Sponsor Personnel



### Protocol 331-10-238



### **Appendix 2 Institutions Concerned With the Trial**

### **Clinical Research Organization**

INC Research 3201 Beechleaf Court, Suite 600 Raleigh, NC 27604-1547 USA

### **Safety Reporting**

Please report SAEs, AEs requiring discontinuation of drug product, and pregnancies to INC Research Pharmacovigilance & Drug Safety as follows:

| Country | Safety Fax Line |
|---------------------|-----------------|
| United States | |
| Canada | |
| France | |
| Germany | |
| Hungary | <u> </u> |
| Poland | |
| Romania | |
| Russia | |
| Slovakia | |
| Ukraine | _ |
| All other countries | |

### **Medical Monitors**

# North America: Primary: r Phone: Mobile: Fax: E-mail:





# Clinical Lab - ECG Central Reader

eResearch Technology 1818 Market Street, Suite 1000 Philadelphia, PA 19103-3638 USA

### **Central Laboratory**

Covance Laboratories 8211 SciCor Drive Indianapolis, IN 46214 USA

### **Subject Recruitment/Retention**

INC Research 3201 Beechleaf Court, Suite 600 Raleigh, NC 27604-1547 USA

### Materials for Subject Recruitment/Retention

Southport Graphics 210 James Jackson Avenue Cary, NC, 27513 USA

Phone: (919) 650-3822

### **Electronic Data Capture**

Medidata Solutions 79 5th Avenue, 8th floor New York, NY 10003 USA

### **Rater Training**

Bracket 575 East Swedesford Road, Suite 200 Wayne, PA 19087 USA

### **IVRS/IWRS**

S-Clinica 6, chaussée de Boondael B-1050 Brussels, Belgium

### **Translation Agency**

Global Language Solutions, Inc. 25 Enterprise, Suite 500 Aliso Viejo, CA 92656 USA

### **Central IRB**

Schulman Associates IRB 4445 Lake Forest Drive Suite 300 Cincinnati, OH 45242 USA

Appendix 3 Criteria for Identifying Vital Signs of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Heart Rate b | > 120 bpm<br>< 50 bpm | ≥ 15 bpm increase<br>≥ 15 bpm decrease |
| Systolic Blood Pressure b | > 180 mmHg<br>< 90 mmHg | ≥ 20 mmHg increase<br>≥ 20 mmHg decrease |
| Diastolic Blood Pressure b | > 105 mmHg<br>< 50 mmHg | ≥ 15 mmHg increase<br>≥ 15 mmHg decrease |
| Orthostatic Hypotension | $\geq$ 20 mmHg decrease in systolic blood<br>pressure and a $\geq$ 25 bpm increase in<br>heart rate from supine to<br>sitting/standing | Not Applicable (baseline status not considered) |
| Weight | <del>-</del> | ≥ 7% increase<br>≥ 7% decrease |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

As defined in "Supplementary Suggestions for Preparing an Integrated Summary of Safety Information in an Original NDA Submission and for Organizing Information in Periodic Safety Updates," FDA Division of Neuropharmacological Drug Products draft (2/27/87).

Appendix 4 Criteria for Identifying Laboratory Values of Potential Clinical Relevance

| Laboratory Tests | Criteria |
|---|---|
| Chemistry | |
| AST (SGOT) | $\geq$ 3 x upper limit of normal (ULN) |
| ALT (SGPT) | $\geq 3 \times ULN$ |
| Alkaline phosphatase | $\geq 3 \text{ x ULN}$ |
| LDH | $\geq$ 3 x ULN |
| BUN | $\geq$ 30 mg/dL |
| Creatinine | $\geq 2.0 \text{ mg/dL}$ |
| Uric Acid | |
| Men | $\geq 10.5 \text{ mg/dL}$ |
| Women | $\geq 8.5 \text{ mg/dL}$ |
| Bilirubin (total) | $\geq 2.0 \text{ mg/dL}$ |
| CPK | $\geq 3 \times ULN$ |
| Prolactin | > ULN |
| Hematology | |
| Hematocrit | |
| Men | $\leq$ 37 % and decrease of $\geq$ 3 percentage points from Baseline |
| Women | $\leq$ 32 % and decrease of $\geq$ 3 percentage points from Baseline |
| Hemoglobin | |
| Men | $\leq 11.5 \text{ g/dL}$ |
| Women | $\leq 9.5 \text{ g/dL}$ |
| White blood count | $\leq 2,800/ \text{ mm}^3 \text{ or } \geq 16,000/ \text{ mm}^3$ |
| Eosinophils | ≥ 10% |
| Neutrophils | ≤ 10%<br>≤ 15% |
| • | 3 |
| Absolute neutrophil count | $\leq 1,000/\text{ mm}^3$ |
| Platelet count | $\leq 75,000/ \text{ mm}^3 \text{ or } \geq 700,000/ \text{ mm}^3$ |
| Urinalysis | |
| Protein | Increase of $\geq 2$ units |
| Glucose | Increase of $\geq 2$ units |
| Casts | Increase of $\geq 2$ units |
| Additional Criteria | |
| Chloride | $\leq$ 90 mEq/L or $\geq$ 118 mEq/L |
| Potassium | $\leq 2.5 \text{ mEq/L or} \geq 6.5 \text{ mEq/L}$ |
| Sodium | $\leq 126 \text{ mEq/L or} \geq 156 \text{ mEq/L}$ |
| Calcium | $\leq 8.2 \text{ mg/dL or} \geq 12 \text{ mg/dL}$ |
| Glucose | |
| Fasting | $\geq 100 \text{ mg/dL}$ |
| Non-Fasting | $\geq 200 \text{ mg/dL}$ |
| Total Cholesterol, Fasting | $\geq$ 240 mg/dL |
| LDL Cholesterol, Fasting | $\geq 160 \text{ mg/dL}$ |
| HDL Cholesterol, Fasting | C |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Triglycerides, Fasting | $\geq 150 \text{ mg/dL}$ |

Appendix 5 Criteria for Identifying ECG Measurements of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Rate | | |
| Tachycardia | ≥ 120 bpm | increase of $\geq 15$ bpm |
| Bradycardia | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Rhythm | | |
| Sinus tachycardia b | ≥ 120 bpm | increase of ≥ 15 bpm |
| Sinus bradycardia c | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Supraventricular premature beat | all | not present → present |
| Ventricular premature beat | all | not present → present |
| Supraventricular tachycardia | all | not present → present |
| Ventricular tachycardia | all | not present → present |
| Atrial fibrillation | all | not present → present |
| Atrial flutter | all | not present → present |
| Conduction | | |
| 1° atrioventricular block | $PR \ge 200 \text{ msec}$ | increase of $\geq 50$ msec |
| 2° atrioventricular block | all | not present → present |
| 3° atrioventricular block | all | not present → present |
| Left bundle-branch block | all | not present → present |
| Right bundle-branch block | all | not present → present |
| Pre-excitation syndrome | all | not present → present |
| Other intraventricular conduction block d | QRS ≥ 120 msec | increase of $\geq 20$ msec |
| Infarction | | |
| Acute or subacute | all | not present → present |
| Old | all | not present $\rightarrow$ present |
| | | ≥ 12 weeks post study entry |
| ST/T Morphological | | |
| Myocardial Ischemia | all | not present $\rightarrow$ present |
| Symmetrical T-wave inversion | all | not present $\rightarrow$ present |
| Increase in QTc | $QTcF \ge 450 \text{ msec}$ (males and females) | |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> No current diagnosis of supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>c</sup> No current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>d</sup> No current diagnosis of left bundle branch block or right bundle branch block.

### **Appendix 6** Clinical Global Impression - Severity of Illness Scale (CGI-S)

Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?

0 = Not assessed 4 = Moderately ill

1 = Normal, not at all ill 5 = Markedly ill

2 = Borderline mentally ill 6 = Severely ill

3 = Mildly ill 7 = Among the most extremely ill patients

### Appendix 7 Clinical Global Impression - Improvement Scale (CGI-I)

Rate total improvement whether or not in your judgment it is due entirely to drug treatment. Compared to his/her condition at the last scheduled visit of the prior double-blind phase 3 trial (ie, prior to enrollment into Trial 331-10-238), how much has patient changed?

0 = Not assessed 4 = No change

1 = Very much improved 5 = Minimally worse

2 = Much improved 6 = Much worse

3 = Minimally improved 7 = Very much worse

### **Appendix 8** Sheehan Disability Scale (SDS)

### **Instructions to the investigator:**

The Sheehan Disability Scale is a measurement of functional disability and impairment due to psychiatric symptoms. It consists of 3 functional impairment items and 2 items related to productivity losses due to the symptoms and impairment.

The Sheehan Disability Scale is a self rated questionnaire and should be administered to the patient to be completed on his/her own without the presence or influence of study investigator/nurse or other individuals.

You should instruct the patient to report the disability and impairment experienced during the **past week** due to his/her **symptoms**. Emphasize that you will not interfere with the completion or have any comments to the patient's responses.

Please note that a questionnaire that has been completed by the patient is considered as source data and cannot be amended by the investigator or any other individual.

### Reference: Sheehan DV. The Anxiety Disease. New York. Charles Scribner and Sons, 1983 Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. International Clinical Psychopharmacology 1996;11:89-95.

### SHEEHAN DISABILITY SCALE

A BRIEF, PATIENT RATED, MEASURE OF DISABILITY AND IMPAIRMENT

Please mark ONE circle for each scale.







### **DAYS LOST**

On how many days in the last week did your symptoms cause you to miss school or work or leave you unable to carry out your normal daily responsibilities?

### DAYS UNDERPRODUCTIVE

On how many days in the last week did you feel so impaired by your symptoms, that even though you went to school or work, your productivity was reduced?\_\_\_\_\_

© Copyright 1983, 2010 David V. Sheehan. All rights reserved. Reproduced with permission of the author

# Appendix 9 Inventory of Depressive Symptomatology (Self-Report) (IDS-SR)

Please circle the one response to each item that best describes you for the past seven days.

### 1. Falling Asleep:

- 0 I never take longer than 30 minutes to fall asleep.
- 1 I take at least 30 minutes to fall asleep, less than half the time.
- 2 I take at least 30 minutes to fall asleep, more than half the time.
- 3 I take more than 60 minutes to fall asleep, more than half the time.

### 2. Sleep During the Night:

- 0 I do not wake up at night.
- 1 I have a restless, light sleep with a few brief awakenings each night.
- I wake up at least once a night, but I go back to sleep easily.
- 3 I awaken more than once a night and stay awake for 20 minutes or more, more than half the time.

### 3. Waking Up Too Early:

- 0 Most of the time, I awaken no more than 30 minutes before I need to get up.
- 1 More than half the time, I awaken more than 30 minutes before I need to get up.
- 2 I almost always awaken at least one hour or so before I need to, but I go back to sleep eventually.
- 3 I awaken at least one hour before I need to, and can't go back to sleep.

### 4. Sleeping Too Much:

- 0 I sleep no longer than 7-8 hours/night, without napping during the day.
- 1 I sleep no longer than 10 hours in a 24-hour period including naps.
- 2 I sleep no longer than 12 hours in a 24-hour period including naps.
- 3 I sleep longer than 12 hours in a 24-hour period including naps.

### 5. Feeling Sad:

- 0 I do not feel sad.
- 1 I feel sad less than half the time.
- 2 I feel sad more than half the time.
- 3 I feel sad nearly all of the time.

### 6. Feeling Irritable:

- 0 I do not feel irritable.
- 1 I feel irritable less than half the time.
- 2 I feel irritable more than half the time.
- 3 I feel extremely irritable nearly all of the time.

### 7. Feeling Anxious or Tense:

- 0 I do not feel anxious or tense.
- I feel anxious (tense) less than half the time.
- 2 I feel anxious (tense) more than half the time.
- 3 I feel extremely anxious (tense) nearly all of the time.

### 8. Response of Your Mood to Good or Desired Events:

- 0 My mood brightens to a normal level which lasts for several hours when good events occur.
- 1 My mood brightens but I do not feel like my normal self when good events occur.
- 2 My mood brightens only somewhat to a rather limited range of desired events.
- 3 My mood does not brighten at all, even when very good or desired events occur in my life.

### 9. Mood in Relation to the Time of Day:

- O There is no regular relationship between my mood and the time of day.
- 1 My mood often relates to the time of day because of environmental events (e.g., being alone, working).
- 2 In general, my mood is more related to the time of day than to environmental events.
- 3 My mood is clearly and predictably better or worse at a particular time each day.
- 9A. Is your mood typically worse in the morning, afternoon or night? (circle one)
- 9B. Is your mood variation attributed to the environment? (yes or no) (circle one)

### 10. The Quality of Your Mood:

- The mood (internal feelings) that I experience is very much a normal mood.
- 1 My mood is sad, but this sadness is pretty much like the sad mood I would feel if someone close to me died or left.
- 2 My mood is sad, but this sadness has a rather different quality to it than the sadness I would feel if someone close to me died or left.
- 3 My mood is sad, but this sadness is different from the type of sadness associated with grief or loss.

Reprinted with permission from A. John Rush Jr., M.D.

### Please complete either 11 or 12 (not both)

### 11. Decreased Appetite:

- 0 There is no change in my usual appetite.
- I eat somewhat less often or lesser amounts of food than usual.
- 2 I eat much less than usual and only with personal effort.
- 3 I rarely eat within a 24-hour period, and only with extreme personal effort or when others persuade me to eat.

### 12. Increased Appetite:

- 0 There is no change from my usual appetite.
- 1 I feel a need to eat more frequently than usual.
- 2 I regularly eat more often and/or greater amounts of food than usual.
- 3 I feel driven to overeat both at mealtime and between meals.

### Please complete either 13 or 14 (not both)

### 13. Decreased Weight (Within the Last Two Weeks):

- 0 I have not had a change in my weight.
- 1 I feel as if I've had a slight weight loss.
- 2 I have lost 2 pounds or more.
- 3 I have lost 5 pounds or more.

### 14. Increased Weight (Within the Last Two Weeks):

- 0 I have not had a change in my weight.
- 1 I feel as if I've had a slight weight gain.
- 2 I have gained 2 pounds or more.
- 3 I have gained 5 pounds or more.

### 15. Concentration/Decision Making:

- O There is no change in my usual capacity to concentrate or make decisions.
- I occasionally feel indecisive or find that my attention wanders.
- 2 Most of the time, I struggle to focus my attention or to make decisions.
- 3 I cannot concentrate well enough to read or cannot make even minor decisions.

### 16. View of Myself:

- I see myself as equally worthwhile and deserving as other people.
- I am more self-blaming than usual.
- 2 I largely believe that I cause problems for others.
- 3 I think almost constantly about major and minor defects in myself.

### 17. View of My Future:

- 0 I have an optimistic view of my future.
- I am occasionally pessimistic about my future, but for the most part I believe things will get better.
- 2 I'm pretty certain that my immediate future (1-2 months) does not hold much promise of good things for me.
- 3 I see no hope of anything good happening to me anytime in the future.

### 18. Thoughts of Death or Suicide:

- 0 I do not think of suicide or death.
- 1 I feel that life is empty or wonder if it's worth living.
- 2 I think of suicide or death several times a week for several minutes.
- 3 I think of suicide or death several times a day in some detail, or I have made specific plans for suicide or have actually tried to take my life.

### 19. General Interest:

- O There is no change from usual in how interested I am in other people or activities.
- 1 I notice that I am less interested in people or activities.
- 2 I find I have interest in only one or two of my formerly pursued activities.
- 3 I have virtually no interest in formerly pursued activities.

### 20. Energy Level:

- 0 There is no change in my usual level of energy.
- 1 I get tired more easily than usual.
- I have to make a big effort to start or finish my usual daily activities (for example, shopping, homework, cooking or going to work).
- 3 I really cannot carry out most of my usual daily activities because I just don't have the energy.

### Capacity for Pleasure or Enjoyment (excluding sex):

- 0 I enjoy pleasurable activities as much as usual.
- 1 I do not feel my usual sense of enjoyment from pleasurable activities.
- 2 I rarely get a feeling of pleasure from any activity.
- 3 I am unable to get any pleasure or enjoyment from anything.

Reprinted with permission from A. John Rush Jr., M.D.

### 22. Interest in Sex (Please Rate Interest, not Activity):

- I'm just as interested in sex as usual.
- My interest in sex is somewhat less than usual or I do not get the same pleasure from sex as I used to.
- I have little desire for or rarely derive pleasure from sex.
- I have absolutely no interest in or derive no pleasure from sex.

### 23. Feeling slowed down:

- I think, speak, and move at my usual rate of speed.
- I find that my thinking is slowed down or my voice sounds dull or flat.
- It takes me several seconds to respond to most questions and I'm sure my thinking is slowed.
- I am often unable to respond to questions without extreme effort.

### 24. Feeling restless:

- I do not feel restless.
- I'm often fidgety, wring my hands, or need to shift how I am sitting.
- I have impulses to move about and am quite restless.
- At times, I am unable to stay seated and need to pace around.

### 25. Aches and pains:

- I don't have any feeling of heaviness in my arms or legs and don't have any aches or pains.
- Sometimes I get headaches or pains in my stomach, back or joints but these pains are only sometime present and they don't stop me from doing what I
- I have these sorts of pains most of the time.
- These pains are so bad they force me to stop what I 30. Leaden Paralysis/Physical Energy: am doing.

### 26. Other bodily symptoms:

- I don't have any of these symptoms: heart pounding fast, blurred vision, sweating, hot and cold flashes, chest pain, heart turning over in my chest, ringing in my ears, or shaking.
- I have some of these symptoms but they are mild and are present only sometimes.
- 2 I have several of these symptoms and they bother me quite a bit.
- I have several of these symptoms and when they occur I have to stop doing whatever I am doing.

# 27. Panic/Phobic symptoms:

- I have no spells of panic or specific fears (phobia) (such as animals or heights).
- I have mild panic episodes or fears that do not usually change my behavior or stop me from functioning.
- I have significant panic episodes or fears that force me to change my behavior but do not stop me from functioning.
- I have panic episodes at least once a week or severe fears that stop me from carrying on my daily activities.

### 28. Constipation/diarrhea:

- There is no change in my usual bowel habits.
- I have intermittent constipation or diarrhea which is mild.
- I have diarrhea or constipation most of the time but it does not interfere with my day-to-day functioning.
- I have constipation or diarrhea for which I take medicine or which interferes with my day-today activities.

### 29. Interpersonal Sensitivity:

- I have not felt easily rejected, slighted, criticized or hurt by others at all.
- I have occasionally felt rejected, slighted, criticized or hurt by others.
- I have often felt rejected, slighted, criticized or hurt by others, but these feelings have had only slight effects on my relationships or work.
- I have often felt rejected, slighted, criticized or hurt by others and these feelings have impaired my relationships and work.

- I have not experienced the physical sensation of feeling weighted down and without physical energy.
- I have occasionally experienced periods of feeling physically weighted down and without physical energy, but without negative effect on work, school, or activity level.
- I feel physically weighted down (without physical energy) more than half the time.
- I feel physically weighted down (without physical energy) most of the time, several hours per day, several days per week.

| Which 3 item | is (questions) were the easiest to understand? | |
|---|---|---|
| Thank you | | |
| Range 0-84 | Score: | Reprinted with permission from A. John Rush Jr., M.D. |

### Appendix 10 Simpson Angus Scale (SAS)

### Circle the appropriate score for each item:

### 1. GAIT

The patient is examined as he walks into the examining room; his gait, the swing of arms, his general posture; all form the basis for an overall score for this item. This is rated as follows:

- 0 Normal
- 1 Mild diminution in swing while the patient is walking
- 2 Obvious diminution in swing suggesting shoulder rigidity
- 3 Stiff gait with little or no arm swing noticeable
- 4 Rigid gait with arms slightly pronated; or stooped-shuffling gait with propulsion and retropulsion.

### 2. ARM DROPPING

The patient and the examiner both raise their arms to shoulder height and let them fall to their sides, in a normal subject a stout slap is heard as the arms hit the sides. In the patient with extreme Parkinson's syndrome, the arms fall very slowly.

- 0 Normal, free fall with loud slap and rebound
- 1 Fall slowed slightly with less audible contact and little rebound
- 2 Fall slowed, no rebound
- 3 Marked slowing, no slap at all
- 4 Arms fall as though against resistance; as though through glue

### 3. SHOULDER SHAKING

The subject's arms are bent at a right angle at the elbow and taken one at a time by the examiner who grabs one hand and also clasps the other around the patient's elbow. The subject's upper arm is pushed to and fro and the humerus is externally rotated. The degree of resistance from normal to extreme rigidity is scored as follows:

- 0 Normal
- 1 Slight stiffness and resistance
- 2 Moderate stiffness and resistance
- 3 Marked rigidity with difficulty in passive movement
- 4 Extreme stiffness and rigidity with almost a frozen joint

### 4. ELBOW RIGIDITY

The elbow joints are separately bent at right angles and passively extended and flexed, with the subject's biceps observed and simultaneously palpated. The resistance to the procedure is rated. (The presence of cogwheel rigidity is noted separately.)

- 0 Normal
- 1 Slight stiffness and resistance
- 2 Moderate stiffness and resistance
- 3 Marked rigidity with difficulty in passive movement
- 4 Extreme stiffness and rigidity with almost a frozen joint

### 5. WRIST RIGIDITY

The wrist is held in one hand and then the fingers held by the examiner's other hand with the wrist moved to extension, and both ulnar and radial deviation. The resistance to this procedure is rated:

- 0 Normal
- 1 Slight stiffness and resistance
- 2 Moderate stiffness and resistance
- 3 Marked rigidity with difficulty in passive movement
- 4 Extreme stiffness and rigidity with almost a frozen joint

### 6. HEAD ROTATION

The patient sits or stands and is told that you are going to move his head from side to side, that it will not hurt and that he should try and relax. (Questions about pain in the cervical area or difficulty in moving his head should be obtained to avoid causing any pain.) Clasp the patient's head between the two hands with fingers on back of the neck. Gently rotate the head in a circular motion 3 times and evaluate the muscular resistance to the movement.

- 0 Loose, no resistance
- 1 Slight resistance to movement although the time to rotate may be normal
- 2 Resistance is apparent and time of rotation is slowed
- 3 Resistance is obvious and rotation is slowed
- 4 Head appears stiff and rotation is difficult to carry out

### 7. GLABELLA TAP

Subject is told to open his eyes and not to blink. The glabella region is tapped at a steady, rapid speed. The number of times patient blinks in succession is noted:

- 0 0-5 blinks
- 1 6-10 blinks
- 2 11-15 blinks
- 3 16-20 blinks
- 4 21 and more blinks

### 8. TREMOR

Patient is observed walking into examining room and then is examined for this item:

- 0 Normal
- 1 Mild finger tremor, obvious to sight and touch
- 2 Tremor of hand or arm occurring spasmodically
- 3 Persistent tremor of one or more limbs
- 4 Whole body tremor

### 9. SALIVATION

Patient is observed while talking and then asked to open his mouth and elevate his tongue. The following ratings are given:

- 0 Normal
- 1 Excess salivation so that pooling takes place if the mouth is open and the tongue raised
- 2 Excess salivation is present and might occasionally result in difficulty in speaking
- 3 Speaking with difficulty because of excess salivation
- 4 Frank drooling

### 10. AKATHISIA

Patient is observed for restlessness. If restlessness is noted, ask: "Do you feel restless or jittery inside; is it difficult to sit still?" Subjective response is not necessary for scoring but patient report can help make the assessment.

- 0 No restlessness reported or observed
- 1 Mild restlessness observed
- 2 Moderate restlessness observed
- 3 Restlessness is frequently observed
- 4 Restlessness persistently observed

Adapted and used with permission by Simpson GN and Angus JWS, "A Rating Scale for Extrapyramidal Side Effects," *Acta Psychiatr Scand*, 1970, 212 (Suppl 44):11-9.

### **Appendix 11 Abnormal Involuntary Movement Scale (AIMS)**

| | crate highest severity observed. Rate tour upon activation one less than those busly. Code for $0 = \text{Nor}$ $1 = \text{Min}$ $2 = \text{Mil}$ $3 = \text{Moo}$ $4 = \text{Sev}$ | e<br>imal, n<br>l<br>lerate | | extren | ne norm | al |
|---|---|---|---|---|---|---|
| | . 50 | | ( | Circle | One) | |
| | 1. MUSCLES OF FACIAL EXPRESSION e.g. movements of forehead, eyebrows, periorbital area, cheeks; include frowning, blinking, smiling, grimacing | 0 | 1 | 2 | 3 | 4 |
| FACIAL AND<br>ORAL | <ol><li>LIPS AND PERIORAL AREA e.g. puckering, pouting,<br/>smacking.</li></ol> | 0 | 1 | 2 | 3 | 4 |
| MOVEMENTS: | <b>3. JAW</b> e.g. biting, clenching, chewing, mouth opening, lateral movement. | 0 | 1 | 2 | 3 | 4 |
| | 4. TONGUE Rate only increase in movement both in and out of mouth, not inability to sustain movement. | 0 | 1 | 2 | 3 | 4 |
| EXTREMITY<br>MOVEMENTS: | 5. UPPER (ARMS, WRISTS, HANDS, FINGERS) include choreic movements (i.e. rapid, objectively purposeless, irregular, spontaneous), athetoid movements (i.e. slow, irregular, complex, serpentine). Do not include tremor (i.e. repetitive, regular, rhythmic). | 0 | 1 | 2 | 3 | 4 |
| 6. | 6. LOWER (LEGS, KNEES, ANKLES, TOES) e.g. lateral knee movement, foot tapping, heel dropping, foot squirming, inversion and eversion of foot | 0 | 1 | 2 | 3 | 4 |
| TRUNK<br>MOVEMENTS: | <ol> <li>NECK, SHOULDERS, HIPS e.g. rocking, twisting, squirming, pelvic gyrations</li> </ol> | 0 | 1 | 2 | 3 | 4 |
| | 8. Severity of abnormal movements | | | | e, normal<br>Minimal<br>Mild<br>Moderate<br>Severe | 1 2 3 |
| GLOBAL<br>JUDGMENTS: | 9. Incapacitation due to abnormal movements | | | | e, normal<br>Minimal<br>Mild<br>Moderate<br>Severe | 1 2 3 |
| | 10. Patient's awareness of abnormal movements Rate only subject's report. | No awareness Aware, no distress Aware, mild distress Aware, moderate distress Aware, severe distress | | 0 1 2 3 | | |
| DENTAL | 11. Any current problems with teeth and/or dentures? | | | , | No<br>Yes | 0 |
| STATUS: | 12. Does patient usually wear dentures? | | | | No<br>Yes | - |

Guy, W. ed. ECDEU Assessment Manual for Psychopharmacology. US Dept of HEW, Publication No. (Adm): 76-338, 1976

### **Appendix 12** Barnes Akathisia Rating Scale (BARS)

Rating scale for drug-induced akathisia (Barnes Akathisia Rating Scale)

### Instructions

Patient should be observed while they are seated, and then standing while engaged in neutral conversation (for a minimum of two minutes in each position). Symptoms observed in other situations, for example while engaged in activity on the ward, may also be rated. Subsequently, the subjective phenomena should be elicited by direct questioning.

### **Objective**

- 0 Normal, occasional fidgety movements of the limbs
- Presence of characteristic restless movements: shuffling or tramping movements of the legs/feet, or swinging one leg while sitting, *and/or* rocking from foot to foot or "walking on the spot" when standing, *but* movements present for less than half the time observed
- Observed phenomena, as described in (1) above, which are present for at least half the observation period
- Patient is constantly engaged in characteristic restless movements, and/or has the inability to remain seated or standing without walking or pacing, during the time observed

### Subjective

Awareness of restlessness

- O Absence of inner restlessness
- 1 Non-specific sense of inner restlessness
- The patient is aware of an inability to keep the legs still, or a desire to move the legs, and/or complains of inner restlessness aggravated specifically by being required to stand still
- Awareness of intense compulsion to move most of the time and/or reports strong desire to walk or pace most of the time

Distress related to restlessness

- 0 No distress
- 1 Mild
- 2 Moderate
- 3 Severe

### Global clinical assessment of akathisia

- O Absent. No evidence of awareness of restlessness. Observation of characteristic movements of akathisia in the absence of a subjective report of inner restlessness or compulsive desire to move the legs should be classified as pseudoakathisia
- 1 Questionable. Non-specific inner tension and fidgety movements
- Mild akathisia. Awareness of restlessness in the legs and/or inner restlessness worse when required to stand still. Fidgety movements present, but characteristic restless movements of akathisia not necessarily observed. Condition causes little or no distress
- 3 *Moderate akathisia*. Awareness of restlessness as described for mild akathisia above, combined with characteristic restless movements such as rocking from foot to foot when standing. Patient finds the condition distressing
- 4 *Marked akathisia*. Subjective experience of restlessness includes a compulsive desire to walk or pace. However, the patient is able to remain seated for at least five minutes. The condition is obviously distressing
- 5 Severe akathisia. The patient reports a strong compulsion to pace up and down most of the time. Unable to sit or lie down for more than a few minutes. Constant restlessness which is associated with intense distress and insomnia

Reproduced from: A rating scale for drug-induced akathisia. T.R.E. Barnes, *British Journal of Psychiatry* (1989), **154**, 672-676.

© 1989 The Royal College of Psychiatrists.

### **Appendix 13** Columbia-Suicide Severity Rating Scale (C-SSRS)

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in **The Columbia Suicide History Form**, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103 -130, 2003.)

| For reprints of the C-SSRS contact | •/ |
|------------------------------------|--------------------------|
| | ; inquiries and training |
| requirements contact | |

# $\ @$ 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEATION | | |
|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | | e Last<br>isit |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. Have you wished you were dead or wished you could go to sleep and not wake up? If yes, describe: | Yes | No |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suicide (e.g., "I've thought about killing myself") without thoughts of ways to kill oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? If yes, describe: | Yes | No |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time, place or method details worked out (e.g., thought of method to kill self but not a specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as to when, where or how I would actually do itand I would never go through with it." Have you been thinking about how you might do this? If yes, describe: | Yes | No 🗆 |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: | Yes | No |
| 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? If yes, describe: | Yes | No 🗆 |

| INTENSITY OF IDEATION | | |
|---|---|---|
| The following features should be rated with respect to the mos above, with 1 being the least severe and 5 being the most seve Most Severe Ideation: | | Most<br>Severe |
| <i>Type # (1-5)</i> | Description of Ideation | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in v (5) Many times each day | week (4) Daily or almost daily | |
| Duration | | |
| | I-8 hours/most of day<br>More than 8 hours/persistent or continuous | |
| (2) Can control thoughts with little difficulty (5) | nting to die if you want to? Can control thoughts with a lot of difficulty Unable to control thoughts Does not attempt to control thoughts | |
| Deterrents Are there things - anyone or anything (e.g., family, religious from wanting to die or acting on thoughts of committing (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | | |
| Reasons for Ideation | | |
| What sort of reasons did you have for thinking about war to end the pain or stop the way you were feeling (in other this pain or how you were feeling) or was it to get attention Or both? (1) Completely to get attention, revenge or a reaction from others. (2) Mostly to get attention, revenge or a reaction from others. (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain. | words you couldn't go on living with on, revenge or a reaction from others? | |
| SUICIDAL BEHAVIOR | Since | |
|---|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Vis | it |
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part | Yes | No |
| thought of as method to kill oneself. Intent does not have to be 100%. If there is <b>any</b> intent/desire to die associated | | |
| with the act, then it can be considered an actual suicide attempt. <i>There does not have to be any injury or</i> | | |
| <b>harm</b> , just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no | | |
| injury results, this is considered an attempt. | | |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or | | |
| circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, | | |
| but they thought that what they did could be lethal, intent may be inferred. | | |
| Have you made a suicide attempt? | Total : | # of |
| Have you done anything to harm yourself? | Atten | npts |
| Have you done anything dangerous where you could have died? | | |
| What did you do? | | _ |
| Did you as a way to end your life? | | |
| Did you want to die (even a little) when you? | | |
| Were you trying to end your life when you? | | |
| Or did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to | | |
| relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior | *** | • |
| without suicidal intent) | Yes | No |
| If yes, describe: | | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for | Yes | No |
| that, actual attempt would have occurred). | _ | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an | | Ш |
| attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by | | |
| someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose | | |
| around neck but has not yet started to hang - is stopped from doing so. | Total | |
| Has there been a time when you started to do something to end your life but someone or | interru | pied |
| something stopped you before you actually did anything? | | _ |
| If yes, describe: | | |
| Aborted Attempt: | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual | П | П |
| stops him/herself, instead of being stopped by something else. | _ | _ |
| Has there been a time when you started to do something to try to end your life but you | Total | # of |
| stopped yourself before you actually did anything? | abort | ted |
| If yes, describe: | | |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization | Yes | No |
| or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death | _ | _ |
| by suicide (e.g., giving things away, writing a suicide note). | | |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such | | |
| as collecting pills, getting a gun, giving valuables away or writing a suicide note)? | | |
| If yes, describe: | | |
| Suicidal Behavior: | Yes | No |
| Suicidal behavior was present during the assessment period? | _ | _ |
| | | N |
| Completed Suicide: | Yes | No |

| Answer for Actual Attempts Only | Most Lethal<br>Attempt<br>Date: |
|---|---|
| <ol> <li>Actual Lethality/Medical Damage: <ol> <li>No physical damage or very minor physical damage (e.g., surface scratches).</li> <li>Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains).</li> <li>Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel).</li> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures).</li> </ol> </li> <li>Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area).</li> <li>Death</li> </ol> | Enter Code |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | Enter Code |

# Appendix 14 Massachusetts General Hospital Sexual Functioning Questionnaire (MSFQ)

Please answer all questions by <u>circling</u> the <u>correct answer</u> or the answer which seems the most <u>appropriate</u> to you (consider "normal" the time in your life prior to the past month when you were most satisfied with your sexual functioning).

| a) How has your interest in sex been over the past month? | | | | | |
|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater<br>than normal | | | moderately<br>diminished | markedly<br>diminished | totally<br>absent |
| b) How has y | our ability to | get sexually aro | used or excited be | en over the pas | t |
| month? | | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater normal than normal | | minimally diminished | moderately<br>diminished | markedly<br>diminished | totally<br>absent |
| c) How has y | our ability to | achieve orgasm | been over the pas | t month? | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater normal than normal | | minimally diminished | moderately<br>diminished | markedly<br>diminished | totally<br>absent |
| d) (for men o | nly) How has | your ability to g | get and maintain a | n erection been | over |
| the past montl | h? | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater normal than normal | | minimally diminished | moderately<br>diminished | markedly<br>diminished | totally<br>absent |
| e) How would you rate your overall sexual satisfaction over the past month? | | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 |
| greater<br>than normal | normal | minimally<br>diminished | moderately diminished | markedly<br>diminished | totally absent |

Copyright 1998, Depression and Clinical Research Program, Massachusetts General Hospital (Derived from the Arizona Sexual Experiences Scale and from the Guided Interview Questionnaire by Segraves and Segraves).

## **Appendix 15 Resource Utilization Form (RUF)**

#### **BASELINE**

We are interested in how often you have sought medical care or were hospitalized for any type of condition. (Note: **Do not include** any research visits.) Please refer to your personal calendar. Enter 0 if there were no visits (Question 1) or no hospitalizations (Questions 2 to 5).

1. In the past 3 months, how many visits did you make to any of the following?

| | | | Number of visits |
|---|---|---|---|
| a. | A primary care doctor | | $\square$ $\square$ visits |
| b. | Psychiatrist | | $\square$ $\square$ visits |
| c. | Counselor, psychologist or other mental health pro | fessional | $\square$ $\square$ visits |
| d. | Physicians other than your primary care doctor or mental health professional | | $\square$ $\square$ visits |
| e. | An emergency room or urgent care facility for the of your emotions, nerves, or mental health | treatment | $\square$ $\square$ visits |
| f. | An emergency room or urgent care facility for any | other reason? | $\square$ $\square$ visits |
| 2. | In the past 12 months, how many times were you be your emotions, nerves, or mental health? | nospitalized for th | ne treatment of |
| | (Enter 0 if there were no hospitalizations.) | $\square$ number of | times hospitalized |
| 3. | In the past 12 months, how many times were you h | nospitalized for a | ny other reason? |
| | (Enter 0 if there were no hospitalizations.) | $\square$ number of | times hospitalized |
| 4. | IF YOU WERE HOSPITALIZED in the past 12 m many days were you in the hospital for your emoti or mental health? | | talized |
| | of mental heartif? | □ □ days nospi | lanzeu |
| 5. | IF YOU WERE HOSPITALIZED in the past 12 m you hospitalized for any other reasons? | $\Box$ $\Box$ days hospi | |

#### **FOLLOW-UP**

We are interested in how often you have sought medical care for any type of condition since you started the study. (Note: **Do not include** any research visits.) Please refer to your personal calendar. Enter 0 if no visits were made.

f. An emergency room or urgent care facility for any other reason?

□ □ visits

## **Appendix 16** Protocol Amendment(s)/Administrative Change(s)

Amendment Number: 1

**Issue Date:** 23 November 2011

## **PURPOSE:**

The sponsor has determined the need for a formal amendment to the original protocol approved on 11 May 2011 to add additional clarity to trial procedures and to make several administrative changes.

#### **BACKGROUND:**

## 1. Clarification of trial procedures

- 1) Clarify dosing schedule of duloxetine 40 mg/day (once daily or 20 mg twice daily).
- 2) Clarify interval between dose adjustments by changing description from "at least one week" to "at least 5 days" and revise wording regarding rechallenge after dose is decreased to 0.5 mg/day.
- 3) Clarify that the serum pregnancy test is the definitive test for determining pregnancy, irrespective of urine pregnancy test result.
- 4) Clarify that subjects who are sterile (ie, women who have had an oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months; or men who have had orchidectomy) are not required to use two different methods of birth control.
- 5) Per recent posting from FDA, add linezolid and methylene blue to list of drugs that may result in serotonin syndrome if coadministered with SSRIs or SNRIs.

## 2. Administrative changes and correction of typographical errors

- 1) Replace OPC-34712 with approved generic name (ie, brexpiprazole)
- 2) Add EudraCT number
- 3) Update primary medical contact for OPDC personnel
- 4) Change name of United BioSource Corporation to Bracket
- 5) Update address of Schulman Associates IRB.

#### **MODIFICATIONS TO PROTOCOL:**

• **Bold and underlined text:** Changed text

• Bold and strikethrough text: Deleted text

• Bold and italicized text: Added text

TITLE PAGE

Brexpiprazole (OPC-34712)

Protocol No. 331-10-238 IND No. 103,958 *EudraCT No. 2011-001351-37* 

## Sponsor Representatives:



Issue Date:

11 May 2011

Date of Amendment 1:

23 November 2011

Entire protocol, Footnote

27 May 2011

## **23 November 2011**

SYNOPSIS, Name of Product:

| Name of Company: Otsuka Pharmaceutical | Protocol #331-10-238 |
|---------------------------------------------------|-------------------------|
| Development & Commercialization, Inc. | IND #103,958 |
| Name of Product: <i>Brexpiprazole</i> (OPC-34712) | EudraCT #2011-001351-37 |

## SYNOPSIS, Objective(s):

Primary: To assess the long-term safety and tolerability of oral OPC-34712 (*hereafter referred to by the generic name "brexpiprazole"*) as adjunctive therapy in the treatment of adults with MDD.

Secondary: To assess the long-term efficacy of oral **OPC-34712 brexpiprazole** as adjunctive therapy in the treatment of adults with MDD.

SYNOPSIS, Trial Design, Paragraph 1, Sentences 1 and 3:

This is a multicenter, 52-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive **OPC-34712** <u>brexpiprazole</u> in depressed adults on concurrent antidepressant therapy (ADT). The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed one of the double-blind, phase 3 efficacy trials (ie, Trial 331-10-227 or Trial 331-10-228) and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral **OPC-34712** <u>brexpiprazole</u> for MDD.

SYNOPSIS, Trial Design, Paragraph 3, Treatment Phase, Sentence 1:

Eligible subjects will receive daily treatment with open-label **OPC-34712** <u>brexpiprazole</u> and ADT as described in the Investigational Medicinal Product, Dose, Formulation, Mode of Administration section.

SYNOPSIS, Subject Population, Paragraph 1, Sentence 1:

The subject population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with **OPC-34712 brexpiprazole** for MDD and who meet one of the following conditions:

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, Paragraph 1:

Trial medication (ie, investigational medicinal product [IMP]) will be provided to the investigator(s) by the sponsor (or designated agent) and will consist of open-label **OPC-34712** brexpiprazole and open-label ADTs.

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, *OPC-34712*, Paragraph 1 and bulleted list:

**OPC-34712 Brexpiprazole**: Open-label **OPC-34712 brexpiprazole** will be supplied as 0.5, 1, 2, and 3-mg tablets packaged in weekly blister cards, each containing sufficient tablets for 7 (+ 2 days). Blister cards will be dispensed at each scheduled visit and at unscheduled visits if the dose of **OPC-34712 brexpiprazole** is changed. All doses of **OPC-34712 brexpiprazole** should be taken orally once daily and can be administered without regard to meals. For convenience, **OPC-34712 brexpiprazole** may be taken with the first daily dose of ADT.

All subjects will be dosed as follows:

• The first dose of open-label OPC-34712 <u>brexpiprazole</u> will be taken one day after the last dose is taken for the double-blind, phase 3 efficacy trial so that adjunctive treatment will continue without interruption. It is anticipated that the last dose of the double-blind, phase 3 efficacy trial will be taken the day of the Week 14 visit of Trial

- 331-10-227 or Trial 331-10-228 (ie, the day of the Screening/Baseline visit for the open-label trial). Subjects will initiate open-label dosing with **brexpiprazole** 0.5 mg/day **OPC-34712** for 1 week. Subjects unable to tolerate **brexpiprazole** 0.5 mg/day **OPC-34712** must be withdrawn from the trial.
- The dose of <u>brexpiprazole</u> <u>OPC-34712</u> will be increased to 1 mg/day at the Week 1 visit. Subjects unable to tolerate <u>brexpiprazole</u> 1 mg/day <u>OPC-34712</u> may decrease to 0.5 mg/day at any time after the Week 1 visit.
- Investigators may further increase the dose to <a href="mailto:brexpiprazole">brexpiprazole</a> 2 mg/day <a href="mailto:OPC-34712">OPC-34712</a>, with an interval of at least <a href="mailto:one-week">one-week</a> 5 days</a> between dose increases. An interval of at least <a href="mailto:one-week">one-week</a> 5 days</a> between dose adjustments is recommended for dose decreases; however, the dose of <a href="mailto:brexpiprazole">brexpiprazole</a> OPC-34712 can be decreased at the investigator's discretion in a stepwise manner at any time after the Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response.
- Subjects who tolerate a reduced dose of <a href="mailto:brexpiprazole">brexpiprazole</a> 0.5 mg/day OPC-34712 at least once during the trial. In addition, the dose of <a href="mailto:brexpiprazole">brexpiprazole</a> OPC-34712 can be reescalated as necessary following any dose decrease if, in the investigator's judgment, rechallenge with a higher dose is warranted in order to identify an optimum dose for the subject. Subjects must return to the clinic for unscheduled visits if changes to the dose of <a href="mailto:brexpiprazole">brexpiprazole</a> OPC-34712 (increases or decreases) are required between scheduled visits.

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, *ADT*, Paragraph 1, Sentences 3 and 4:

It is recommended that the dose of ADT not be changed while the dose of <a href="mailto:becapture">becapture</a> DPC-34712 is being optimized (ie, no change to ADT up to and including the Week 4 visit). After the Week 4 visit, the dose of ADT can be modified if necessary to achieve optimum efficacy and tolerability for the treatment regimen using the following rules: 1) at least <a href="mailto:one-week 5 days">one-week 5 days</a> must elapse between dose increases (either <a href="mailto:brexpiprazole">brexpiprazole</a> OPC-34712 or ADT), 2) an interval of at least <a href="mailto:one-week 5 days">one-week 5 days</a> between dose adjustments (either <a href="mailto:brexpiprazole">brexpiprazole</a> OPC-34712 or ADT) is recommended for dose decreases; however, the ADT dose can be decreased at the investigator's discretion at any time as needed for tolerability, and 3) subjects must return to the clinic for unscheduled visits if changes to the ADT dose are required between scheduled visits.

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, *ADT*, Paragraph 3:

All doses of ADT will be administered orally once daily except for duloxetine 40 mg/day that **is can be** administered **once daily or** as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily.

SYNOPSIS, Criteria for Evaluation, Primary Outcome Variable:

The primary outcome variable is the safety and tolerability of <u>brexpiprazole</u> <u>OPC-34712</u> which will be assessed by examining the frequency and severity of adverse events (AEs).

List of Abbreviations and Definitions of Terms:

## EudraCT European Clinical Trial Data Base

Investigational medicinal product (IMP)

For the purposes of this protocol, IMP refers to all trial medication supplied to the sites by the sponsor (or designated agent) and includes bottles of protocol-specified ADTs and blister cards containing **brexpiprazole OPC-34712**.

Section 1, Introduction, Paragraph 3:



Results from initial phase 2 trials showed **OPC-34712** <u>brexpiprazole</u> to be well tolerated by subjects with MDD and schizophrenia (see Section 1.3).

Section 1.1.1, Efficacy Pharmacology:

OPC-34712 Brexpiprazole functions as a partial agonist at the D2 receptor. In in vitro assay systems based on forskolin-induced cyclic AMP accumulation and calcium (Ca<sup>2+</sup>) mobilization in human dopamine D2L receptor-expressing cells, its intrinsic activity at the D2 receptor was slightly lower than that of aripiprazole, another D2 receptor partial agonist. OPC-34712 Brexpiprazole inhibited apomorphine (APO)-induced hyperlocomotion, APO-induced stereotyped behavior, and conditioned avoidance response in rats, which are predictive animal models for antipsychotic-like efficacy. The inhibitory effects of OPC-34712 brexpiprazole were more potent than those of aripiprazole. Moreover, in contrast to the D2 receptor antagonist risperidone, OPC-34712 brexpiprazole did not increase plasma prolactin levels in reserpine-treated rats, thus demonstrating a D2 receptor partial agonistic profile in vivo. Despite its lower intrinsic activity at the D2 receptor, the in vivo catalepsy liability of OPC-34712 brexpiprazole, an index of EPS, was similar to that of aripiprazole, but still lower than that of the typical antipsychotic haloperidol. Furthermore, OPC-34712 brexpiprazole showed high binding affinity for the 5-HT2A receptor and dose-dependently inhibited  $(\pm)$ -2,5-dimethoxy-4-iodoamphetamine-induced head twitch response in rats, indicating that the compound has 5-HT2A receptor antagonistic activity; the effect of **OPC-34712** brexpiprazole was more potent than that of aripiprazole. In addition, OPC-34712 brexpiprazole exhibited high binding affinities for the D3 and 5-HT1A receptors, acting as a partial agonist at these receptors.

#### Section 1.1.2, Safety Pharmacology:

In safety pharmacology studies in rats at an oral dose of 30 mg/kg or higher, OPC-34712 brexpiprazole induced pharmacologically mediated clinical signs considered to be due to depression of the central nervous system (CNS) and dose-dependent decreases in body temperature. When orally administered at up to 30 mg/kg in conscious male beagle dogs, OPC-34712 brexpiprazole showed no effect on respiratory parameters or heart rate at any dose tested. OPC-34712 Brexpiprazole decreased blood pressure at doses of 3 mg/kg or higher and prolonged both QT interval and corrected QT interval (QTc, by Van de Water's formula) at 30 mg/kg. OPC-34712 Brexpiprazole inhibited human ether-ago-go related gene (hERG) current in Chinese hamster ovary cells (CHO-K1) at concentrations of 10<sup>-8</sup> mol/L or higher, with a 50% inhibitory concentration of 1.17 ×

brexpiprazole was suggested to result from a blockade of the α<sub>1</sub>-adrenoceptor in peripheral blood vessels, which is a part of the compound's pharmacological profile. Proarrhythmic risk was also evaluated by examining the effects of OPC-34712 brexpiprazole on monophasic action potential parameters in halothane-anesthetized dogs. OPC-34712 Brexpiprazole did not affect the terminal repolarization period even at an intravenous dose of 3 mg/kg, suggesting a low potential for proarrhythmic effects. In general, the changes in the CNS, respiratory, and cardiovascular systems observed with OPC-34712 brexpiprazole occurred at doses or exposure levels higher than those at which efficacy was confirmed in rats (3 mg/kg), and similar changes were shown to occur after administration of risperidone at similar or lower doses.

## Section 1.2.1, Pharmacokinetics/pharmacodynamics:

The pharmacokinetics of single and multiple doses of OPC-34712 brexpiprazole was studied in healthy subjects and in subjects with MDD, attention-deficit/hyperactivity disorder (ADHD), and schizophrenia or schizoaffective disorder. Based on preclinical data and human clinical trials, brexpiprazole (OPC-34712) and one metabolite, DM-3411, were identified as the major analytes that are present in human plasma. In vitro, the activity of DM-3411 is 17 times lower than that of OPC-34712 brexpiprazole and thus is considered as an inactive metabolite. Both OPC-34712 brexpiprazole and DM-3411 pharmacokinetics were linear following single oral doses of brexpiprazole 0.2 to 8 mg OPC-34712 to healthy subjects. The terminal phase elimination half-life of OPC-34712 brexpiprazole-and DM-3411 was 48.3 to 80.8 hours and 48.6 to 77.5 hours, respectively. The median time to maximum (peak) plasma concentration (t<sub>max</sub>) occurred at approximately 2 to 6 hours postdose for OPC-34712 brexpiprazole and at approximately 10 to 24 hours postdose for DM-3411. In healthy subjects, administration of single-dose OPC-34712 brexpiprazole with a high-fat meal did not affect its rate and extent of absorption.

Steady state pharmacokinetics also appeared to be linear following multiple daily doses of  $\overline{OPC-34712}$   $\underline{brexpiprazole}$  in the range of 0.5 to 2 mg to healthy subjects. The accumulation factor based on maximum (peak) plasma concentration ( $C_{max}$ ) and area under the concentration-time curve calculated to the last observable concentration at time t ( $AUC_t$ ) was approximately 4 times. After multiple dose administration of  $\underline{OPC-34712}$   $\underline{brexpiprazole}$  (1 to 12 mg/day) to subjects with schizophrenia or schizoaffective disorder,  $\underline{OPC-34712}$   $\underline{brexpiprazole}$  and DM-3411 mean terminal elimination half-life

at steady state was 95.4 and 89.3 hours, respectively; median  $t_{max}$  was 3.0 and 8.0 hours, respectively.

In drug interaction trials in healthy subjects, **OPC-34712** <u>brexpiprazole</u> was shown to be metabolized by CYP3A4 and CYP2D6 isozymes and was not an inhibitor of CYP3A4, CYP2B6, CYP2D6, or P-glycoprotein. Coadministration of potent CYP3A4 or CYP2D6 inhibitors with **OPC-34712** <u>brexpiprazole</u> resulted in about a 2-fold higher exposure and about a 1.5-fold increase in the terminal elimination half life of **OPC-34712** <u>brexpiprazole</u> with fluoxetine, paroxetine, or duloxetine (MDD medications coadministered in this trial) may potentially increase **OPC-34712** <u>brexpiprazole</u> plasma concentrations by up to 2-fold.

In a single-dose trial in healthy subjects, approximately 46.0% and 24.6% of administered radioactivity following an oral dose of  $^{14}\text{C-}\text{OPC-}34712 \text{ brexpiprazole}$  was excreted in feces and urine, respectively. In this same trial, OPC-34712 brexpiprazole did not preferentially bind to red blood cells. OPC-34712 Brexpiprazole showed high protein binding in human serum ( $\geq 99.8\%$ ) in vitro.

The binding of **OPC-34712** <u>brexpiprazole</u> to dopamine receptors was assessed using positron emission tomography (PET). The mean D2/D3 receptor occupancies at 4 and 24 hours postdose after 0.25, 0.5, 1, 2, 4, 5, and 6 mg single dose administration of **OPC-34712** <u>brexpiprazole</u> to healthy subjects were 11.4% to 17.4%, 36.5% to 46.3%, 45.6% to 60.2%, 52.7% to 68.6%, 67.9% to 79.5%, 71.9% to 88.2%, and 69.5% to 92.6%, respectively (Trial 331-07-202). Based on the single-dose D2/D3 receptor occupancy data and steady-state pharmacokinetic/pharmacodynamic (PK/PD) modeling, it was predicted that the D2/D3 receptor occupancy after multiple daily dose administration of 1 to 2 mg and higher doses of **OPC-34712** <u>brexpiprazole</u> will result in at least 80% to 90% D2/D3 receptor occupancy.

Additional information on the pharmacokinetics/pharmacodynamics of **OPC-34712 brexpiprazole** and its metabolites in humans can be found in the Investigator Brochure. 

Section 1.2.2, Major Depressive Disorder

The efficacy of **OPC-34712 brexpiprazole** as adjunctive therapy for the treatment of MDD has been studied in one completed placebo-controlled trial (Trial 331-08-211). An additional placebo-controlled efficacy trial (Trial 331-09-222) and one long-term openlabel safety trial (Trial 331-08-212) are ongoing. Trial 331-08-211 was a multicenter, randomized, double-blind, placebo-controlled trial designed to assess the safety and

efficacy of OPC-34712 brexpiprazole (0.15 to 2 mg daily) as adjunctive treatment to an assigned open-label ADT in subjects with MDD who have demonstrated an incomplete response to prospective treatment with the same ADT. Subjects with an incomplete response after 8 weeks of treatment with single-blind placebo plus open-label ADT were randomized to 6 weeks of double-blind treatment with either OPC-34712 brexpiprazoleplus-ADT or placebo-plus-ADT. Responders continued to receive placebo-plus-ADT for an additional 6 weeks. Randomized subjects received brexpiprazole 0.15 mg/dayOPC-34712,  $0.50 \pm 0.25$  mg/day OPC-34712,  $1.5 \pm 0.50$  mg/day OPC-34712, or matching placebo. Subjects randomized to the **brexpiprazole**  $0.50 \pm 0.25$  mg/day **OPC-34712** and **brexpiprazole**  $1.5 \pm 0.50$  mg/day **OPC-34712** arms were titrated to the target doses (0.50) and 1.5 mg, respectively) over a 2-week period. Dose adjustments were permitted after the subjects received 1 week of treatment at the target dose. Subjects who could not tolerate the lowest dose (**brexpiprazole** 0.15, 0.25, or 1.0 mg/day **OPC-34712** or matching placebo, respectively) were to be discontinued from the trial. In this trial, adjunctive  $\frac{OPC-34712}{OPC}$  brexpiprazole dosed at  $1.5 \pm 0.50$  mg/day was superior to adjunctive placebo with respect to the primary endpoint (change from Week 8 to Week 14 in Montgomery Asberg Depression Rating Scale [MADRS] Total Score) and several secondary efficacy endpoints. Ongoing Trial 331-09-222 is of similar design to Trial 331-08-211, but is exploring an expanded dose range (brexpiprazole 1 to 3 mg/day<del>OPC-34712</del>).

Section 1.2.3, Schizophrenia, Sentence 2:

The outcome of this trial suggests an active dose range of **brexpiprazole** 1 to 6 mg/day **OPC-34712** for the treatment of schizophrenia.<sup>21</sup>

Section 1.2.4, Other Indications, Sentences 1 and 2:

OPC-34712 <u>Brexpiprazole</u> is being investigated in a proof-of-concept trial in adult ADHD (Trial 331-08-213). This is a multicenter, randomized, double-blind, placebo-controlled, flexible-dose trial in which adults with ADHD who have an incomplete/partial response to stimulant therapy in a prospective treatment phase are randomized to double-blind treatment with either OPC-34712 <u>brexpiprazole</u>-plus-stimulant or placebo-plus-stimulant.

Section 1.3, Known and Potential Risks and Benefits, Paragraph 1, Sentences 1, 4, and 5:

As of 31 Dec 2010, 14 clinical trials involving **OPC-34712** <u>brexpiprazole</u> have been completed worldwide, including 10 in the United States (US), 1 in multiple countries (including the US), 2 in Japan, and 1 in Korea.

OPC-34712 <u>Brexpiprazole</u> has been well tolerated by healthy volunteers at single doses up to 6 mg and at multiple doses up to 2 mg/day. In patient trials, OPC-34712 <u>brexpiprazole</u> has been well tolerated at multiple doses up to 12 mg/day in subjects with schizophrenia or schizoaffective disorder, up to 4 mg/day in subjects with MDD who received concomitant ADT, and up to 4 mg/day in adults with ADHD who received concomitant stimulant therapy.

Section 1.3, Known and Potential Risks and Benefits, Paragraph 2, Sentences 1 and 2:

In the 11 completed phase 1 and 2 clinical trials performed under the US IND (two phase 2 trials, one phase 1b trial, and eight phase 1 trials), 673/973 (69.2%) subjects who received **OPC-34712 brexpiprazole** either alone or coadministered with another marketed medication reported at least one treatment-emergent adverse event (TEAE) compared to 158/253 (62.5%) subjects who received placebo either alone or coadministered with another marketed medication. The most common TEAEs reported for **OPC-34712 brexpiprazole** in the completed trials ( $\geq 5\%$  in the total **OPC-34712 brexpiprazole** group and more than the total placebo group) were headache (10.6%), dizziness (8.0%), anxiety (7.1%), akathisia (7.0%), and nausea (5.5%).

Section 1.3, Known and Potential Risks and Benefits, Paragraph 3, Sentences 3 and 4:

The incidence of serious TEAEs (fatal and non-fatal) that were reported during treatment with OPC-34712 <u>brexpiprazole</u> administered either alone or coadministered with another medication (19/973 subjects, 2.0%) was comparable to placebo administered either alone or coadministered with another medication (4/253 subjects, 1.6%). Furthermore, treatment with OPC-34712 <u>brexpiprazole</u> does not appear to promote suicidal behavior in subjects with MDD or schizophrenia.

Section 1.3, Known and Potential Risks and Benefits, Paragraph 4:

OPC-34712 <u>Brexpiprazole</u> did not result in any consistent, clinically relevant changes in laboratory values, vital signs (blood pressure or heart rate), or electrocardiogram (ECG) parameters in the completed phase 1 and 2 clinical trials in subjects with MDD or schizophrenia. Statistically significant increases in weight were observed with OPC-34712 <u>brexpiprazole</u> relative to placebo in both sample populations. OPC-34712 <u>Brexpiprazole</u> exhibited a favorable profile with respect to movement disorders in subjects with MDD at doses up to 3 mg/day (Trial 331-09-221) and in subjects with

schizophrenia at doses up to 12 mg/day (Trial 331-08-205). In the dose-ranging trial that enrolled subjects who were experiencing an acute exacerbation of schizophrenia (Trial 331-07-203), an increase in the incidence of EPS was observed at the highest dose (ie, **brexpiprazole**  $5.0 \pm 1.0$  mg/day **OPC-34712**).

Section 2.1, Trial Rationale, Paragraph 1, Sentence 4:

As **OPC-34712** <u>brexpiprazole</u> demonstrated antagonism at 5-HT2A receptors, the attenuated response to SSRIs may be reversed with coadministration of **OPC-34712** <u>brexpiprazole</u> and SSRIs, thus enhancing clinical outcomes.

Section 2.1, Trial Rationale, Paragraph 2:

Because the management of MDD may require prolonged administration of ADT(s) with or without an augmenting agent, safety monitoring for longer than the period required to achieve initial response is warranted. In the **OPC-34712 brexpiprazole** clinical development program for MDD, phase 2 and phase 3 trials examined the 6-week safety and efficacy of **OPC-34712 brexpiprazole** augmentation of ADTs. For phase 2, subjects who completed either of the trials had the option to enroll into an open-label rollover trial in which they received **OPC-34712 brexpiprazole** for up to 52 weeks (Trial 331-08-212). The current trial (Trial 331-10-238) provides an open-label rollover option for the double-blind phase 3 trials (ie, Trial 331-10-227 and Trial 331-10-228) and will expand on the knowledge gained in these trials by assessing the long-term safety, tolerability, and efficacy of **OPC-34712 brexpiprazole** when administered concomitantly with antidepressant medications.

Section 2.2, Dosing Rationale, Paragraph 1:

A dose range of <u>brexpiprazole</u> 0.5 to 3 mg/day <del>OPC-34712</del> was selected for the current open-label trial to encompass the dose range of the double-blind efficacy trials (ie, <u>brexpiprazole</u> 1 to 3 mg/day <del>OPC-34712</del>) and to include an option for a reduced dose for tolerability (ie, 0.5 mg/day) in order to maximize subject retention in the long-term trial. Therapeutic dose ranges of ADT are based on product labels and clinical practice. Data from phase 1 drug interaction trials (Trial 331-08-207 and Trial 331-08-208) indicated that coadministration of CYP2D6 inhibitors (eg, paroxetine, fluoxetine, and duloxetine) with <del>OPC-34712</del> <u>brexpiprazole</u> could cause potentially higher plasma concentrations of <del>OPC-34712</del> <u>brexpiprazole</u> (up to 2-fold). In order to limit the potential higher exposure of <del>OPC-34712</del> <u>brexpiprazole</u> when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine in the current trial.

Section 2.3, Trial Objectives:

Primary: To assess the long-term safety and tolerability of oral **OPC-34712** 

**brexpiprazole** as adjunctive therapy in the treatment of adults with MDD.

Secondary: To assess the long-term efficacy of oral **OPC-34712 brexpiprazole** as

adjunctive therapy in the treatment of adults with MDD.

## Section 3.1, Type/Design of Trial, Paragraph 1, Sentences 1 and 3:

This is a multicenter, 52-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive **OPC-34712** <u>brexpiprazole</u> in depressed adults on concurrent antidepressant therapy (ADT). The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed one of the double-blind, phase 3 efficacy trials (ie, Trial 331-10-227 or Trial 331-10-228) and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral **OPC-34712** <u>brexpiprazole</u> for MDD.

Section 3.1, Type/Design of Trial, Paragraph 3, *Treatment Phase*, Sentence 1:

Eligible subjects will receive daily treatment with open-label **OPC-34712** <u>brexpiprazole</u> and ADT as described in Section 3.2.

Figure 3.1-1, Population and treatment group descriptions:

Eligible subjects who completed one of the double-blind phase 3 trials (ie, Trial 331-10-227 or Trial 331-10-228) and who could potentially benefit from adjunctive treatment with OPC-34712 brexpiprazole for MDD

per investigator

Open-label OPC-34712 Brexpiprazole (0.5 to 3 mg/day) + ADT

## Section 3.2.1.1, OPC-34712 Brexpiprazole:

The first dose of open-label **OPC-34712** <u>brexpiprazole</u> will be taken one day after the last dose is taken for the double-blind, phase 3 efficacy trial so that adjunctive treatment will continue without interruption. It is anticipated that the last dose of the double-blind, phase 3 efficacy trial will be taken the day of the Week 14 visit of Trial 331-10-227 or

Trial 331-10-228 (ie, the day of the Screening/Baseline visit for the open-label trial). Subjects will initiate open-label dosing with <a href="mailto:brexpiprazole">brexpiprazole</a> 0.5 mg/day OPC-34712 for 1 week. Subjects unable to tolerate <a href="mailto:brexpiprazole">brexpiprazole</a> 0.5 mg/day OPC-34712 must be withdrawn from the trial. The dose of OPC-34712 <a href="mailto:brexpiprazole">brexpiprazole</a> will be increased to 1 mg/day at the Week 1 visit. Subjects unable to tolerate <a href="mailto:brexpiprazole">brexpiprazole</a> 1 mg/day OPC-34712 may decrease to 0.5 mg/day at any time after the Week 1 visit.

Investigators may further increase the dose to <a href="brexpiprazole">brexpiprazole</a> 2 mg/day OPC 34712 and then to <a href="brexpiprazole">brexpiprazole</a> 3 mg/day OPC 34712, with an interval of at least one week 5 days between dose adjustments is recommended for dose decreases; however, the dose of OPC 34712 <a href="brexpiprazole">brexpiprazole</a> can be decreased at the investigator's discretion in a step-wise manner at any time after the Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response. Subjects must return to the clinic for unscheduled visits if changes to the dose of OPC-34712 <a href="brexpiprazole">brexpiprazole</a> (increases or decreases) are required between scheduled visits. The dosing schedule is summarized in Table 3.2.1.1-1. Additional information on dose adjustments is provided in Section 3.2.2.1.

All doses of **OPC-34712** <u>brexpiprazole</u> should be taken orally once daily and can be administered without regard to meals. For convenience, **OPC-34712** <u>brexpiprazole</u> may be taken with the first daily dose of ADT.

| Table 3.2.1.1-1 Dosing Schedule for OPC-34712 Brexpiprazole | | | | | |
|---|---|---|---|---|---|
| | Trial Visit | | | | |
| IMP | Screening/<br>Baseline | Week 1 <sup>a</sup> | Week 2 <sup>b</sup> | Week 4 <sup>b</sup> | Visits at Weeks 8, 14, 20, 26, 32, 38, and 44 |
| OPC-34712<br>Brexpiprazole<br>(mg/day) <sup>c</sup> | 0.5 | 1 | 0.5, 1 or 2 | 0.5, 1, 2 or 3 | 0.5, 1, 2, or 3 |
| ADT | Final dose<br>from double-<br>blind trial | No change | No change | No change | Change to ADT dose is permitted as described in Section 3.2.2.2. |

Subjects unable to tolerate **brexpiprazole** 1 mg/day **OPC-34712** may decrease to 0.5 mg/day at any time after the Week 1 visit.

Step-wise increases in the dose of **OPC-34712** <u>brexpiprazole</u> must be separated by at least <u>one week</u> <u>5 days</u>. Although step-wise decreases in the <u>OPC-34712</u> <u>brexpiprazole</u> dose are permitted at any time after the Week 1 visit to a minimum of 0.5 mg/day, an interval of at least <u>one week 5 days</u> between dose adjustments is recommended. See Section 3.2.2.1 for additional information on dose adjustments. Subjects must return to the clinic for unscheduled visits if changes to the dose of <u>OPC-34712</u> <u>brexpiprazole</u> (increases or decreases) are required between scheduled visits.

#### Section 3.2.1.2, ADT, Sentence 7:

All doses of ADT will be administered orally once daily except for duloxetine 40 mg/day that **is can be** administered **once daily or** as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily.

#### Table 3.2.1.2-1, Footnote a:

#### Section 3.2.2, Dose Adjustments

Dose modifications to both **OPC-34712** <u>brexpiprazole</u> and ADT will be permitted to optimize therapeutic benefit according to the rules described below for each treatment. However, the dose of **OPC-34712** <u>brexpiprazole</u> and the dose of ADT should not both be changed at the same visit.

#### Section 3.2.2.1, **OPC-34712** Brexpiprazole

Allowable dose modifications to the daily dose of OPC-34712 brexpiprazole are summarized in Table 3.2.2.1-1. At least one week 5 days must elapse between dose increases for OPC-34712 brexpiprazole. An interval of at least one week 5 days between dose adjustments is recommended for dose decreases; however, the dose of OPC-34712 brexpiprazole can be decreased at the investigator's discretion in a stepwise manner at any time after the Week 1 visit as needed for tolerability to a minimum of 0.5 mg/day. Subjects must return to the clinic for unscheduled visits if changes to the dose of OPC-34712 brexpiprazole (increases or decreases) are required between scheduled visits.

Subjects who are unable to tolerate the 0.5-mg/day dose of **OPC-34712** <u>brexpiprazole</u> must be withdrawn from the trial. However, subjects whose <u>OPC-34712</u> <u>brexpiprazole</u>

Subjects unable to tolerate the minimum dose of **OPC-34712** <u>brexpiprazole</u> (ie, 0.5 mg/day) must be withdrawn from the trial.

<sup>&</sup>lt;sup>d</sup>Throughout Trial 331-10-238, the subject must remain on the same ADT that was assigned in the double-blind phase 3 trial (ie, Trial 331-10-227 or Trial 331-10-228).

<sup>&</sup>lt;sup>e</sup>It is recommended that the dose of ADT not be changed while the dose of **OPC-34712** <u>brexpiprazole</u> is being optimized.

All doses are to be administered orally once daily except for duloxetine 40 mg/day that **is can be** administered **once daily or** as duloxetine 20 mg twice daily, duloxetine 60 mg/day that can be administered once daily or as duloxetine 30 mg twice daily, and fluoxetine 40 mg/day that can be administered once daily or in divided doses twice daily. All doses should be taken at approximately the same time each day, if possible.

dose is decreased to 0.5 mg/day and who demonstrate adequate tolerability at this dose should be rechallenged with a 1-mg/day dose within approximately 6 to 8 weeks after starting the dose is decreased to 0.5 mg/day dose. If tolerability issues arise following the rechallenge, the dose may be decreased again to 0.5 mg/day. Further rechallenge at 1 mg/day may be performed at the investigator's discretion. The dose of OPC-34712 brexpiprazole can be re-escalated as necessary following a dose decrease at any other dose if, in the investigator's judgment, rechallenge with a higher dose is warranted in order to identify an optimum dose for the subject. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response.

| <b>Table 3.2.2.1-1 Dose M</b> | lodifications for OPC-34712 | Brexpiprazole |
|---|---|---|
| | Dose Increases a,b | |
| Current Dose of OPC-34712 | Incremental Increase | Adjusted OPC-34712 |
| <u>Brexpiprazole</u> | | Brexpiprazole dose |
| 0.5 mg | 0.5 mg | 1 mg |
| 1 mg | 1 mg | 2 mg |
| 2 mg | 1 mg | 3 mg |
| Dose Decreases b,c | | |
| Current Dose of OPC-34712 | Incremental Decrease | Adjusted OPC-34712 |
| Brexpiprazole | | Brexpiprazole dose |
| 0.5 mg | Not permitted <sup>d</sup> | 0.5 mg <sup>d</sup> |
| 1 mg | 0.5 mg | 0.5 mg |
| 2 mg | 1 mg | 1 mg |
| 3 mg | 1 mg | 2 mg |

<sup>&</sup>lt;sup>a</sup>At least <del>one week <u>5 days</u></del> must elapse between dose increases.

## Section 3.2.2.2, ADT:

It is recommended that the dose of ADT not be changed while the dose of OPC-34712 brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). After the Week 4 visit, the dose of ADT can be modified if necessary to achieve optimum efficacy and tolerability for the treatment regimen using the following rules:

1) at least one week 5 days must elapse between dose increases (either OPC-34712)

bSubjects must return to the clinic for unscheduled visits if changes to the dose of **OPC-34712**brexpiprazole (increases or decreases) are required between scheduled visits.

An interval of at least one week 5 days between dose adjustments is recommended for dose decreases; however, the investigator may decrease the dose of OPC 34712 brexpiprazole at any time after the Week 1 visit for tolerability.

<sup>&</sup>lt;sup>d</sup>Subjects unable to tolerate 0.5 mg/day of **OPC-34712** <u>brexpiprazole</u> must be withdrawn from the trial.

<u>brexpiprazole</u> or ADT), 2) an interval of at least <u>one week 5 days</u> between dose adjustments (either <u>OPC-34712 brexpiprazole</u> or ADT) is recommended for dose decreases; however, the ADT dose can be decreased at the investigator's discretion at any time as needed for tolerability, and 3) subjects must return to the clinic for unscheduled visits if changes to the ADT dose are required between scheduled visits.

## Section 3.3, Trial Population, Paragraph 1, Sentence 1:

The trial population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with **OPC-34712** <u>brexpiprazole</u> for MDD and who meet one of the following conditions:

#### Table 3.4.2-1, Criterion 3:

- 3. Subjects who, in the opinion of the investigator, could potentially benefit from administration of **OPC 34712** <u>brexpiprazole</u> as adjunctive therapy to their antidepressant therapy and who meet one of the following criteria:
  - a) Subjects who completed participation in the Double-blind Randomization Phase (ie, Week 14 visit of Phase B) in Trial 331-10-227 or Trial 331-10-228 or
  - b) Subjects who met criteria for a response at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227 or Trial 331-10-228, **BUT DID NOT** meet criteria for remission (defined as a MADRS Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227 or Trial 331-10-228.

#### Table 3.4.3-1, Criterion 2 and Footnote a:

2. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving open-label **OPC-34712 brexpiprazole** in Trial 331-10-238.

## Section 3.5.1, Primary Outcome Variable:

The primary outcome variable is the safety and tolerability of **OPC-34712** <u>brexpiprazole</u> which will be assessed by examining the frequency and severity of adverse events (AEs).

## Table 3.6-1, Footnotes o, s and u:

All positive urine pregnancy test results must be confirmed by a serum test. Subjects with <u>a</u> positive <u>urine and</u> serum pregnancy test results at Screening/Baseline must not be enrolled in Trial 331-10-238- and <u>Ss</u>ubjects with <u>a</u> positive <u>urine and</u> serum pregnancy test results during the trial must discontinue treatment and be withdrawn from the trial. Pregnancy tests can be performed at any point during the trial if pregnancy is suspected.

<sup>&</sup>lt;sup>a</sup>Use of CYP2D6 inhibitors or CYP3A4 inhibitors and inducers is prohibited during the trial. Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs that are also CYP2D6 inhibitors. In order to limit the potential higher exposure of **OPC-34712** <u>brexpiprazole</u> when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine.

Adjustments to the dose of OPC-34712 brexpiprazole or ADT are permitted to optimize efficacy and tolerability as described in Section 3.2. It is recommended that the dose of ADT not be changed while the dose of OPC-34712 brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). At least one week 5 days must elapse between dose increases for OPC-34712 brexpiprazole and ADT. An interval of at least one week 5 days between dose adjustments is also recommended for dose decreases; however, the investigator may decrease the dose of OPC-34712 brexpiprazole or ADT as needed for tolerability according to the rules described in Section 3.2.2. Subjects must return to the clinic for unscheduled visits if changes to the dose of OPC-34712 brexpiprazole or ADT (increases or decreases) are required between scheduled visits.

<sup>u</sup>The IVRS/IWRS will be accessed at unscheduled visits if new blister cards are dispensed for dose adjustment of **OPC-34712 brexpiprazole**.

## Section 3.6.1.1, Screening/Baseline, Bullet 7:

Trial personnel will call the interactive voice response system (IVRS) or access the interactive web response system (IWRS) to register the visit and to obtain blister card and ADT bottle number assignments. The assigned open-label OPC-34712 brexpiprazole and ADT will be dispensed. Treatment will begin with brexpiprazole 0.5 mg/day OPC-34712 for 1 week. The ADT will be the same as the one taken during the double-blind phase 3 trial (ie, Trial 331-10-227 of Trial 331-10-228). The dose of ADT should not be changed at this time.

#### Section 3.6.1.2, Week 1, Bullets 10, 11, and 12:

- Women of childbearing potential (WOCBP) will be given a urine pregnancy test.
   Any positive result must be confirmed by a serum pregnancy test. WOCBP with <u>a</u> positive <u>urine and</u> serum pregnancy test results must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for OPC-34712 brexpiprazole and ADT.
- The dose of OPC-34712 <u>brexpiprazole</u> will be increased to 1 mg/day. Subjects unable to tolerate <u>brexpiprazole</u> 1 mg/day OPC-34712 may decrease to 0.5 mg/day at any time after the Week 1 visit. It is recommended that the dose of ADT not be changed while the dose of OPC-34712 <u>brexpiprazole</u> is being optimized. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for OPC-34712 <u>brexpiprazole</u> and ADT, and to obtain blister card and bottle number assignments. The assigned open-label OPC-34712 <u>brexpiprazole</u> and ADT will be dispensed to the subject.

#### Section 3.6.1.3, Week 2, Bullets 6, 7 and 8:

- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with <u>a positive urine and</u> serum pregnancy test results must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for **OPC-34712** brexpiprazole and ADT.

- The investigator will adjust the dose of OPC-34712 <a href="brexpiprazole">brexpiprazole</a> as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. It is recommended that the dose of ADT not be changed while the dose of OPC-34712 <a href="brexpiprazole">brexpiprazole</a> is being optimized. Any subject unable to tolerate the minimum dose of OPC-34712 <a href="brexpiprazole">brexpiprazole</a> (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for OPC-34712 <a href="brexpiprazole">brexpiprazole</a> and ADT, and to obtain blister card and bottle number assignments. The assigned open-label OPC-34712 <a href="brexpiprazole">brexpiprazole</a> and ADT will be dispensed to the subject.
- Section 3.6.1.4, Week 4, Bullets 9, 10 and 11:
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with <u>a</u> positive <u>urine and</u> serum pregnancy test results must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for **OPC-34712** <u>brexpiprazole</u> and ADT.
- The investigator will adjust the dose of **OPC-34712 brexpiprazole** as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. If necessary, the dose of ADT can be changed after the Week 4 visit, but not at the same visit as a change to the dose of **OPC-34712 brexpiprazole** (see Section 3.2.2.2). Any subject unable to tolerate the minimum dose of **OPC-34712 brexpiprazole** (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for **OPC-34712 brexpiprazole** and ADT, and to obtain blister card and bottle number assignments. The assigned openlabel **OPC-34712 brexpiprazole** and ADT will be dispensed to the subject.
- Section 3.6.1.5, Week 8, Bullets 11, 12 and 13:
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with <u>a positive urine and</u> serum pregnancy test results must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for **OPC-34712** brexpiprazole and ADT.
- The investigator will adjust the dose of OPC-34712 <u>brexpiprazole</u> as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for OPC-34712 <u>brexpiprazole</u> and ADT, and to obtain blister card and bottle number assignments. The assigned open-label OPC-34712 <u>brexpiprazole</u> and ADT will be dispensed to the subject.
- Section 3.6.1.6, Long-term Treatment Visits (Weeks 14, 20, 26, 32, 38, and 44), Bullets 7, 8 and 9 after Paragraph 1:

- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with <u>a positive urine and</u> serum pregnancy test results must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for OPC-34712 <u>brexpiprazole</u> and ADT.
- The investigator will adjust the dose of OPC-34712 brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for OPC-34712 brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label OPC34712 brexpiprazole and ADT will be dispensed to the subject.

Table 3.6.2.1-1, Footnote a:

Section 3.6.2.4, Other Safety Assessments, Sentence 5:

Training and materials for rating will be provided by **United BioSource Corporation Bracket**.

Section 3.6.3, Efficacy Assessments, Sentence 5:

Training, certification, and materials for rating will be provided by **United BioSource Corporation Bracket**.

Section 3.7.3, Individual Subject, Item f:

f) subject cannot tolerate the minimum dose of **OPC-34712** <u>brexpiprazole</u> (ie, 0.5 mg/day), the minimum protocol-defined therapeutic dose of ADT (see Table 3.2.1.2-1), or requires a different ADT; or

Section 3.8, Screen Failures, Sentence 2:

For the purposes of Trial 331-10-238, treatment begins with the first dose of open-label **OPC-34712** <u>brexpiprazole</u> in the Treatment Phase.

Section 3.11, Subject Compliance, Sentence 1:

Responsible trial personnel will dispense the IMP (ie, OPC-34712 brexpiprazole and ADTs).

Table 4.1-1, Footnote c:

<sup>&</sup>lt;sup>a</sup>All positive urine pregnancy test results must be confirmed by a serum test. Subjects with <u>a</u> positive <u>urine and</u> serum pregnancy test results at Screening/Baseline must not be enrolled in Trial 331-10-238-<u>and Ssubjects</u> with <u>a</u> positive <u>urine and</u> serum pregnancy test results during the trial must discontinue treatment and be withdrawn from the trial.

## Section 4.2.1, Restricted Therapies and Precautions, Bullet 2 after Paragraph 1:

Triptans (eg, sumatriptan, naratriptan, almotriptan, frovatriptan, rizatriptan, eletriptan, and zolmitriptan), *linezolid, and methylene blue* since there have been rare post-marketing reports of serotonin syndrome or serotonin syndrome-like reactions (eg, mental status changes, weakness, hyperreflexia, autonomic effects, and lack of coordination, and diarrhea) following the concomitant use of SSRIs or SNRIs and triptans these drugs.

## Section 4.2.1, Restricted Therapies and Precautions, Paragraphs 7 and 8:

Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs in this trial; however, they are also CYP2D6 inhibitors. Data from Trial 331-08-207 and Trial 331-08-208 indicate that coadministration of CYP2D6 inhibitors with **OPC-34712 brexpiprazole** can cause potentially higher plasma concentrations of **OPC-34712 brexpiprazole** (up to 2-fold). In order to limit the potential higher exposure of **OPC-34712 brexpiprazole** when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine. The investigator should consider the potential for higher **OPC-34712 brexpiprazole** plasma concentrations when adjusting the dose of **OPC-34712 brexpiprazole** for subjects who are receiving fluoxetine, paroxetine CR, or duloxetine as the assigned ADT.

All trial personnel should be familiar with the content of the Investigator Brochure for **OPC-34712 brexpiprazole** in order to manage the subject's condition adequately and select appropriate concomitant medications, if needed.

Section 5.1, Definitions, Last sentence:

Investigators will assess IMP causality based on OPC-34712 brexpiprazole.

Section 5.5, Pregnancy, Paragraph 1, Sentence 2:

Unless the subject and his/her partner(s) are <u>is</u> sterile (ie, women who have had an oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months; or men who have had orchidectomy) or remain<u>s</u> abstinent, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pills, birth control depot injection, birth control implant, condom or sponge with spermicide.

Fluoxetine, paroxetine, and duloxetine are protocol-defined ADTs that are also CYP2D6 inhibitors. In order to limit the potential higher exposure of **OPC 34712** <u>brexpiprazole</u> when coadministered with such inhibitors, the upper limit of the therapeutic ADT dose is limited to 40 mg for fluoxetine, 50 mg for paroxetine CR, and 60 mg for duloxetine (see Section 4.2.1).

Section 7.1.1, Data Sets for Analysis, Safety Sample definition:

Safety Sample: comprises those subjects who receive at least one dose of open-label **OPC-34712** brexpiprazole as adjunctive therapy to one of the allowed ADTs.

Section 7.4, Safety Analyses, Last sentence:

In general, baseline measurements of safety variables are defined as their last measurements prior to the first dose of open-label **OPC-34712** brexpiprazole.

Section 8.1, Packaging and Labeling, Paragraph 1:

Trial drugs will be provided to the investigator(s) by the sponsor (or designated agent). The IMP will consist of open-label **OPC-34712 brexpiprazole** and open-label ADTs. Open-label **OPC-34712 brexpiprazole** will be supplied as 0.5, 1, 2, and 3-mg tablets packaged in weekly blister cards, each containing sufficient tablets for 7 (+ 2 days). Blister cards will contain single tablet strengths (ie, **brexpiprazole** 0.5, 1, 2, or 3 mg/day **OPC-34712**) and subjects will take 1 tablet daily. When accessed by the site, the IVRS or IWRS will assign a specific blister card number to be dispensed to a subject. New weekly blister cards will be dispensed at each scheduled visit and at unscheduled visits if the dose of **OPC-34712 brexpiprazole** is changed.

Section 8.2, Storage, Paragraph 2, Sentence 1:

**OPC-34712 Brexpiprazole** should be stored according to the storage conditions indicated on the clinical label.

Section 8.3, Accountability:

The investigator, or designee, must maintain an inventory record of trial drugs (including **OPC-34712 brexpiprazole** and ADTs) received, dispensed, administered, and returned.

Section 8.4, Returns and Destruction, Paragraph 1:

Upon completion or termination of the trial, all unused and/or partially used IMP (including OPC-34712 brexpiprazole and ADTs) must be returned to Otsuka Pharmaceutical Development & Commercialization, Inc. (OPDC) (or a designated contractor).

Section 14, References:

US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Public Health Advisory 2006 19 Jul [updated 2006 24 Nov; cited 4 Nov 2008 24 Oct 2011]. Available at

US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Drug Safety Communication 2011 26 Jul [updated 2011 21 Oct; cited 24 Oct 2011]. Available at
 US Food and Drug Administration [homepage on the Internet]. Rockville, MD: FDA Drug Safety Communication 2011 26 Jul [updated 2011 21 Oct; cited 24 Oct 2011]. Available at

Appendix 1, Names of Sponsor Personnel, Primary Medical Contact:



Appendix 2, Institutions Concerned With the Trial

Rater Training
United BioSource Corporation
Specialty Clinical Services
Bracket
575 East Swedesford Road, Suite 200
Wayne, PA 19087
USA

## **Central IRB**

Schulman Associates IRB

4290 Glendale-Mulford Road

4445 Lake Forest Drive

Suite 300

Cincinnati, OH 45242

USA

Protocol 331-10-238

Add:

Appendix 16 Protocol Amendment(s)/Administrative Change(s)

## ADDITIONAL RISK TO THE SUBJECT:

There is no additional risk to the subjects as a result of this protocol amendment.

**Amendment Number:** 2

**Issue Date:** 16 November 2012

#### **PURPOSE:**

The sponsor has determined the need for a formal amendment to amendment 1 approved on 23 November 2011 to allow enrollment of eligible subjects who completed the last scheduled visit of a double-blind phase 3 brexpiprazole MDD trial, to remove the definitions of incomplete response and response, to match the specifications for potential Hy's Law cases, to clarify that the contraceptive methods of vasectomy and tubal ligation apply to the subject and partner, to update study duration and the estimated number of enrolled subjects, and to make administrative changes.

#### **BACKGROUND:**

- 1. Enrollment of subjects who completed the last scheduled visit of a doubleblind phase 3 brexpiprazole MDD trial
- 1) Add subjects who completed the last scheduled visit of double-blind phase 3 brexpiprazole MDD trials as those eligible for enrollment into Trial 331-10-238
- 2) Add statement that all assessments listed under screening need to be performed at Screening/Baseline of Trial 331-10-238; and that if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238

## 2. Definitions of incomplete response and response

• 1) Remove the definitions for incomplete response and response for Trial 331-10-227 and Trial 331-10-228

## 3. Hy's Law specifications

• 1) Update the specifications for potential Hy's Law cases

## 4. Contraceptive methods of vasectomy and tubal ligation

1) Clarify that that the contraceptive methods of vasectomy and tubal ligation apply to the subject and partner

## 5. Study duration and number of enrolled subjects

- 1) Update the study duration to approximately 63 months, of which approximately 51 months are allotted for rollover of subjects from the prior double-blind phase 3 trials
- 2) Update number of estimated enrolled subjects to 3,000

## 6. Administrative changes and correction of typographical errors

- 1) Update primary and backup medical contact for OPDC personnel
- 2) Remove safety reporting information for Czech Republic and add safety reporting information for "All Other Countries"

#### MODIFICATIONS TO PROTOCOL:

• **Bold and underlined text:** Changed text

Bold and strikethrough text: Deleted text
 Bold and italicized text: Added text

#### TITLE PAGE

Issue Date: 11 May 2011
Date of Amendment 1: 23 November 2011
Date of Amendment 2: 16 November 2012

Entire protocol, Footnote

#### 23 November 2011

#### **16 November 2012**

SYNOPSIS, Trial Design, Paragraph 1, Sentence 3:

This is a multicenter, 52-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive <u>brexpiprazole</u> in depressed adults on concurrent antidepressant therapy (ADT). The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed *the last scheduled visitone* of *thea* double-blind, phase 3 <u>efficacy-brexpiprazole MDD</u> trials (ie, Trial 331-10-227 or Trial 331-10-228) and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral brexpiprazole for MDD.

SYNOPSIS, Trial Design, Paragraph 3, Screening/Baseline, Sentences 1 and 3:

Subjects will be screened for eligibility at the last scheduled visit of the prior double-blind phase 3 trialof Trial 331-10-227 or Trial 331-10-228 (ie, Week 14). Subjects will sign a separate informed consent form for participation in Trial 331-10-238 before any procedures specific to the open-label trial are performed. The assessments from the last scheduled visit of the prior double-blind phase 3 trial Week 14 visit of Trial 331-10-227 or Trial 331-10-228 will serve as the baseline measures for Trial 331-10-238 for any assessment that is not unique to the open-label trial.

SYNOPSIS, Trial Design, Paragraph 3, Follow-up:

Subjects will be followed **up** for safety via telephone contact or clinic visit 30 (+ 2) days after the last dose of open-label medication.

SYNOPSIS, Subject Population:

The subject population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with brexpiprazole for MDD *according to the following criteria* who meet one of the following conditions:

- Subjects who participated in Trial 331-10-227 or Trial 331-10-228 only will be eligible for the 331-10-238 study if they meet one of the following conditions:
  - Subjects who completed participation in the double-blind randomization phase (ie, Week 14 visit of Phase B) in Trial 331-10-227 or Trial 331-10-228 or
  - Subjects who met criteria for a response continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227 or Trial 331-10-228, BUT DID NOT meet criteria for remission (defined as a Montgomery Asberg Depression Rating Scale MADRS Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227 or Trial 331-10-228.
- Subjects who participated in another double-blind phase 3 brexpiprazole MDD trial will be eligible for the 331-10-238 study if they have completed the last scheduled visit of the prior double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last *scheduled* visit of the *prior* double-blind *phase 3* trial and must be able to continue therapy without interruption between the double-blind and open label trials. Based on the projected enrollment estimates for the *prior* double-blind phase 3 *brexpiprazole MDD* trials (ie, Trial 331-10-227 and Trial 331-10-228), *up to approximately* to 12803,000 subjects may enroll into Trial 331-10-238.

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, *Brexpiprazole*, bulleted list, Paragraph 1, Sentences 1 and 2:

• The first dose of open-label brexpiprazole will be taken one day after the last dose is taken for the *prior* double-blind, phase 3 *brexpiprazole MDD* efficacy trial so that adjunctive treatment will continue without interruption. It is anticipated that

the last dose of the double-blind, phase 3 *brexpiprazole MDD* efficacy trial will be taken the day of the *last scheduled visit* Week 14 visit of Trial 331-10-227 or Trial 331-10-228, (ie, the day of the Screening/Baseline visit for the open-label trial).

SYNOPSIS, Investigational Medicinal Product, Dose, Formulation, Mode of Administration, *ADT*, Paragraph 1, Sentences 1 and 2:

ADT: During the Treatment Phase of Trial 331-10-238, subjects will remain on the same assigned open-label ADT from the *prior* double-blind, phase 3 *brexpiprazole*MDDefficacy trial (ie, Trial 331-10-227 or Trial 331-10-228). The initial dose of ADT will be the same as the ADT dose taken on the last *scheduled* visit of *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228.

SYNOPSIS, Trial Duration, Sentence 1:

The duration of this trial from first subject enrolled to last subject completed is estimated to be approximately 3063 months, of which approximately 1751 months are allotted for rollover of subjects from the *prior* double-blind phase 3 *brexpiprazole MDD* trials—(ie, Trial 331-10-227 or Trial 331-10-228).

List of Abbreviations and Definitions of Terms:

# Incomplete response

A term employed to assess prospective response to ADT during Phase A of the double-blind phase 3 trials (ie, Trial 331-10-227 and Trial 331-10-228) as part of eligibility criteria for entrance into Phase B. Incomplete response is defined as <50% reduction in depressive symptom severity between baseline and the Week 8 visit as measured by the 17-item Hamilton Depression Rating Scale (HAM-D17) Total Score; AND a HAM-D17 Total Score ≥ 14 at the Week 8 visit; AND a Clinical Global Impression - Improvement scale (CGI-I) score ≥3 at the Week 8 visit. Note: The visit of interest for this definition is the Week 8 visit of the double-blind phase 3 trial (ie, Trial 331-10-227 and Trial 331-10-228).

#### Response

A term employed to assess prospective response to ADT during Phase A of the double-blind phase 3 trials (ie, Trial 331-10-227 and Trial 331-10-228) and representing the logical complement of "incomplete response." Response is defined as ≥ 50% reduction in depressive symptom severity between baseline and the Week 8 visit as measured by the HAM-D17 Total Score; OR a HAM-D17 Total Score of < 14 at the Week 8 visit; OR a CGI-I score of < 3 at the Week 8 visit. Note: The visit of interest for this definition is the Week 8 visit of the double-blind phase 3 trial (ie, Trial 331-10-227 and Trial 331-10-228).

Section 2.1, Trial Rationale, Paragraph 2, Sentence 4:

The current trial (Trial 331-10-238) provides an open-label rollover option for **the** double-blind phase 3 *brexpiprazole MDD* trials-(ie, Trial 331-10-227 and Trial 331-10-228) and will expand on the knowledge gained in these trials by assessing the long-term safety, tolerability, and efficacy of brexpiprazole when administered concomitantly with antidepressant medications.

Section 3.1, Type/Design of Trial, Paragraph 1, Sentence 3:

This is a multicenter, 52-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive <u>brexpiprazole</u> in depressed adults on concurrent ADT. The trial will be conducted on an outpatient basis. Enrollment into the trial will be drawn from eligible subjects who have completed <del>onethe last scheduled visit</del> of the double-blind, phase 3 **efficacy brexpiprazole MDD** trials (ie, Trial 331-10-227 or Trial 331-10-228) and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral <u>brexpiprazole</u> for MDD.

Section 3.1, Type/Design of Trial, Paragraph 3, Screening/Baseline, Sentences 1 and 3:

Subjects will be screened for eligibility at the last scheduled visit of the prior double-blind phase 3 trial Trial 331-10-227 or Trial 331-10-228 (ie, Week 14). Subjects will sign a separate informed consent form for participation in Trial 331-10-238 before any procedures specific to the open-label trial are performed. The assessments from the last scheduled visit of the prior double-blind phase 3 trial (Week 14 visit of Trial 331-10-228) will serve as the baseline measures for Trial 331-10-238 for any assessment that is not unique to the open-label trial.

Section 3.1, Type/Design of Trial, Paragraph 3, *Follow-up*:

Subjects will be followed **up** for safety via telephone contact or clinic visit 30 (+ 2) days after the last dose of open-label medication.

Figure 3.1-1, Population and screening/baseline visit descriptions:

Eligible subjects who completed *the last scheduled visitene* of *thea* double-blind phase 3 *brexpiprazole MDD* trials (ie, Trial 331-10-228) and who could potentially benefit from adjunctive treatment with brexpiprazole for MDD per investigator

Last scheduled visit of a double-blind phase 3 brexpiprazole MDD

Ttrial 331-10-227 or

Trial 331-10-228

## Section 3.2.1.1, Brexpiprazole, Paragraph 1, Sentence 2:

The first dose of open-label brexpiprazole will be taken one day after the last dose is taken for the *prior* double-blind, phase 3 efficacy trial so that adjunctive treatment will continue without interruption. It is anticipated that the last dose of the double-blind, phase 3 efficacy trial will be taken the day of the *last scheduled visit* Week 14 visit of Trial 331-10-227 or Trial 331-10-228, (ie, the day of the Screening/Baseline visit for the open-label trial).

Table 3.2.1.1-1, Footnote d:

<sup>d</sup>Throughout Trial 331-10-238, the subject must remain on the same ADT that was assigned in the *prior* double-blind phase 3 trial (ie, Trial 331-10-227 or Trial 331-10-228).

Section 3.2.1.2, ADT, Sentences 1 and 3:

<sup>&</sup>lt;sup>a</sup>Occurs simultaneously with **the** last scheduled visit of **a** double-blind phase 3 brexpiprazole MDD **T**trial-**331-10-227** or **Trial 331-10-228**.

During the Treatment Phase of Trial 331-10-238, subjects will remain on the same assigned open-label ADT from the *prior* double-blind, phase 3 efficacy trial (ie, Trial 331-10-227 or Trial 331-10-228). Numbered ADT bottles to be dispensed to the subject will be assigned by the IVRS or IWRS. The initial dose of ADT for the open-label trial will be the same as the ADT dose taken on the last *scheduled* visit of the prior double-blind *phase 3* trial.

Section 3.2.2.1, Brexpiprazole, Paragraph 2:

Subjects who are unable to tolerate the 0.5 -mg/day dose of brexpiprazole must be withdrawn from the trial. However, subjects whose brexpiprazole dose is decreased to 0.5 mg/day and who demonstrate adequate tolerability at this dose should be rechallenged with a 1 -mg/day dose within approximately 6 to 8 weeks after the dose is decreased to 0.5 mg/day. If tolerability issues arise following the rechallenge, the dose may be decreased again to 0.5 mg/day. Further rechallenge at 1 mg/day may be performed at the investigator's discretion. The dose of brexpiprazole can be *increasedre-escalated* as necessary following a dose decrease at any other dose if, in the investigator's judgment, rechallenge with a higher dose is warranted in order to identify an optimum dose for the subject. Dose adjustments must ultimately be made based upon the clinical judgment of the investigator as it relates to tolerability and therapeutic response.

Section 3.2.2.2, ADT, Paragraph 2:

The Sponsor reserves the right to use a generic equivalent should any marketed antidepressant become unavailable during the course of the trial.

Section 3.3, Trial Population, Paragraphs 1, 2, 4, 5, 6, and 7:

The subject trial population will consist of eligible subjects who, in the investigator's judgment, could potentially benefit from adjunctive treatment with brexpiprazole for MDD *according to the following criteria* who meet one of the following conditions:

- Subjects who participated in Trial 331-10-227 or Trial 331-10-228 will be eligible for the 331-10-238 study if they meet one of the following conditions:
  - Subjects who completed participation in the **D**double-blind **R**randomization
     **P**phase (ie, Week 14 visit of Phase B) in Trial 331-10-227 or Trial 331-10-228 or
  - Subjects who met criteria for a response continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227 or Trial 331-10-228, BUT DID NOT meet criteria for remission (defined as a Montgomery Asberg Depression Rating Scale MADRS Total Score of ≤ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227 or Trial 331-10-228.

- Subjects who participated in another double-blind phase 3 brexpiprazole MDD trial will be eligible for the 331-10-238 study if they have completed the last scheduled visit of the prior double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last *scheduled* visit of the *prior* double-blind *phase 3* trial and must be able to continue therapy without interruption between the double-blind and open label trials. Based on the projected enrollment estimates for the *prior* double-blind phase 3 *brexpiprazole MDD* trials-(ie, Trial 331-10-228), *up to approximately* to 12803,000 subjects may enroll into Trial 331-10-238.

Section 3.4.1, Informed Consent, Paragraph 2, Sentence 3:

The ICF for the open-label trial may be provided to potential candidates for review and discussion toward completion of the *prior* double-blind *phase 3* trial, but the form must not be signed until the day of the Screening/Baseline visit for Trial 331-10-238 (ie, the *the last scheduled visit of the prior double-blind phase 3 trial*\(\text{Week 14 visit of Trial}\) 331-10-227 or Trial 331-10-228).

Table 3.4.2-1, Inclusion Criteria 3, 4, 5, and 6:

| | ANG 11 A |
|---|---|
| | All Subjects |
| <i>3.5</i> 4. | Male and female outpatients 18 to 65 years of age, inclusive, at the time of informed consent for |
| | Trial 331-10-238. |
| 4. <del>65</del> . | Subjects willing to discontinue all prohibited psychotropic medications starting from the time of |
| | signing the ICF and during the trial period (refer to Section 4). |
| | 331-10-227 and 331-10-228 Subjects Only |
| 5. <del>3</del> . | Subjects who, in the opinion of the investigator, could potentially benefit from administration of |
| | brexpiprazole as adjunctive therapy to their antidepressant therapy and who meet one of the |
| | following criteria: |
| | a) Subjects who completed participation in the dDouble-blind rRandomization pPhase (ie, Week |
| | 14 visit of Phase B) in Trial 331-10-227 or Trial 331-10-228 or |
| | b) Subjects who met criteria for a response continued into Phase A+ (were not randomized |
| | into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227 |
| | or Trial 331-10-228, <b>BUT DID NOT</b> meet criteria for remission (defined as a MADRS Total Score |
| | of $\leq$ 10) at the Week 14 visit of Phase A+ in Trial 331-10-227 or Trial 331-10-228. |
| | Eligible Subjects From Other Double-Blind Phase 3 Brexipiprazole MDD Trials |
| 6.4 <del>.</del> | Subjects who completed <del>participation</del> the last scheduled visit of the prior double-blind phase 3 |
| | trial and who in the opinion of the investigator, could potentially benefit from administration of |
| | brexpiprazole as adjunctive therapy to their antidepressant therapy. |

## Section 3.4.3, Exclusion Criteria, Paragraph 1:

Subjects entering the open-label trial at the last *scheduled* visit *of the prior double-blind phase 3 trialof* Trial 331-10-227 or Trial 331-10-228 (ie, Week 14) will be excluded from Trial 331-10-238 if they meet any of the following exclusion criteria.

Table 3.4.3-1, Exclusion Criteria 1, 3, 6, 10, 11, 15, and 20:
## Sex and Reproductive Status

1. Sexually active females of childbearing potential (see Section 5.5) and male subjects who are not practicing two different methods of birth control with their partner during the trial and for 30 days after the last dose of trial medication or who will not remain abstinent during the trial and for 30 days after the last dose. If employing birth control, each couple must use two of the following precautions: vasectomy, tubal ligation (*subject or partner*), vaginal diaphragm, IUD, birth control pill, birth control implant, birth control depot injections, condom, or sponge with spermicide.

#### Administrative

3. Subjects with a major protocol violation during the course of their participation in the *prior* double-blind phase 3 trial-(ie, Trial 331-10-227 or Trial 331-10-228). Minor violations such as occasional visits outside of the acceptable window or a missing blood draw will not exclude a subject from participation in Trial 331-10-238; however, continual lack of compliance with the visit schedule, trial assessments, or treatment regimen in the prior double-blind *phase 3* trial-(ie, Trial 331-10-227 or Trial 331-10-228) would be considered a major violation that would result in exclusion from Trial 331-10-238. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility.

## **Target Disease**

- 6. Subjects with a current need for involuntary commitment or who have been hospitalized during *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228 for the current major depressive episode.
- 10. Subjects receiving new onset psychotherapy (individual, group, marriage, or family therapy) during *the prior double-blind phase 3 trial*Trial 331-10-227 or Trial 331-10-228.

## **Medical History and Concurrent Diseases**

11. Subjects with a response of "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) at entry, **OR**Subjects with a response of "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) at entry, **OR**Subjects with a response of "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) at entry, **OR**Subjects who, in the opinion of the investigator (including consideration of responses on the C-SSRS throughout *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228), present a serious risk of suicide.

Note: "Entry" is defined as the last scheduled visit of the prior double-blind phase 3 trial Week 14 of Trial 331-10-227 or Trial 331-10-228.

- 15. Subjects with IDDM (ie, any subjects using insulin) are excluded. Subjects with non-IDDM may be eligible for the trial if their condition is stable as determined by satisfying **ALL** of the following criteria:
  - Screening/baseline HbA1c < 7.0%, **AND**
  - Screening/baseline fasting glucose must be ≤ 125 mg/dL, AND
  - Subject has been maintained on a stable regimen of oral anti-diabetic medication(s) or diabetes has been well-controlled by diet during *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228, AND
  - Subject has not had any hospitalizations during Trial 331-10-227 or Trial 331-10-228 due to diabetes or complications related to diabetes during the prior double-blind phase 3 trial Trial 331-10-227, or Trial 331-10-228, AND
  - Subject's diabetes is not newly diagnosed during screening/baseline for Trial 331-10-238.

# **Physical and Laboratory Results**

- 20. The following laboratory test and ECG results are exclusionary:
  - 1) Platelets  $\leq 75,000/\text{mm}^3$
  - 2) Hemoglobin  $\leq 9 \text{ g/dL}$
  - 3) Neutrophils, absolute ≤ 1000/mm<sup>3</sup>
  - 4) AST  $> 2 \times ULN$

- 5) ALT  $> 2 \times ULN$
- 6) CPK > 3  $\times$  ULN, unless discussed with and approved by the medical monitor
- 7) Creatinine  $\geq 2 \text{ mg/dL}$
- 8) HbA1c  $\geq 7.0\%$
- 9) Abnormal free T<sub>4</sub>, unless discussed with and approved by the medical monitor. (Note: Free T<sub>4</sub> is measured only if result for TSH is abnormal.)
- 10) QTcF  $\geq$  450 msec

NOTE: In addition, subjects should be excluded if they have any other abnormal laboratory tests, vital sign results, or ECG findings which in the investigator's judgment are medically significant and that would impact the safety of the subject or the interpretation of the trial results. Criteria are provided in Appendix 3, Appendix 4, and Appendix 5 to assist investigators in their assessments of results that may be potentially medically significant, depending on the subject's medical history and clinical presentation. Eligibility should be based on the last available measurement during *the prior double-blind phase 3 trial*Trial 331-10-227 or Trial 331-10-228. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility.

22. Subjects with a history of neuroleptic malignant syndrome (NMS) or serotonin syndrome.

## Section 3.4.3, Exclusion Criteria, Paragraph 2, Sentence 2:

Subjects who do not qualify for the open-label trial at the Screening/Baseline visit may not be rescreened at a later date. If results of clinical laboratory tests from the last *scheduled* visit of the prior double-blind *phase 3* trial (ie, Week 14 of Trial 331-10-227 or Trial 331-10-228) are not available to assess eligibility, the assessment for the affected criteria should be based on the last available measurement during the respective double-blind trial.

## Section 3.6, Trial Procedures, Sentence 1:

The duration of this trial from first subject enrolled to last subject completed is estimated to be approximately 6330 months, of which approximately 5117 months are allotted for rollover of subjects from the *prior* double-blind phase 3 *brexpiprazole MDD* trials-(ie, Trial 331-10-227 or Trial 331-10-228).

| Γable 3.6-1 Schedule of Assessments | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>A</b> | Screening/ | | Open-Label Treatment Phase Visit Week (± 2 days) | | | | | | | Follow-up <sup>c</sup> | | | |
| Assessment | Baseline <sup>a</sup> | 1 | 2 | 4 | 8 | 14 | 20 | 26 | 32 | 38 | 44 | <b>52/ET</b> <sup>b</sup> | 30 (+2) days |
| ENTRANCE CRITERIA | | | | • | • | | | | | • | | | |
| Informed consent d | X | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | | | | | |
| Medical history | X <sup>e</sup> | | | | | | | | | | | | |
| EFFICACY | • | | | • | • | | | | • | • | • | | |
| CGI-S | $X^{\mathbf{f}}$ | X | X | X | X | X | X | X | X | X | X | X | |
| CGI-I <sup>gf</sup> | | X | X | X | X | X | X | X | X | X | X | X | |
| SDS | $X^{\mathbf{f}}$ | | | | X | | | X | | | | X | |
| IDS-SR | X <sup>fq</sup> | | | | X | X | X | X | | X | | X | |
| SAFETY | | | | | | | | | | | | | |
| Physical examination | $X^{\mathbf{f}}$ | | | | X | | | X | | | | X | |
| Waist circumference | X <sup>f</sup> | | | | X | X | X | X | X | X | X | X | |
| Vital signs hg | $X^{\mathbf{f}}$ | X | X | X | X | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>ih</sup> | X <sup>f</sup> | X | | X | X | X | | X | | X | | X | |
| Clinical laboratory tests <sup>ji</sup> | X <sup>f,kj</sup> | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | $X^{lk}$ | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | | X <sup>1</sup> k | |
| ACTH, cortisol, and HbA1c | X <sup>m</sup> | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | $X^{lk}$ | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | | $X^{\mathbf{l}k}$ | | $X^{\mathbf{i}k}$ | |
| Drug screen/blood alcohol** | X <sup>f</sup> | X | | X | X | X | | X | | X | | X | |
| Urine pregnancy test (WOCBP only) <sup>6m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| SAS | X | X | X | X | X | X | X | X | X | X | X | X | |
| AIMS | X <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | |
| BARS | X <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | |
| C-SSRS <sup>pn</sup> | $X^{\mathbf{f}}$ | X | X | X | X | X | X | X | X | X | X | X | |
| MSFQ | X <sup>f</sup> | X | X | | X | | | X | | | | X | |

| Table 3.6-1 Schedule of Assessments | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Screening/ Open-Label Treatment Phase Visit Week (± 2 day | | | | | | ± 2 days | ys) | | Follow-up <sup>c</sup> | | | | |
| Assessment | Baseline <sup>a</sup> | 1 | 2 | 4 | 8 | 14 | 20 | 26 | 32 | 38 | 44 | <b>52/ET</b> <sup>b</sup> | 30 (+2) days |
| Adverse events | X <sup>qo</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications **p | X | X | X | X | X | X | X | X | X | X | X | X | X |
| OTHER | | | | | | | | | | | | | |
| Dose adjustments sq | | X | X | X | X | X | X | X | X | X | X | | |
| RUF <sup>tr</sup> | X | | | | X | | | X | | | | X | |
| Register visit in IVRS/IWRS *** | X | X | X | X | X | X | X | X | X | X | X | X | |
| IMP dispensing | X | X | X | X | X | X | X | X | X | X | X | | |
| IMP accountability | | X | X | X | X | X | X | X | X | X | X | X | |

IVRS = interactive voice response system; IWRS = interactive web response system; WOCBP = women of childbearing potential.

<sup>&</sup>lt;sup>a</sup>Screening for Trial 331-10-238 occurs simultaneously with Baseline at the *last scheduled visit of the prior double-blind trial*<del>Week 14 visit of Trial 331-10-228. All assessments listed under screening need to be performed at Screening/Baseline of Trial 331-10-238; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.</del>

<sup>&</sup>lt;sup>b</sup>If a subject discontinues prematurely before Week 52, procedures noted for Week 52 must be completed at the early termination (ET) visit.

<sup>&</sup>lt;sup>c</sup>Consists of telephone contact or clinic visit (investigator's discretion) for evaluation of safety and applies to all subjects (completers and early withdrawals).

d Informed consent for Trial 331-10-238 will occur at Screening/Baseline and must be obtained before any trial-related procedures specific to the open-label trial are performed.

<sup>&</sup>lt;sup>e</sup>Update, if necessary.

f Screening/Baseline value will be obtained from the Week 14 visit of Trial 331-10-227 or Trial 331-10-228.

Improvement should be based on the subject's status at the last *scheduled* visit of the *prior* double-blind phase 3 trial-(ie, the Week 14 visit of Trial 331-10-227 or Trial 331-10-228).

hg Vital signs include body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Blood pressure and heart rate will be measured in the following order: supine, sitting, and standing after the subject has been in each position for at least 3 minutes. Vital signs scheduled for the same visit as blood samples are to be completed before blood is drawn.

Standard 12-lead ECGs will be performed after the subject has been supine and at rest for ≥ 5 minutes prior to the ECG. A central ECG service will be utilized to review all ECGs in order to standardize interpretations for the safety analysis. In addition, ECG results will be evaluated at the investigational site to monitor safety during the trial. Subjects will be enrolled in Trial 331-10-238 based on the screening/baseline ECG results from the trial site. If the

- screening/baseline ECG results from the central reader (ie, Week 14 visit of Trial 331-10-227 or Trial 331-10-228the last scheduled visit of the prior double-blind phase 3 trial), when available, indicate a QTcF  $\geq$  450 msec at screening/baseline, the investigator must contact the medical monitor to discuss the subject's continued participation in the trial. ECGs scheduled for the same visit as blood samples are to be completed before blood is drawn.
- ji Includes hematology (including PT, aPTT, and INR), serum chemistry (including prolactin and TSH, with reflex to free thyroxine [T4] if the result for TSH is abnormal), and urinalysis.
- kkj Subjects must be fasting for a minimum of 8 hours prior to blood draws for screening/baseline laboratory assessments (ie, Week 14 visit of Trial 331-10-227 and Trial 331-10-228the last scheduled visit of the prior double-blind phase 3 trial).
- Clinical laboratory tests should be drawn fasting, if possible, but must be drawn after a minimum 8-hour fast at Week 52/ET. Vital sign and ECG assessments should be completed before any blood samples are collected.
- <sup>m</sup>A fasting blood sample for analysis of ACTH, cortisol, and HbA1c must be drawn at Screening/Baseline from subjects entering Trial 331–10-238 after completing Phase A+ of Trial 331–10-227 or Trial 331–10-228. This is not required for subjects entering Trial 331–10-238 from Phase B of Trial 331–10-227 or Trial 331–10-228 because the screening/baseline values will be obtained from the last visit of the double-blind protocols.
- A urine drug screen and a blood alcohol test are required at the designated times, but either or both can be conducted at any time during the trial at the discretion of the investigator.
- All positive urine pregnancy test results must be confirmed by a serum test. Subjects with a positive serum pregnancy test result at Screening/Baseline must not be enrolled in Trial 331-10-238 and subjects with a positive serum pregnancy test result during the trial must discontinue treatment and be withdrawn from the trial. Pregnancy tests can be performed at any point during the trial if pregnancy is suspected.
- pn. "Since Last Visit" C-SSRS form.
- **qro** AE recording will begin with the signing of the ICF for Trial 331-10-238.
- All prescription and non-prescription medications taken during the trial will be recorded as concomitant medications. Details of prohibited and restricted medications are provided in Section 4.
- Adjustments to the dose of brexpiprazole or ADT are permitted to optimize efficacy and tolerability as described in Section 3.2. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). At least 5 days must elapse between dose increases for brexpiprazole and ADT. An interval of at least 5 days between dose adjustments is also recommended for dose decreases; however, the investigator may decrease the dose of brexpiprazole or ADT as needed for tolerability according to the rules described in Section 3.2.2. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole or ADT (increases or decreases) are required between scheduled visits. All eligible subjects entering from prior double-blind phase 3 brexpiprazole MDD trials must be able to continue therapy without interruption between the double-blind and open label trials.
- <sup>rt</sup>Baseline RUF is completed at Screening/Baseline for all subjects. The Follow-up RUF is completed at all other visits.
- sumant The IVRS/IWRS will be accessed at unscheduled visits if new blister cards are dispensed for dose adjustment of brexpiprazole.

## Section 3.6.1.1, Screening/Baseline, Paragraph 1 and bulleted list:

Subjects entering Trial 331-10-238 must sign the ICF for the open-label trial before any procedures specific to Trial 331-10-238 can be performed. Subjects will retain the same subject identification (Subject ID) number assigned in the *prior* double-blind phase 3 trial (ie, Trial 331-10-227 or Trial 331-10-228). Screening/baseline values will be derived from the last visit of the double-blind phase 3 trial (ie, Week 14 visit of Trial 331-10-227 or Trial 331-10-228) for the following assessments: CGI-S, SDS, IDS-SR, MSFQ, SAS, AIMS, BARS, C-SSRS, physical examination, waist circumference, vital signs, ECG, clinical laboratory tests (except for ACTH, cortisol, and HbA1c for some subjects), urine drug screen, blood alcohol, and urine pregnancy test. The only additional following procedures need to be performed at Screening/Baseline of Trial 331-10-238the open-label trial are as follows:; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.

- Inclusion/exclusion criteria for Trial 331-10-238 will be reviewed to assure the subject's eligibility.
- Medical history will be updated, if necessary, using information from the prior double-blind phase 3 trial.
- Subjects will submit to a physical examination and assessments of waist circumference, vital signs, and ECG.
- The investigator (or qualified designee) will administer any scale (ie, CGI-I and CGI-S).
- Subjects will complete any Baseline instrument (ie, SDS, IDS-SR, and MSFQ).
- An adequately trained and experienced clinician will administer any EPS scale (ie, SAS, AIMS, and BARS).
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Concomitant medications will be reviewed to assure that the subject is not receiving any prohibited medications.
- Subjects will complete the Baseline RUF.
- For subjects entering Trial 331-10-238 after completing the last scheduled visit of the prior double-blind phase 3 trial Phase A+ of Trial 331-10-227 or Trial 331-10-228, a fasting blood sample will be drawn for analysis of any clinical laboratory parameter (ie, the clinical laboratory parameters specified in Table 3.6.2.1-1) that was not analyzed at the last scheduled visit of the prior double-blind phase 3 trial ACTH, cortisol, and HbA1c to obtain screening/baseline values for these parameters. For all other, the screening/baseline values for these parameters will be obtained from the last visit of the double-blind trial.

- AE recording will begin with the signing of the ICF for Trial 331-10-238.
- Trial personnel will call the interactive voice response system (IVRS) or access the interactive web response system (IWRS) to register the visit and to obtain blister card and ADT bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed. Treatment will begin with brexpiprazole 0.5 mg/day for 1 week. The ADT will be the same as the one taken during the *prior* double-blind phase 3 trial-(ie, Trial 331-10-227 or Trial 331-10-228). The dose of ADT should not be changed at this time.

Section 3.6.2.1, Clinical Laboratory Tests, Paragraph 1, Sentences 1 and 3:

As it is unlikely that the final laboratory test results from *the last scheduled visit of the prior* double-blind phase 3 trial (ie, Week 14 of Trial 331-10-227 and Trial 331-10-228) will be available at the time of enrollment in Trial 331-10-238, the investigator is to review the subject's most recent laboratory test results from the *prior* double-blind *phase 3* trial (ie, Trial 331-10-227 or Trial 331-10-228) for compliance with the exclusion criteria and the presence of abnormal laboratory test results that, in the investigator's judgment, are medically significant and would impact the safety of the subject or the interpretation of the trial results. Subjects meeting any of these criteria will be excluded from Trial 331-10-238. Appendix 4 is included to assist investigators in their assessments of results that may be potentially medically significant, depending on the subject's medical history and clinical presentation. If one or more results from the screening/baseline sample are clinically significant and/or exclusionary when the results from the last *scheduled* visit of the *prior* double-blind *phase 3* trial become available, the test(s) should be repeated.

Section 3.6.2.2.1, Physical Examination, Paragraph 1, Sentences 1 and 3:

The complete physical examination at the last *scheduled* visit of the *prior* double-blind phase 3 trial (ie, Week 14 visit of Trial 331-10-228) will serve as the screening/baseline physical examination for the current protocol. A complete physical examination will consist of a review of the following body systems: HEENT, thorax, abdomen, urogenital, extremities, neurological, and skin and mucosae. Repeat measurement of height is not required during Trial 331-10-238 if a *Ss*creening/*Bb*aseline value is available from the last *scheduled* visit of the *prior* double-blind phase 3 trial.

Section 3.6.2.2.1, Physical Examination, Paragraph 5, Sentences 1, 3, and 4:

The principal investigator or his/her appointed designee is primarily responsible to perform the physical exam*ination*. If the appointed designee is to perform the physical exam*ination*, he/she must be permitted by local regulations and his/her name must be included on the FDA Form 1572. Whenever possible, the same individual should perform all physical exam*inations*. Any condition present at the post-treatment physical exam*ination* that was not present at the screening/baseline exam*ination* should be documented as an AE and followed to a satisfactory conclusion.

## Section 3.6.2.4.4

Suicidality will be monitored during the trial using the C-SSRS. Subjects completed the "Baseline/Screening" C-SSRS form at the beginning of the *prior* double-blind phase 3 trial (ie, Trial 331-10-227 or Trial 331-10-228); therefore, only the "Since Last Visit" C-SSRS form will be used in Trial 331-10-238. A copy of the "Since Last Visit" C-SSRS form is provided in Appendix 13.

Section 3.6.3.2, Clinical Global Impression - Improvement Scale (CGI-I), Sentence 2

The efficacy of trial treatment will be rated for each subject using the CGI-I.26 The rater or investigator will rate the subject's total improvement whether or not it is due entirely to drug treatment. All responses will be compared to the subject's condition at Screening/Baseline (ie, Week 14 last scheduled visit of the prior double-blind phase 3 trialTrial 331-10-227 or Trial 331-10-228). Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. A sample of the CGI-I is provided in Appendix 7.

Section 3.6.3.3.3, Resource Utilization Form (RUF), Sentences 2 and 3:

The RUF is a self-report tool designed to collect information regarding the extent of medical care sought by subjects while participating in the trial (Appendix 15). The number of hospitalizations and days of hospitalization within the past 12 months will be collected on the Baseline Form at Screening/Baseline, including any hospitalizations that may have occurred during the subject's participation in *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228. The number of visits to various practitioners for mental health and other reasons within the 3 months prior to Screening/Baseline (excluding any visits from *the prior* 

*double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228) will be collected on the Baseline Form and the number of such visits occurring during the trial (excluding visits related to the trial) will be collected on the Follow-up Form at Weeks 8, 26, and 52/ET.

Section 3.8, Screen Failures, Sentence 3:

A screen failure subject is one from whom informed consent is obtained and is documented in writing (ie, subject signs an ICF), but who is not started on treatment, whether through randomization or open assignment. For the purposes of Trial 331-10-238, treatment begins with the first dose of open-label brexpiprazole in the Treatment Phase. Subjects who do not qualify for Trial 331-10-238 at the last *scheduled* visit of the *prior* double-blind phase 3 trial (ie, Week 14 of Trial 331-10-227 or Trial 331-10-228) may not be rescreened.

Section 4.1, Prohibited Medications, Sentence 1:

Concomitant medications taken by subjects who are rolling over into Trial 331-10-238 from one of thea prior double-blind phase 3 trials (ie, Trial 331-10-227 or Trial 331-10-228) should be reviewed for the prohibited medications listed in Table 4.1-1.

Section 4.2.1, Restricted Therapies and Precautions, Paragraph 4, Sentence 1:

ECT was prohibited during the *prior* double-blind phase 3 trials (ie, Trial 331-10-227 and Trial 331-10-228) and is also prohibited for the duration of Trial 331-10-238.

Section 4.2.2.2, Restrictions, Paragraph 1:

Subjects may only receive psychotherapy (eg, individual, group, marriage, or family therapy) if they initiated the therapy at least 42 days before enrollment in **one of** the *prior* double-blind phase 3 trials (ie, Trial 331-10-227 or Trial 331-10-228), participated in the therapy regularly during the *prior* double-blind phase 3 trial, and commit to maintain their participation during the course of Trial 331-10-238, or unless permission is obtained from the medical monitor.

Section 5.4, Potential Hy's Law Cases:

For a subject that experiences an elevation in AST or ALT that is  $\geq 3$  times the upper normal limit-or whose levels increase  $\geq 3$  times their initial screening value, a total bilirubin level should also be evaluated. If the total bilirubin is  $\geq 2$  times the upper normal limit or  $\geq 2$  times their screening value, confirmatory repeat laboratory samples should be drawn within 48 to 72 hours of the initial draw. If these values are confirmed, trial personnel will complete an IRE form with all values listed and also report as an AE on the eCRFs. Please note: If the subject was enrolled into the trial with non-exclusionary elevated transaminase levels at baseline, please discuss any potential drug-induced liver injury events with the Medical Monitor.

Section 5.5, Pregnancy:

WOCBP and men who are sexually active must use an effective method of birth control during the course of the trial and for at least 30 days after the last dose in a manner such that risk of failure is minimized. Unless the subject is sterile (ie, women who have had an oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months; or men who have had orchidectomy) or remains abstinent, two of the following precautions must be used: vasectomy *or*<sub>5</sub> tubal ligation (*subject and partner*), vaginal diaphragm, intrauterine device, birth control pills, birth control depot injection, birth control implant, condom or sponge with spermicide. Any single method of birth control, including vasectomy and tubal ligation, may fail, leading to pregnancy.

Section 7.2, Sample Size:

The sample size is not based on statistical power considerations. The trial population will be derived from eligible subjects from the *prior* double-blind phase 3 *brexpiprazole MDD* trials (ie, Trial 331-10-227 and Trial 331-10-228). Therefore, the number of eligible subjects will be limited by the number of subjects enrolled into these protocols. Based on the projected enrollment estimates for the *prior* double-blind phase 3 trials (ie, Trial 331-10-227 and Trial 331-10-228), *up to approximately* up to 3,0001280 subjects may enroll into Trial 331-10-238.

Section 8.1, Packaging and Labeling, Paragraph 3, Sentence 2:

ADTs will be supplied as bulk drug in commercial packaging (eg, bottles) with an ancillary trial-specific label that will be positioned such that it will not obscure the original commercial label. *The sponsor reserves the right to use a generic equivalent, should any marketed antidepressant become unavailable during the course of the trial.* 

Appendix 1, Names of Sponsor Personnel:



| | п |
|-----------------|---|
| LOW | ı |
| <del>l'ax</del> | ŀ |

Appendix 2, Institutions Concerned with the Trial, Safety Reporting:

| Country | Safety Fax Line |
|---------------------|-----------------|
| United States | |
| Canada | |
| Czech Republic | |
| France | |
| Germany | |
| Hungary | |
| Poland | |
| Romania | |
| Russia | |
| Slovakia | |
| Ukraine | _ |
| All other countries | |

Appendix 7, Clinical Global Impression - Improvement Scale (CGI-I), Sentence 2:

Rate total improvement whether or not in your judgment it is due entirely to drug treatment. Compared to his/her condition at the last *scheduled* visit of *the prior double-blind phase 3 trial* Trial 331-10-227 or Trial 331-10-228 (ie, prior to enrollment into Trial 331-10-238), how much has patient changed?

## ADDITIONAL RISK TO THE SUBJECT:

There is no additional risk to the subjects as a result of this protocol amendment.

Protocol 331-10-238

**Amendment Number:** 3

Issue Date: 11 Apr 2014

## **PURPOSE:**

The sponsor has determined the need for a third formal amendment to the original protocol. Due to a well-established safety profile in the completed double-blind and long-term Phase 2 and Phase 3 trials the study duration has been reduced from 52 weeks to 26 weeks and the number of assessments has been decreased. In addition, administrative clarifications were made, including changes to text to enhance readability and consistency and correct typographical errors. The purpose of amending Protocol 331-10-238, issued on 16 Nov 2012 (amendment 2), was to:

- reduce the trial duration from 52 weeks to 26 weeks.
- reduce the number of visits to match the reduction in trial duration.
- minimize safety assessments performed at each visit.
- reduce the safety scale administration performed at each visit.
- reduce the efficacy scale administration performed at each visit.
- make administrative changes.

## **BACKGROUND:**

Due to a well-established safety profile in the completed double-blind and long-term Phase 2 and Phase 3 trials the study duration has been reduced from 52 weeks to 26 weeks and the number of assessments has been decreased. In addition, administrative clarifications were made, including changes to text to enhance readability and consistency and correct typographical errors.

## **MODIFICATIONS TO PROTOCOL:**

## **General Revisions:**

- Changes made to Protocol 331-10-238 in this third amendment are as outlined above.
- All the references to Week 52 were changed to Week 26. The word "study" was replaced by "trial" throughout the document.
- All visits and assessments from Week 26 to Week 52 were removed.
- Reference to Trial 331-13-214 was added wherever Trial 331-10-227 and Trial 331-10-228 were referred.
- Sections 8.5 to 8.5.4 (Reporting of Product Quality Complaints) were added.

# **General Revisions:**

Changes made to Protocol 331-10-238 in this third amendment are as outlined above. Changes by section are provided below.

# **Revisions by Protocol Section:**

| Location | Current Text | Revised Text |
|---|---|---|
| Title Page | Phone Fax E-mail | Phone Fax E-mail: |
| Synopsis: Trial Design | This is a multicenter, 52-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive brexpiprazole in depressed adults on concurrent antidepressant therapy (ADT). Visits will occur at the end of | This is a multicenter, 26-week, open-label trial designed to assess the long-term safety, tolerability, and efficacy of adjunctive brexpiprazole in depressed adults on concurrent antidepressant therapy (ADT). The trial will be conducted on an outpatient basis. Enrollment into the trial will be |

Weeks 1, 2, 4, 8, 14, 20, 26, 32, 38, 44, and 52. All subjects will receive up to 52 weeks of openlabel treatment in Trial 331-10-238.

drawn from eligible subjects who have completed the last scheduled visit of a double-blind, phase 3 brexpiprazole MDD trial and who, in the investigator's judgment, could potentially benefit from adjunctive treatment with oral brexpiprazole for MDD.

The original 52 week open-label trial design has been modified in this Amendment 3 to shorten the duration of the trial to 26 weeks; ongoing subjects who have not reached their Week 26 visit will be re-consented and will follow Amendment 3 schedule of assessments. Ongoing subjects who have already completed their Week 26 visit at the time of Amendment 3 will follow Amendment 3 week 26/ET schedule of assessments at their next scheduled visit

Visits will occur at the end of Weeks 1, 2, 4, 8, 14, 20 and 26. All subjects will receive up to 26 weeks of open-label treatment in Trial 331-10-238.

| <b>Synopsis: Trial Duration</b> | The duration of this trial from | The duration of this trial from |
|---|---|---|
| | first subject enrolled to last | first subject enrolled to last |
| | subject completed is estimated to | subject completed is estimated to |
| | be approximately 63 months, of | be approximately 57 months, of |
| | which approximately 51 months | which approximately 51 months |
| | are allotted for rollover of | are allotted for rollover of |
| | subjects from the prior double- | subjects from the prior double- |
| | blind phase 3 brexpiprazole MDD | blind phase 3 brexpiprazole MDD |
| | trials. Individual participation for | trials. Individual participation for |
| | subjects who complete the trial | subjects who complete the trial |
| | without early withdrawal will be | without early withdrawal will be |
| | approximately 56 weeks (52 | approximately 30 weeks (26 |
| | weeks of treatment and 30-day | weeks of treatment and 30-day |
| | follow-up). | follow-up). |
| Section 3.1: | Visits will occur at the end of | Visits will occur at the end of |
| Type/Design of Trial | Weeks 1, 2, 4, 8, 14, 20, 26, 32, | Weeks 1, 2, 4, 8, 14, 20, and 26. |
| | 38, 44, and 52. All subjects will | All subjects will receive up to 26 |
| | receive up to 52 weeks of open- | weeks of open-label treatment in |
| | label treatment in Trial 331-10- | Trial 331-10-238 and follow the |
| | 238 and follow the schedule of | schedule of assessments |
| | assessments described in Table | described in Table 3.6-1. |
| | 3.6-1. | Car Daviand Figure 444 and 4 |
| | Sac Cumment Figure at the sulf-f | See Revised Figure at the end of |
| | See Current Figure at the end of the table. | the table. |
| | the table. | Figure 3.1-1 Trial Design |
| | Figure 3.1-1 Trial Design | Schematic |

| | Schematic | |
|---|---|---|
| | See current Table 3.2.1.1-1 | See revised Table 3.2.1.1-1 |
| | Dosing Schedule for | Dosing Schedule for |
| | Brexpiprazole at the end of this | Brexpiprazole at the end of this |
| | table. | table. |
| | See curent Table 10.2-1 Schedule | See revised Table 10.2-1 |
| | of Assessments at the end of this | Schedule of Assessments at |
| | table | the end of this table. |
| | | the end of this table. |
| Section 3.3: Trial | The trial population will consist | The trial population will consist |
| Population | of eligible subjects who, in the | of eligible subjects who, in the |
| | investigator's judgment, could | investigator's judgment, could |
| | potentially benefit from | potentially benefit from |
| | adjunctive treatment with | adjunctive treatment with |
| | brexpiprazole for MDD | brexpiprazole for MDD |
| | according to the following | according to the following |
| | criteria: | criteria: |
| | Subjects who | Subjects who |
| | participated in Trial 331-10-227, | participated in Trial 331-10-227, |
| | Trial 331-10-228 or Trial 331 13 | Trial 331-10-228 or Trial 331 13 |
| | 214 will be eligible for Trial 331- | 214 will be eligible for Trial 331- |
| | 10-238 if they meet one of the | 10-238 if they meet one of the |
| | following conditions: | following conditions: |
| | Subjects who completed | Subjects who completed |
| | participation in the double-blind | participation in the double-blind |
| | randomization phase (ie, Week | randomization phase (ie, Week |
| | 14 visit of phase B) in Trial 331- | 14 visit of phase B) in Trial 331- |
| | 10-227, Trial 331-10-228 or | 10-227, Trial 331-10-228 or |

Trial 331 13 214 or

Subjects who continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214, BUT DID NOT meet criteria for remission (defined as a MADRS Total Score of  $\leq$  10) at the Week 14 visit of Phase A+ in Trial 331 10 227, Trial 331-10-228 or Trial 331-13-214.

- Subjects who participated in a double-blind phase 3 brexpiprazole MDD trial will be eligible for the 331-10-238 trial if they have completed the last scheduled visit of the double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last scheduled visit of the prior double-blind phase 3 trial and must be able to continue therapy without interruption between the double-blind and open label

Trial 331 13 214 or

Subjects who continued into Phase A+ (were not randomized into Phase B) at the end of prospective treatment (ie, Week 8 visit of Phase A) in Trial 331-10-227, Trial 331-10-228 or Trial 331-13-214, BUT DID NOT meet criteria for remission (defined as a MADRS Total Score of  $\leq$  10) at the Week 14 visit of Phase A+ in Trial 331 10 227, Trial 331-10-228 or Trial 331-13-214.

- Subjects who participated in a double-blind phase 3 brexpiprazole MDD trial will be eligible for the 331-10-238 trial if they have completed the last scheduled visit of the double-blind phase 3 trial.
- Subjects must qualify for Trial 331-10-238 at the last scheduled visit of the prior double-blind phase 3 trial and must be able to continue therapy without interruption between the double-blind and open label

| | trials. Based on the projected | trials. Based on the projected |
|---|---|---|
| | enrollment estimates for the prior | enrollment estimates for the prior |
| | double-blind phase 3 | double-blind phase 3 |
| | brexpiprazole MDD trials, up to | brexpiprazole MDD trials, up to |
| | approximately 3,000 subjects | approximately 3,000 subjects |
| | may enroll into Trial 331-10-238. | may enroll into Trial 331-10-238. |
| Section 3.4.2: Inclusion | Subjects willing to discontinue all | Subjects willing to discontinue all |
| Criteria | prohibited psychotropic | prohibited psychotropic |
| | medications starting from the | medications starting from the |
| | time of signing the ICF and | time of signing the ICF and |
| | during the trial period (refer to | during the trial period (refer to |
| | Section 4). | Section 4). |
| | 331-10-227 331-10-228 Subjects | 331-10-227 331-10-228 and 331- |
| | Only. | 13-214 Subjects Only. |
| Section 3.4.3: Exclusion | 5. Subjects who have had an | 5. Subjects who have had an |
| Criteria. | inadequate response to ECT at | inadequate response to ECT at |
| | any time in the past or who have | any time in the past or who have |
| | had a vagus nerve stimulation or | had a vagus nerve stimulation or |
| | deep brain stimulation device | deep brain stimulation device |
| | implanted for management of | implanted at any time for |
| | treatment-resistant depression. | management of treatment- |
| | | resistant depression. Subjects |
| | | who have had Transcranial |
| | | Magnetic Stimulation during the |
| | | current major depressive episode. |
| | | 15. Continuation of subjects |
| | | excluded based on abnormal test |
| | | results from the |

| | 20. Eligibility should be based on the last available measurement during the prior double-blind phase 3 trial. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility. | screening/baseline visit should be discussed with the medical monitor, if in the investigator's judgement, the subject is a suitable candidate for the trial. 20. Eligibility should be based on the Screening/baseline laboratory test and ECG results. The medical monitor should be contacted if the investigator is unsure of a subject's eligibility. Continuation of subjects excluded based on abnormal test and ECG results should be discussed with the medical monitor, if in the investigator's judgement, the subject is a suitable candidate for the trial. |
|---|---|---|
| Section 3.5.2.2: Safety | Mean change from baseline will | Mean change from baseline will |
| Variables | be calculated for coagulation parameters (prothrombin time | be calculated for coagulation parameters (prothrombin time |
| | [PT], activated partial | [PT], activated partial |
| | thromboplastin time [aPTT], and | thromboplastin time [aPTT], and |
| | International Normalized Ratio [INR]), glycosylated hemoglobin | International Normalized Ratio [INR]), glycosylated hemoglobin |

| | (HbA1c), cortisol, | (HbA1c), thyroid-stimulating |
|---|---|---|
| | adrenocorticotropic hormone | hormone (TSH), waist |
| | (ACTH), thyroid-stimulating | circumference, and body mass |
| | hormone (TSH), waist | index (BMI; derived |
| | circumference, and body mass | programmatically from body |
| | index (BMI; derived | weight and height |
| | programmatically from body | measurements). |
| | weight and height | |
| | measurements). | |
| Section 3.6: Trial | The duration of this trial from | The duration of this trial from |
| Procedures | first subject enrolled to last | first subject enrolled to last |
| | subject completed is estimated to | subject completed is estimated to |
| | be approximately 63 months, of | be approximately 57 months, of |
| | which approximately 51 months | which approximately 51 months |
| | are allotted for rollover of | are allotted for rollover of |
| | subjects from prior double-blind | subjects from prior double-blind |
| | phase 3 brexpiprazole MDD | phase 3 brexpiprazole MDD |
| | trials. Individual participation for | trials. Individual participation for |
| | subjects who complete the trial | subjects who complete the trial |
| | without early withdrawal will be | without early withdrawal will be |
| | approximately 56 weeks (52 | approximately 30 weeks (26 |
| | weeks of treatment and 30-day | weeks of treatment and 30-day |
| | follow-up). | follow-up). |
| Section 3.6.1: | The investigator (or qualified | The investigator (or qualified |
| Screening/Baseline | designee) will administer any scale (ie,the CGI-I and CGI S). | designee) will administer the CGI-S and CGI. |
| Section 3.6.1.2: Week 1 | The investigator (or qualified designee) will administer the | The investigator (or qualified designee) will administer the |

#### CGI-S and CGI-I.

- An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- The subject will complete the MSFQ.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry,

#### CGI-S.

- An adequately trained and experienced clinician will administer the SAS AIMS, and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- Women of childbearing potential (WOCBP) will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum

- including prolactin, HbA1c, ACTH, cortisol, and TSH, with reflex to free thyroxine [T<sub>4</sub>] if the result for TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- Women of childbearing potential (WOCBP) will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The dose of brexpiprazole will be increased to 1 mg/day. Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit. It is recommended that the dose of ADT not be changed

- pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The dose of brexpiprazole will be increased to 1 mg/day. Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

| | • | while the dose of brexpiprazole is being optimized. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject. AEs and concomitant medications will be recorded. | | |
|---|---|---|---|---|
| Section 3.6.1.3: Week 2 | • | The investigator (or qualified designee) will administer the CGI-S and CGI-I. | • | The investigator (or qualified designee) will administer the CGI-S. |
| | • | An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS. | • | An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS. |
| | • | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. | • | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. |
| | • | The subject will complete the MSFQ. | • | Vital sign measurements (body weight, body |
| | • | Vital sign measurements<br>(body weight, body<br>temperature, blood pressure,<br>and heart rate) will be<br>recorded. Blood pressure<br>and heart rate are to be<br>measured in the following<br>order: supine, sitting, and | | temperature, blood pressure,<br>and heart rate) will be<br>recorded. Blood pressure and<br>heart rate are to be measured<br>in the following order:<br>supine, sitting, and standing<br>after the subject has been in<br>each position at least 3 |

- standing after the subject has been in each position at least 3 minutes.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized. Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain

- minutes.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
  - The investigator will adjust the dose of brexpiprazole as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized. Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-labelbrexpiprazole and

| | • | blister card and bottle<br>number assignments. The<br>assigned open-label<br>brexpiprazole and ADT will<br>be dispensed to the subject.<br>AEs and concomitant<br>medications will be recorded. | • | ADT will be dispensed to the subject. AEs and concomitant medications will be recorded. |
|---|---|---|---|---|
| Section 3.6.1.4: Week 4 | • | The investigator (or qualified designee) will administer the CGI-S and CGI-I. | • | The investigator (or qualified designee) will administer the CGI-S. |
| | • | An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS. | • | An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS. |
| | • | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. | • | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. |
| | • | Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn. | • | Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn. |
| | • | A standard 12-lead ECG will<br>be performed after the<br>subject has been supine and<br>at rest for at least 5 minutes. | • | Samples will be obtained for blood alcohol testing. Urine will be collected for urine screen(s) for drugs of |

- The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, ACTH, cortisol, and TSH, with reflex to free T4 if the result for TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary as described in

- abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary as described in Section 3.2 to achieve optimal efficacy and tolerability. If necessary, the dose of ADT can be changed after the Week 4 visit, but not at the same visit as a change to the dose of brexpiprazole (see Section 3.2.2.2). Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned

| | | Section 3.2 to achieve optimal efficacy and tolerability. If necessary, the dose of ADT can be changed after the Week 4 visit, but not at the same visit as a change to the dose of brexpiprazole (see Section 3.2.2.2). Any subject unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial. Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject. AEs and concomitant | • | open-label brexpiprazole and ADT will be dispensed to the subject. AEs and concomitant medications will be recorded. |
|---|---|---|---|---|
| | | medications will be recorded. | | |
| Section 3.6.1.5: Week 8 | • | The investigator (or qualified designee) will administer the CGI-S and CGI-I. | • | The investigator (or qualified designee) will administer the CGI-S. |
| | • | An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS. | • | An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS. |
| | • | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS | • | Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be |

form.

- The subject will complete the MSFQ, SDS, IDS-SR, and the Follow-up RUF.
- A complete physical examination (including waist circumference) will be performed.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, ACTH, cortisol, and TSH, with reflex to free T4 if TSH

- recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the

- is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle

- IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.

| | number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject. • AEs and concomitant medications will be recorded. | |
|---|---|---|
| Section 3.6.1.6: | Section 3.6.1.6: Long-term | Section 3.6.1.6 Week 14 |
| | Treatment Visits (Weeks 14, 20, | All subjects will attend a visit at |
| | 26, 32, 38, and 44) | Week 14 (± 2 days) where the following evaluations will be performed: |
| | All subjects will attend visits at | |
| | Weeks 14, 20, 26, 32, 38, and 44 | |
| | (± 2 days). The following evaluations will be performed at each visit, unless otherwise | • The investigator (or qualified designee) will administer the CGI-S and CGI-I. |
| | specified: | Waist circumference will be measured. |
| | <ul> <li>The investigator (or qualified designee) will administer the CGI-S and CGI-I.</li> <li>Waist circumference will be</li> </ul> | An adequately trained and experienced clinician will administer the SAS, AIMS, and BARS to assess EPS. |
| • | An adequately trained and | • The subject will complete the IDS-SR and SDS. |
| | experienced clinician will administer the SAS, AIMS, and BARS to assess EPS. | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS |
| | The subject will complete the IDS-SR (except for Weeks | form. |
| | <ul> <li>32 and 44).</li> <li>The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.</li> </ul> | Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured |

- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- WOCBP will be given a
  urine pregnancy test. Any
  positive result must be
  confirmed by a serum
  pregnancy test. WOCBP
  with a positive serum
  pregnancy test result must
  discontinue the IMP and be
  withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter

- in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, and TSH, with reflex to free T4 if the result for TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
   Additional blood alcohol testing may be performed at any other time at the discretion of the investigator.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
   Additional urine drug screens may be performed at any

- dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.
- The following additional evaluations will be performed at Weeks 14, 26, and 38 only:
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, ACTH, cortisol, and TSH, with reflex to free T4 if the result for TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
   Additional blood alcohol

- other time at the discretion of the investigator.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject.
- AEs and concomitant medications will be recorded.
| | testing may be performed at any other time at the discretion of the investigator. • Urine will be collected for urinalysis and urine screen(s) for drugs of abuse. Additional urine drug screens may be performed at any other time at the discretion of the investigator. | |
|---|---|---|
| | The following additional evaluations will be performed at Week 26 only: • A complete physical examination will be performed. | |
| | The subject will complete the MSFQ, SDS, and the Follow-up RUF. | |
| Section 3.6.1.7: Week 20 | Section 3.6.1.7: End of<br>Treatment (Week 52/ET) | Section 3.6.1.7: |
| | Treatment (Week 32/E1) | All subjects will attend a visit at Week 20 (± 2 days) where the following evaluations will be performed: • The investigator (or qualified designee) will administer the CGI-S. |

- An adequately trained and experienced clinician will administer the SAS and BARS to assess EPS.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test. WOCBP with a positive serum pregnancy test result must discontinue the IMP and be withdrawn from the trial.
- Drug accountability will be performed for brexpiprazole and ADT.
- The investigator will adjust the dose of brexpiprazole as necessary within the range of 0.5 to 3 mg daily as described in Section 3.2. If necessary, the dose of ADT can also be adjusted (see

| | | Section 3.2.2.2). Trial personnel will call the IVRS or access the IWRS to register the visit, to enter dose details for brexpiprazole and ADT, and to obtain blister card and bottle number assignments. The assigned open-label brexpiprazole and ADT will be dispensed to the subject. • AEs and concomitant medications will be recorded |
|---|---|---|
| Section 3.6.1.8: End of Treatment (Week 26/ET) | NA | • The Week 26 visit signifies the end of treatment. Therefore, all subjects will undergo a complete evaluation at Week 26 (±2 days). In addition, Week 26 evaluations are to be completed, if possible, for any subject withdrawn from the trial prematurely. Since the original 52 week openlabel trial design has been modified as a part of Amendment 3 to shorten the duration of the trial to 26 weeks; ongoing subjects who have not reached their Week 26 visit will be re-consented and will follow Amendment 3 schedule of assessments. Ongoing subjects who have |

already completed their Week 26 visit at the time Amendment 3 is approved will follow Amendment 3 week 26/ET schedule of assessments at their next scheduled visit. The following activities and assessments will occur at Week 26 (or at the ET visit, if applicable):The investigator (or qualified designee) will administer the CGI-S and CGI-I. An adequately trained and experienced clinician will

- administer the SAS, AIMS, and BARS to assess EPS.
- The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form.
- The subject will complete the MSFQ, SDS, IDS-SR, and the Follow-up RUF.
- A complete physical examination (including waist circumference) will be performed.
- Vital sign measurements (body weight, body temperature, blood pressure, and heart rate) will be recorded. Blood pressure and heart rate are to be measured

- in the following order: supine, sitting, and standing after the subject has been in each position at least 3 minutes. Vital signs are to be completed before any blood is drawn.
- A standard 12-lead ECG will be performed after the subject has been supine and at rest for at least 5 minutes. The ECG is to be completed before any blood is drawn.
- A fasting blood draw will be collected for clinical laboratory tests (hematology, including PT, aPTT, and INR; and serum chemistry, including prolactin, HbA1c, ACTH,cortisol and TSH, with reflex to free T<sub>4</sub> if TSH is abnormal). Vital sign and ECG assessments should be completed before any blood samples are collected.
- Samples will be obtained for blood alcohol testing.
- Urine will be collected for urinalysis and urine screen(s) for drugs of abuse.
- WOCBP will be given a urine pregnancy test. Any positive result must be confirmed by a serum pregnancy test.

| | | <ul> <li>Final drug accountability will be performed.</li> <li>Trial personnel will call the IVRS or access the IWRS to register completion or discontinuation from the trial.</li> <li>AEs and concomitant medications will be recorded.</li> </ul> |
|---|---|---|
| Section 3.6.2.1: Clinical | See the current table at the end of | See the revised table at the end of |
| <b>Laboratory Tests</b> | this table | this table |
| Section 3.6.2.2.1: | Repeat measurement of height is | Repeat measurement of height is |
| Physical Examination | not required during Trial 331-10- | not required during Trial 331-10- |
| | 238 if a Screening/Baseline value | 238 if a Screening/Baseline value |
| | is available from the last | is available from the prior double |
| | scheduled visit of the prior | blind phase 3 trial. |
| | double blind phase 3 trial. | Waist circumference will be measured at Screening/Baseline |
| | Waist circumference will be | |
| | measured at each physical | Week 14 and Week 26/ET. |
| | examination (ie, Weeks 8, 26, and | |
| | 52), and in addition, at Weeks 14, | |
| | 20, 32, 38, and 44. | |
| Section 3.10: Definition | Subjects who cannot be contacted | Subjects who cannot be contacted |
| of Lost to Follow-up | on or before the Week 52 visit | on or before the Week 26 visit |
| | during the treatment period and | during the treatment period and |
| | who do not have a known reason | who do not have a known reason |
| | for discontinuation (eg, withdrew | for discontinuation (eg, withdrew |
| | consent or AE) will be classified | consent or AE) will be classified |
| | as "lost to follow-up" as the | as "lost to follow-up" as the |

| | reason for discontinuation. | reason for discontinuation. The site will make three attempts to contact the subject by telephone and in the event the site is unable to reach the subject by telephone, the site will attempt to contact the |
|---|---|---|
| | | subject via certified mail or an alternative similar method where appropriate. |
| <b>Section 5.1: Definitions</b> | Examples of AEs that are | Examples of AEs that are |
| | considered extrapyramidal | considered extrapyramidal |
| | symptoms include, but are not | symptoms include, but are not |
| | limited to: generalized rigidity, | limited to: generalized rigidity, |
| | hyperkinesia, bradykinesia, | hyperkinesia, dyskinesia, |
| | akinesia, dystonia, hypertonia, | bradykinesia, akinesia, dystonia, |
| | akathisia, tremor, flexed posture, | hypertonia, akathisia, tremor, |
| | involuntary muscle contractions, | <ul> <li>flexed posture, involuntary muscle contractions, athetosis, and chorea.</li> <li>Potential Hy's Law cases (Any increase of AST or ALT ≥ 3 times the upper normal limit with an increase in total bilirubin ≥ 2 times the upper normal limit.</li> </ul> |
| | athetosis, and chorea. | |
| | Potential Hy's Law cases | |
| | (Any increase of AST or ALT ≥ 3 times the upper normal limit or screening value with an increase in total bilirubin ≥ 2 times the upper normal limit or screening value.) | |
| Section 7.1.2: | In order to assess sensitivity of | In order to assess sensitivity of |
| | results due to missing data, two | results due to missing data, two |
| | types of analyses will be | types of analyses will be |
| | performed for analyses by visit: | performed for analyses by visit: |

| | LOCF and OC. The LOCF and | LOCF and OC. The LOCF and |
|---|---|---|
| | OC data sets are defined in | OC data sets are defined in |
| | Section 7.1.1. The OC data set | Section 7.1.1. The OC data set |
| | will be used for analyses at each | will be used for analyses at each |
| | visit and the LOCF data set will | visit and the LOCF data set will |
| | be used for the last visit analyses | be used for the last visit analyses |
| | (ie, Week 26, LOCF). | |
| Section 7.1.4: Secondary | Secondary efficacy endpoints are | Secondary efficacy endpoints are |
| outcome analysis | as follows: | as follows: |
| | 1) Change from baseline in | 1) Change from baseline in |
| | CGI-S score, by trial week and at | CGI-S score, by trial week and at |
| | the last visit (ie, Week 26/ET); | the last visit. |
| | 2) Mean CGI-I score, by | 2) Mean CGI-I score, by |
| | trial week and at the last visit (ie, | trial week and at the last visit. |
| | Week 26/ET); | 3) Change from baseline in |
| | 3) Change from baseline in | SDS score, by trial week and at |
| | SDS score, by trial week and at | the last visit. |
| | the last visit (ie, Week 26/ET); | 4) Change from baseline in |
| | 4) Change from baseline in | IDS-SR Total Score, by trial week |
| | IDS-SR Total Score, by trial | and at the last visit |
| | week and at the last visit (ie, | Descriptive statistics will be |
| | Week 26/ET). | Descriptive statistics will be provided for each endpoint. The |
| | Descriptive statistics will be | analysis will be carried out on the |
| | provided for each endpoint. The | Efficacy Sample. Descriptive |
| | analysis will be carried out on the | statistics will be summarized at |
| | Efficacy Sample. Descriptive | each trial visit using the OC data |
| | statistics will be summarized at | set and at the last visit. |
| | statistics will be summarized at | Set and at the fast visit. |

| | each trial visit using the OC data | trial visit using the OC data |
|---|---|---|
| | set and at the last visit using the | |
| | LOCF data set. | |
| | | Descriptive statistics will be |
| Section 74.5: Other | Descriptive statistics will be | Descriptive statistics will be |
| Safety Data | summarized at each visit using | summarized at each visit using the |
| | the OC data set and at the last OC data set and at the last visit | |
| | visit (Week 26/ET) using the using the LOCF data set. | |
| | LOCF data set. Suicidality | Suicidality monitored during the |
| | monitored during the trial using | trial using the C-SSRS |
| | the C-SSRS | |
| Section 8.1: Packaging | Each blister card used in the trial | Each blister card used in the trial |
| and Labeling | will be given an identifying | will be given an identifying |
| | number and will be labeled to | number and will be labeled to |
| | clearly disclose the blister card | clearly disclose the blister card |
| | number, Subject ID (to be filled | number, Subject ID (to be filled in |
| | in by the site staff/investigator), | by the site staff/investigator), |
| | subject's initials, name of the | subject's initials or other unique |
| | investigator (to be filled in by the | identifier, name of the |
| | site staff/investigator), site | investigator (to be filled in by the |
| | number (to be filled in by the site | site staff/investigator), site |
| | staff/investigator), subject's | number (to be filled in by the site |
| | initials (to be filled in by the site | staff/investigator), subject's |
| | staff/investigator), date dispensed | initials (to be filled in by the site |
| | (to be filled in by the site | staff/investigator), date dispensed |
| | staff/investigator), compound ID, | (to be filled in by the site |
| | protocol number, the sponsor's | staff/investigator), compound ID, |
| | name and address, instructions | protocol number, the sponsor's |
| | for use, route of administration, | name and address, instructions for |
| | and appropriate precautionary | use, route of administration, and |

| | statements. | appropriate precautionary |
|---|---|---|
| | | statements. |
| | Subjects must remain on the same ADT for the duration of the trial (ie, Screening/Baseline through Week 52/ET). | Subjects must remain on the same ADT for the duration of the trial (ie, Screening/Baseline through Week 26/ET). |
| Section 8.5: Reporting | | A Product Quality Complaint |
| of Product Quality | | (PQC) is any written, electronic, |
| Complaints | | or verbal communication by a |
| | | healthcare professional, |
| | | consumer, subject, medical |
| | | representative, Competent |
| | | Authority, regulatory agency, |
| | | partner, affiliate or other third |
| | | party that alleges deficiencies or |
| | | dissatisfaction related to identity, |
| | | quality, labeling, packaging, |
| | | reliability, safety, durability, |
| | | tampering, counterfeiting, theft, |
| | | effectiveness or performance of a |
| | | drug product or medical device |
| | | after it is released for distribution. |
| | | Examples include, but are not |
| | | limited to, communications |
| | | involving: |
| | | Failure/malfunction of a product to meet any of its specifications |

| | Incorrect or missing labeling |
|---|---|
| | Packaging issues (eg,<br>damaged, dirty, crushed,<br>missing product) |
| | Blister defects (eg, missing, empty blisters) |
| | Bottle defects (eg,<br>under/over-fill, no safety<br>seal) |
| | Vial defects |
| | Product defect (eg, odor, chipped, broken, embossing illegible) |
| | Loss or theft of product |
| Section 8.5.1: Eliciting | The investigator or designee must |
| and Reporting Product | record all PQCs identified |
| <b>Quality Complaints</b> | through any means from the |
| | receipt of the IMP from sponsor |
| | through and including |
| | reconciliation and up to |
| | destruction, including subject |
| | dosing. The investigator or |
| | designee must notify the sponsor |
| | (or sponsor's designee) must be |
| | notified within 24 hours of |
| | becoming aware of the PQC by e- |
| | mail or telephone and according |
| | to the procedure outlined below: |
| | Online – Send information |

| | required for reporting purposes (listed below) to OAPI- EQCProductComplaints@Ot suka-us.com • Phone - Rocky Mountain Call Center at 1-800-438-6055. Identification of a PQC by the subject should be reported to the site investigator, who should then follow one of the reporting mechanisms above. |
|---|---|
| Section 8.5.2: | Description of compliant |
| Information Required | Reporter identification (eg, |
| for Reporting Purposes | subject, investigator, site, etc) Reporter contact information (eg, address, phone number, e-mail address.) ID of material (product/compound name, coding) Clinical protocol reference (number and/or trial name) Dosage form/strength (if known) Pictures (if available) Availability for return |
| Section 8.5.3: Return | Indicate during the report of the |
| Process | PQC if the complaint sample is |
| | available for return. If complaint sample is available for return, |

| | | return it in the product retrieval |
|---|---|---|
| | | package, which will be provided |
| | | by OAPI-EQC. |
| | | It should be documented in the site accountability record that a |
| | | complaint sample for a dispensed |
| | | kit has been forwarded to OAPI- |
| | | EQC for complaint investigation. |
| Section 8.5.4: | | Assessment and evaluation of |
| Assessment/Evaluation | | Product Quality complaints will |
| | | be handled by OAPI EQC QM |
| | | group. |
| Section 9.4: Records | FDA regulations require all | Regulatory requirements for the |
| Retention at the Trial | investigators participating in | archival of records for this trial |
| Site | clinical drug trials to maintain | necessitate that participating |
| | detailed clinical data for one of | investigators maintain detailed |
| | the following periods: | clinical data for the longest of the |
| | A period of at least 3 years | following three periods |
| | following the date on which a New Drug Application is approved by the FDA. A period of 3 years after the sponsor notifies the investigator that no further application is to be filed with the FDA. | • A period of at least 2 years following the date on which approval to market the drug is obtained (or if IMP development is discontinued, the date regulatory authorities were notified of discontinuation); OR |
| | | A period of at least 3 years<br>after the sponsor notifies the<br>investigator that the final<br>report has been filed with |

The investigator must not dispose of any records relevant to this trial without either (1) written permission from the sponsor or (2) provision of an opportunity for the sponsor or designated agent to collect such records. The investigator will be responsible to maintain adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial, including the eCRF data on the CD-ROM and any data clarification forms received from the sponsor (or sponsor's designee). Such documentation is subject to inspection by the sponsor, sponsor's designee, and relevant regulatory agencies. If the investigator withdraws from the trial (eg, due to relocation or retirement), all trial related records should be transferred to a

- regulatory authorities.
- Longer, region-specific storage requirements, if applicable.

The investigator must not dispose of any records relevant to this trial without either (1) written permission from the sponsor or (2) provision of an opportunity for the sponsor or designated agent to collect such records. The investigator will be responsible to maintain adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial, including the eCRF data on the CD ROM and any data clarification forms received from the sponsor (or sponsor's designee). Such documentation is subject to inspection by the sponsor, sponsor's designee, and relevant regulatory agencies. If the investigator withdraws from the trial (eg, due to relocation or retirement), all trial related records should be transferred to a mutually agreed upon designee

| | mutually agreed upon designee. | within a sponsor-specified |
|---|---|---|
| | Notice of such transfer will be | timeframe. Notice of such |
| | given to the sponsor (or designee) | transfer will be given to the |
| | in writing. | sponsor (or designee) in writing. |
| Section 12: | Subjects will be identified only Subjects will be identified only | |
| Confidentiality | by initials and unique subject | initials and unique subject |
| | numbers in eCRFs. Their full | numbers in eCRFs. Per country |
| | names may, however, be made | regulations, if subject initials |
| | known to a regulatory agency or | cannot be collected, another |
| | other authorized officials if | unique identifier will be used. |
| | necessary. | Their full names may, however, |
| | | be made known to a regulatory |
| | | agency or other authorized |
| | | officials if necessary. |
| Appendix 1 | Current Contacts | Revised Contacts |
| Appendix 1 | | Revised Contacts |
| Appendix 1 | Current Contacts Primary Medical Contact: | Revised Contacts |
| Appendix 1 | | Revised Contacts |
| Appendix 1 | | Revised Contacts |
| Appendix 1 | | Revised Contacts |
| Appendix 1 | | Revised Contacts |
| Appendix 1 | | Revised Contacts Phone |
| Appendix 1 | Primary Medical Contact: | |
| Appendix 1 | Primary Medical Contact: | Phone<br>Mobile |
| Appendix 1 | Primary Medical Contact: Phone Fax | Phone |
| Appendix 1 | Primary Medical Contact: | Phone<br>Mobile |





Protocol 331-10-238

# **Current Figure 3.1-1**



# **Revised Figure 3.1-1**



| Table 4.2.2.2-2 Dosing Schedule for Brexpiprazole | | | | | |
|---|---|---|---|---|---|
| | Trial Visit | | | | |
| IMP | Screening/<br>Baseline | Week 1 <sup>a</sup> | Week 2 <sup>b</sup> | Week 4 <sup>b</sup> | Visits at Weeks 8, 14, 20, 26, 32, 38, and 44 |
| Brexpiprazole (mg/day) <sup>c</sup> | 0.5 | 1 | 0.5, 1 or 2 | 0.5, 1, 2 or 3 | 0.5, 1, 2, or 3 |
| ADT <sup>d</sup> | Final dose<br>from double-<br>blind trial | No change | No change | No change | Change to ADT dose is permitted as described in Section 3.2.2.2. |

<sup>&</sup>lt;sup>a</sup>Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit.

bStep-wise increases in the dose of brexpiprazole must be separated by at least 5 days. Although step-wise decreases in the brexpiprazole dose are permitted at any time after the Week 1 visit to a minimum of 0.5 mg/day, an interval of at least 5 days between dose adjustments is recommended. See Section 3.2.2.1 for additional information on dose adjustments. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

<sup>&</sup>lt;sup>c</sup>Subjects unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial.

<sup>&</sup>lt;sup>d</sup>Throughout Trial 331-10-238, the subject must remain on the same ADT that was assigned in the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>e</sup>It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized.

| Revised Tal | ble 4.2.2.2- | for Brexpi | prazole | | |
|---|---|---|---|---|---|
| | Trial Visit | | | | |
| IMP | Screening/<br>Baseline | Week 1 <sup>a</sup> | Week 2 <sup>b</sup> | Week 4 <sup>b</sup> | Visits at Weeks 8, 14, and 20 b |
| Brexpiprazole (mg/day) <sup>c</sup> | 0.5 | 1 | 0.5, 1 or 2 | 0.5, 1, 2 or 3 | 0.5, 1, 2, or 3 |
| ADT | Final dose from double-blind trial | No change e | No change | No change | Change to ADT dose is permitted as described in Section 3.2.2.2. |

<sup>&</sup>lt;sup>a</sup>Subjects unable to tolerate brexpiprazole 1 mg/day may decrease to 0.5 mg/day at any time after the Week 1 visit.

bStep-wise increases in the dose of brexpiprazole must be separated by at least 5 days. Although step-wise decreases in the brexpiprazole dose are permitted at any time after the Week 1 visit to a minimum of 0.5 mg/day, an interval of at least 5 days between dose adjustments is recommended. See Section 3.2.2.1 for additional information on dose adjustments. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole (increases or decreases) are required between scheduled visits.

<sup>&</sup>lt;sup>c</sup>Subjects unable to tolerate the minimum dose of brexpiprazole (ie, 0.5 mg/day) must be withdrawn from the trial.

d Throughout Trial 331-10-238, the subject must remain on the same ADT that was assigned in the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>e</sup>It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized.

| Current Table 3.6.1 | Schedule o | of Asse | ssmen | ts | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening/ Open-Label Treatment Phase Visit Week (± 2 days) | | | | | | | | | | Follow-up <sup>c</sup> | | |
| Assessment | Baseline | 1 | 2 | 4 | 8 | 14 | 20 | 26 | 32 | 38 | 44 | <b>52/ET</b> <sup>b</sup> | 30 (+2) days |
| ENTRANCE CRITERIA | | | | | | • | l | | | • | • | ' | |
| Informed consent d | X | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | | | | | |
| Medical history | xe | | | | | | | | | | | | |
| EFFICACY | | I | I | | | | I | | I | | | <u> </u> | |
| CGI-S | X | X | X | X | X | X | X | X | X | X | X | X | |
| CGI-I <sup>f</sup> | | X | X | X | X | X | X | X | X | X | X | X | |
| SDS | X | | | | X | | | X | | | | X | |
| IDS-SR | X | | | | X | X | X | X | | X | | X | |
| SAFETY | | | | | | | | | | | | | |
| Physical examination | X | | | | X | | | X | | | | X | |
| Waist circumference | X | | | | X | X | X | X | X | X | X | X | |
| Vital signs <sup>g</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>h</sup> | X | X | | X | X | X | | X | | X | | X | |
| Clinical laboratory tests | X <sup>j</sup> | $X^k$ | | X <sup>k</sup> | X <sup>k</sup> | $X^k$ | | X <sup>k</sup> | | $X^k$ | | $X^k$ | |
| ACTH, cortisol, and HbA1c | X | $X^k$ | | X <sup>k</sup> | X <sup>k</sup> | X <sup>k</sup> | | X <sup>k</sup> | | X <sup>k</sup> | | $X^k$ | |
| Drug screen/blood alcohol | X | X | | X | X | X | | X | | X | | X | |
| Urine pregnancy test (WOCBP only) <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| SAS | X | X | X | X | X | X | X | X | X | X | X | X | |
| AIMS | X | X | X | X | X | X | X | X | X | X | X | X | |
| BARS | X | X | X | X | X | X | X | X | X | X | X | X | |
| C-SSRS <sup>n</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| MSFQ | X | X | X | | X | | | X | | | | X | |

| Current Table 3.6.1 | Schedule o | f Asse | ssmen | ts | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening/ | | Open-Label Treatment Phase Visit Week (± 2 days) | | | | | | | | | | Follow-up <sup>c</sup> |
| Assessment | Baseline <sup>a</sup> | 1 | 2 | 4 | 8 | 14 | 20 | 26 | 32 | 38 | 44 | <b>52/ET</b> <sup>b</sup> | 30 (+2) days |
| Adverse events | X <sup>o</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| OTHER | | | • | | • | | | • | | • | | | |
| Dose adjustments <sup>q</sup> | | X | X | X | X | X | X | X | X | X | X | | |
| RUF <sup>r</sup> | X | | | | X | | | X | | | | X | |
| Register visit in IVRS/IWRS <sup>S</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| IMP dispensing | X | X | X | X | X | X | X | X | X | X | X | | |
| IMP accountability | | X | X | X | X | X | X | X | X | X | X | X | |

IVRS = interactive voice response system; IWRS = interactive web response system; WOCBP = women of childbearing potential.

<sup>&</sup>lt;sup>a</sup>Screening for Trial 331-10-238 occurs simultaneously with Baseline at the last scheduled visit of the prior double-blind phase 3 trial. All assessments listed under screening need to be performed at Screening/Baseline of Trial 331-10-238; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.

<sup>&</sup>lt;sup>b</sup>If a subject discontinues prematurely before Week 52, procedures noted for Week 52 must be completed at the early termination (ET) visit.

<sup>&</sup>lt;sup>c</sup>Consists of telephone contact or clinic visit (investigator's discretion) for evaluation of safety and applies to all subjects (completers and early withdrawals).

<sup>&</sup>lt;sup>d</sup>Informed consent for Trial 331-10-238 will occur at Screening/Baseline and must be obtained before any trial-related procedures specific to the open-label trial are performed.

<sup>&</sup>lt;sup>e</sup>Update, if necessary.

fImprovement should be based on the subject's status at the last scheduled visit of the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>g</sup>Vital signs include body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Blood pressure and heart rate will be measured in the following order: supine, sitting, and standing after the subject has been in each position for at least 3 minutes. Vital signs scheduled for the same visit as blood samples are to be completed before blood is drawn.

h Standard 12-lead ECGs will be performed after the subject has been supine and at rest for ≥ 5 minutes prior to the ECG. A central ECG service will be utilized to review all ECGs in order to standardize interpretations for the safety analysis. In addition, ECG results will be evaluated at the investigational site to monitor safety during the trial. Subjects will be enrolled in Trial 331-10-238 based on the screening/baseline ECG results from the trial site. If the screening/baseline ECG results from the central reader (ie, the last scheduled visit of the prior double-blind phase 3 trial), when available, indicate a QTcF

- $\geq$  450 msec at screening/baseline, the investigator must contact the medical monitor to discuss the subject's continued participation in the trial. ECGs scheduled for the same visit as blood samples are to be completed before blood is drawn.
- <sup>1</sup>Includes hematology (including PT, aPTT, and INR), serum chemistry (including prolactin and TSH, with reflex to free thyroxine [T<sub>4</sub>] if the result for TSH is abnormal), and urinalysis.
- <sup>J</sup>Subjects must be fasting for a minimum of 8 hours prior to blood draws for screening/baseline laboratory assessments (ie, the last scheduled visit of the prior double-blind phase 3 trial).
- <sup>k</sup>Clinical laboratory tests should be drawn fasting, if possible, but must be drawn after a minimum 8-hour fast at Week 52/ET. Vital sign and ECG assessments should be completed before any blood samples are collected.
- A urine drug screen and a blood alcohol test are required at the designated times, but either or both can be conducted at any time during the trial at the discretion of the investigator.
- <sup>m</sup>All positive urine pregnancy test results must be confirmed by a serum test. Subjects with a positive serum pregnancy test result at Screening/Baseline must not be enrolled in Trial 331-10-238 and subjects with a positive serum pregnancy test result during the trial must discontinue treatment and be withdrawn from the trial. Pregnancy tests can be performed at any point during the trial if pregnancy is suspected.
- <sup>n</sup> "Since Last Visit" C-SSRS form.
- <sup>o</sup>AE recording will begin with the signing of the ICF for Trial 331-10-238.
- <sup>p</sup>All prescription and non-prescription medications taken during the trial will be recorded as concomitant medications. Details of prohibited and restricted medications are provided in Section 4.
- <sup>q</sup>Adjustments to the dose of brexpiprazole or ADT are permitted to optimize efficacy and tolerability as described in Section 3.2. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). At least 5 days must elapse between dose increases for brexpiprazole and ADT. An interval of at least 5 days between dose adjustments is also recommended for dose decreases; however, the investigator may decrease the dose of brexpiprazole or ADT as needed for tolerability according to the rules described in Section 3.2.2. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole or ADT (increases or decreases) are required between scheduled visits. All eligible subjects entering from prior double-blind phase 3 brexpiprazole MDD trials must be able to continue therapy without interruption between the double-blind and open label trials.

<sup>&</sup>lt;sup>r</sup>Baseline RUF is completed at Screening/Baseline for all subjects. The Follow-up RUF is completed at all other visits.

<sup>&</sup>lt;sup>S</sup>The IVRS/IWRS will be accessed at unscheduled visits if new blister cards are dispensed for dose adjustment of brexpiprazole.

| Assessment | Screening/<br>Baseline <sup>a</sup> | O | days) | Follow-up <sup>c</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseinie | 1 | 2 | 4 | 8 | 14 | 20 | <b>26/ET</b> <sup>b</sup> | 30 (+2) days |
| ENTRANCE CRITERIA | | • | | | | • | | | |
| Informed consent d | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | |
| Medical history | X <sup>e</sup> | | | | | | | | |
| EFFICACY | | 1 | | | | | | | |
| CGI-S | X<br>X | X | X | X | X | X | X | X<br>X | |
| CGI-I <sup>f</sup> | X | | | | | X | | X | |
| SDS | X | | | | | X | | X | |
| IDS-SR | X | | | | | X | | X | |
| SAFETY | | | | | | | | | |
| Physical examination | X | | | | | | | X | |
| Waist circumference | X | | | | | X | | X | |
| Vital signs <sup>g</sup> | X | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>h</sup> | X | | | | | X | | X | |
| Clinical laboratory tests <sup>1</sup> | X <sup>j</sup> | | | | | X <sup>k</sup> | | X <sup>k</sup> | |
| HbA1c | X <sup>j</sup> | | | | | $X^k$ | | $X^k$ | |
| Drug screen/blood alcohol | X | X | | X | X | X | | X | |
| Urine pregnancy test | X | X | X | X | X | X | X | X | |
| (WOCBP only) <sup>m</sup> | | | | | | | | | |
| SAS | X | X | X | X | X | X | X | X | |
| AIMS | X | | | | | X | | X | |
| BARS | X | X | X | X | X | X | X | X | |
| C-SSRS <sup>n</sup> | X | X | X | X | | X | | X | |
| MSFQ | X | | | | | | | X | |
| Adverse events | X <sup>o</sup> | X | X | X | X | X | X | X | X |

| Concomitant medications <sup>p</sup> | X | X | X | X | X | X | X | X | X |
|------------------------------------------|---|---|---|---|---|---|---|---|---|
| OTHER | | | | | | | | | |
| Dose adjustments <sup>q</sup> | | X | X | X | X | X | X | | |
| RUF <sup>r</sup> | X | | | | | | | X | |
| Register visit in IVRS/IWRS <sup>S</sup> | X | X | X | X | X | X | X | X | |
| IMP dispensing | X | X | X | X | X | X | X | | |
| IMP accountability | | X | X | X | X | X | X | X | |

IVRS = interactive voice response system; IWRS = interactive web response system; WOCBP = women of childbearing potential.

<sup>&</sup>lt;sup>a</sup>Screening for Trial 331-10-238 occurs simultaneously with Baseline at the last scheduled visit of the prior double-blind phase 3 trial. All assessments listed under screening need to be performed at Screening/Baseline of Trial 331-10-238; if any of these assessments were conducted at the last scheduled visit of the prior double-blind phase 3 trial, then Screening/Baseline values for those assessments will be derived from that visit and those assessments will not need to be repeated at Screening/Baseline of Trial 331-10-238.

If a subject discontinues prematurely before Week 26, procedures noted for Week 26 must be completed at the early termination (ET) visit. Subjects who have completed 26 weeks or more, will have the Week 26/ET procedures at their next scheduled visit.

<sup>&</sup>lt;sup>c</sup>Consists of telephone contact or clinic visit (investigator's discretion) for evaluation of safety and applies to all subjects (completers and early withdrawals).

d Informed consent for Trial 331-10-238 will occur at Screening/Baseline and must be obtained before any trial-related procedures specific to the open-label trial are performed.

<sup>&</sup>lt;sup>e</sup>Update, if necessary.

Improvement should be based on the subject's status at the last scheduled visit of the prior double-blind phase 3 trial.

<sup>&</sup>lt;sup>g</sup>Vital signs include body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Blood pressure and heart rate will be measured in the following order: supine, sitting, and standing after the subject has been in each position for at least 3 minutes. Vital signs scheduled for the same visit as blood samples are to be completed before blood is drawn.

h Standard 12-lead ECGs will be performed after the subject has been supine and at rest for ≥ 5 minutes prior to the ECG. A central ECG service will be utilized to review all ECGs in order to standardize interpretations for the safety analysis. In addition, ECG results will be evaluated at the investigational site to monitor safety during the trial. Subjects will be enrolled in Trial 331-10-238 based on the screening/baseline ECG results from the trial site. If the screening/baseline ECG results from the central reader (ie, the last scheduled visit of the prior double-blind phase 3 trial), when available, indicate a QTcF ≥ 450 msec at screening/baseline, the investigator must contact the medical monitor to discuss the subject's continued participation in the trial. ECGs scheduled for the same visit as blood samples are to be completed before blood is drawn.

Includes hematology (including PT, aPTT, and INR), serum chemistry (including prolactin and TSH, with reflex to free thyroxine [T<sub>4</sub>] if the result for TSH is abnormal), and urinalysis.

<sup>&</sup>lt;sup>J</sup>Subjects must be fasting for a minimum of 8 hours prior to blood draws for screening/baseline laboratory assessments (ie, the last scheduled visit of the prior double-blind phase 3 trial).

k Clinical laboratory tests should be drawn fasting, if possible, but must be drawn after a minimum 8-hour fast at Week 26/ET. Vital sign and ECG assessments should be completed before any blood samples are collected.

A urine drug screen and a blood alcohol test are required at the designated times, but either or both can be conducted at any time during the trial at the discretion of the investigator.

<sup>&</sup>lt;sup>m</sup>All positive urine pregnancy test results must be confirmed by a serum test. Subjects with a positive serum pregnancy test result at Screening/Baseline must not be enrolled in Trial 331-10-238 and subjects with a positive serum pregnancy test result during the trial must discontinue treatment and be withdrawn from the trial. Pregnancy tests can be performed at any point during the trial if pregnancy is suspected.

<sup>&</sup>quot;Since Last Visit" C-SSRS form.

<sup>&</sup>lt;sup>o</sup>AE recording will begin with the signing of the ICF for Trial 331-10-238.

<sup>&</sup>lt;sup>p</sup>All prescription and non-prescription medications taken during the trial will be recorded as concomitant medications. Details of prohibited and restricted medications are provided in Section 4.

<sup>&</sup>lt;sup>q</sup>Adjustments to the dose of brexpiprazole or ADT are permitted to optimize efficacy and tolerability as described in Section 3.2. It is recommended that the dose of ADT not be changed while the dose of brexpiprazole is being optimized (ie, no change to ADT up to and including the Week 4 visit). At least 5 days must elapse between dose increases for brexpiprazole and ADT. An interval of at least 5 days between dose adjustments is also recommended for dose decreases; however, the investigator may decrease the dose of brexpiprazole or ADT as needed for tolerability according to the rules described in Section 3.2.2. Subjects must return to the clinic for unscheduled visits if changes to the dose of brexpiprazole or ADT (increases or decreases) are required between scheduled visits. All eligible subjects entering from prior double-blind phase 3 brexpiprazole MDD trials must be able to continue therapy without interruption between the double-blind and open label trials.

Baseline RUF is completed at Screening/Baseline for all subjects. The Follow-up RUF (as well as hospitalization questions) is completed at ET visit.

The IVRS/IWRS will be accessed at unscheduled visits if new blister cards are dispensed for dose adjustment of brexpiprazole.

| Section 3.6.2.1: Clinical | |
|---|---|
| Laboratory Tests | |
| Current Table | |
| Table 3.6.2.1-1 Safety Clinical Laboratory Tests | |
| Hematology: | Serum Chemistry: |
| WBC count with differential | ALP |
| RBC count | ALT or SGPT |
| Hematocrit | AST or SGOT |
| Hemoglobin | BUN |
| Platelet count | CPK |
| | Creatinine |
| <u>Urinalysis:</u> | LDH |
| рН | Total bilirubin |
| Specific gravity | Triglycerides |
| Protein | Cholesterol (total, LDL, and HDL) |
| Ketones | Calcium |
| Glucose | Chloride |
| Blood | Glucose |
| Microscopic exam (performed only if any part o | f Insulin |
| the urinalysis is not negative) | Magnesium |
| | Bicarbonate |
| <u>Urine Drug Screens:</u> | Inorganic phosphorous |
| Amphetamines | Sodium |
| Barbiturates | Potassium |
| Benzodiazepines | Total protein |
| Cannabinoids | Uric acid |
| Cocaine | GGT |
| Marijuana | Prolactin |
| Methadone | Albumin |
| Opiates | |
| Phencyclidine | Additional Tests: |
| Propoxyphene | Urine pregnancy (WOCBP) <sup>a</sup> |
| Other: | TSH, with reflex to free T <sub>4</sub> if TSH is abnormal |
| Blood alcohol | PT, aPTT, and INR |
| Dioog alcolloi | ACTH |
| | Cortisol |
| | HbA1c |
| | 1101110 |

#### **Revised Table**

### **Table 3.6.2.1-1** Safety Clinical Laboratory Tests

Hematology: Serum Chemistry:

WBC count with differential ALP

RBC count ALT or SGPT
Hematocrit AST or SGOT
Hemoglobin BUN

Platelet count

CPK

Creatinine

<u>Urinalysis:</u> pH Total bilirubin

Specific gravity
Protein
Triglycerides
Cholesterol (total, LDL, and HDL)

Ketones Calcium
Glucose Chloride
Blood Glucose

Microscopic exam (performed only if any part of the urinalysis is not negative)

Insulin

Magnesium

 Urine Drug Screens:
 Inorganic phosphorous

 Amphetamines
 Sodium

 Post scrippe

Barbiturates Potassium
Benzodiazepines Total protein
Cannabinoids Uric acid
Cocaine GGT
Marijuana Prolactin
Methadone Albumin

Opiates
Phencyclidine
Propoxyphene

Additional Tests:
Urine pregnancy (WOCBP)

Other: TSH, with reflex to free T<sub>4</sub> if TSH is abnormal

Bicarbonate

Blood alcohol PT, aPTT, and INR

HbA1c

**Amendment Number:** 4

**Issue Date:** 13 Jun 2014

#### **PURPOSE:**

The sponsor has determined the need for a fourth Amendment to make the following administrative changes:

- include C-SSRS assessment at week 8 and week 20 (removed in error from amendment 3 issued on 11 Apr 2014)
- update sponsor contact details

## **General Revisions:**

• Changes made to Protocol 331-10-238 in this fourth amendment are as outlined above. Changes by section are provided below.

| Location | Current Text | Revised Text |
|---|---|---|
| Title Page | Phone Fax E-mail: | Phone Fax E-mail: |
| Table 3.6-1<br>Schedule of<br>Assessments | | C-SSRS added X at week 8 and 20 |
| 3.6.1.5<br>Week 8 | | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. |
| 3.6.1.7<br>Week 20 | | The investigator (or qualified designee) will complete the "Since Last Visit" C-SSRS form. |

#### Agreement

I, the undersigned principal investigator, have read and understand the protocol (including the Investigator's Brochure) and agree that it contains all the ethical, legal and scientific information necessary to conduct this trial in accordance with the principles of Good Clinical Practices and as described herein and in the sponsor's (or designee's) Clinical Research Agreement.

I will provide copies of the protocol to all physicians, nurses and other professional personnel to whom I delegate trial responsibilities. I will discuss the protocol with them to ensure that they are sufficiently informed regarding the investigational new drug, OPC-34712, the concurrent medications, the efficacy and safety parameters and the conduct of the trial in general. I am aware that this protocol must be approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) responsible for such matters in the clinical trial facility where 331-10-238 will be tested prior to commencement of this trial. I agree to adhere strictly to the attached protocol (unless amended in the manner set forth in Paragraph I of the sponsor's Clinical Research Agreement, at which time I agree to adhere strictly to the protocol as amended).

I understand that this IRB- or IEC-approved protocol will be submitted to the appropriate regulatory authority/ies by the sponsor. I agree that clinical data entered on case report forms by me and my staff will be utilized by the sponsor in various ways such as for submission to governmental regulatory authorities and/or in combination with clinical data gathered from other research sites, whenever applicable. I agree to allow sponsor monitors and auditors full access to all medical records at the research facility for subjects screened or enrolled in the trial.

I agree to await IRB/IEC approval before implementation of any protocol amendments to this protocol. If, however, there is an immediate hazard to subjects, I will implement the amendment immediately, and provide the information to the IRB/IEC within 5 working days. Administrative changes to the protocol will be transmitted to the IRB/IEC for informational purposes only.

I agree to provide all subjects with informed consent forms, as required by the applicable regulations and by ICH guidelines. I agree to report to the sponsor any adverse experiences in accordance with the terms of the sponsor's Clinical Research Agreement and the relevant regional regulation(s) and guideline(s). I further agree to provide all required information regarding financial certification or disclosure to the sponsor for all investigators and sub-investigators in accordance with the terms of the relevant regional regulation(s). I understand that participation in the protocol involves a commitment to publish the data from this trial in a cooperative publication prior to publication of efficacy and safety results on an individual basis.

| <b>-</b> | | | |
|-------------------|-----------------|-----------------|--------------|
| Principal or Coor | dinatina Invest | idator Sidnatur | e and I )ate |

# Otsuka Pharmaceutical Development & Commercialization, Inc. This page is a manifestation of an electronically captured signature

OPC-34712

SIGNATURE PAGE

Document Name: 331-10-238 Amendment 04

Document Number: 0001108835

**Document Version: 3.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'GMT'Z) |
|-----------|------------------------|----------------------------------------|
| | Biostatistics Approval | 13-Jun-2014 21:02 GMT+00 |
| | Clinical Approval | 13-Jun-2014 21:04 GMT+00 |